Previous Version (Amendment 03): V6.0 Current Version (Amendment 04): V7.0

Date of Revisions: 05 Feb 2018

| Change | Rationale | <b>Affected Protocol Sections</b> |
|---|---|---|
| Revised order of key | To incorporate feedback | Synopsis – Objectives |
| secondary objectives and | from regulatory authorities | Synopsis – Statistical |
| related endpoints | | Methods |
| - | | Synopsis – Sample Size |
| | | Rationale |
| | | Section 8.2.1 |
| | | Section 9.7.1.1.2 |
| | | Section 9.7.1.6 |
| | | Figure 2 |
| | | Section 9.7.1.6.2 |
| | | Section 9.7.2 |
| Added sensitivity analysis | To incorporate feedback | Section 9.7.1.6.1 |
| | from regulatory authorities | |
| Revised process for Control | To align with revised order | Section 9.7.1.6 |
| of Type I Error | of objectives and endpoints | |
| Revised age ranges for | Correction | Synopsis – Statistical |
| categorical variables | | Methods |
| | | Section 9.7.1.4 |
| | | Section 9.7.1.6.1 |

Revision History:
Previous Version (Amendment 02): V5.0
Current Version (Amendment 03): V6.0

Date of Revisions: 16 Jun 2017

| Change | Rationale | <b>Affected Protocol Sections</b> |
|---|---|---|
| Revised order of Primary, Key | To incorporate feedback | Synopsis – Objectives |
| Secondary, Additional | from regulatory | Synopsis – Statistical |
| Secondary, and Exploratory | authorities | Methods |
| objectives and related endpoints | | Synopsis – Sample Size |
| | | Rationale |
| | | Section 7.2 |
| | | Section 8.1 |
| | | Section 8.2 |
| | | Section 8.3 |
| | | Section 9.2.2 |
| | | Section 9.2.3 |
| | | Section 9.2.7 |
| | | Section 9.7.1.1.1 |
| | | Section 9.7.1.1.2 |
| | | Section 9.7.1.1.3 |
| | | Section 9.7.1.6.1 |
| | | Section 9.7.1.6.2 |
| | | Section 9.7.1.6.3 |
| | | Section 9.7.1.8.6 |
| | | Section 9.7.2 |
| Revised process for Control of | To align with revised | Synopsis – Statistical |
| Type I Error | order of objectives and | Methods |
| | endpoints | Section 9.7.1.6 |
| Added WASO1H as a sleep | Correction | Synopsis – Assessments |
| architecture parameter | | Section 9.5.1.3.1 |
| (efficacy) | | |
| Revised description of mornings | Correction | Section 9.5.1.3.2 |
| sleepiness scale | | |
| Revised age groups for analysis | In response to request | Section 9.7.1.4 |
| | from regulatory | |
| | authorities | |
| Revised analysis covariate from | To ensure adequate | Throughout |
| country to region | number of subjects per | |
| | analysis group | |
| Revised Sponsor Signature Page | To reflect current | Sponsor Signature Page |
| | sponsor signatories | |

Previous Version (Amendment 01): V4.0 Current Version (Amendment 02): V5.0 Date of Revisions: 16 Feb 2017

| Date of Revisions: 16 Feb 2017 | | |
|---|---|---|
| Change | Rationale | Affected Protocol Sections |
| Revised approximate<br>number of sites from 90 to<br>105 | To facilitate study enrollment | Synopsis – Site(s) Section 6 Section 9.3 |
| Revised text to allow<br>Sleep Diary entries may be<br>to be maintained in paper<br>format as a backup to the<br>electronic Sleep Diary, if<br>necessary | To allow flexibility in diary data collection in the event electronic diary is not available | Synopsis – Assessments<br>Section 9.5.1.3.2 |
| Revised to Screening Period from up to -28 days to up to -35 days | To allow flexibility in scheduling | Synopsis – Study Design<br>Section 9.1<br>Section 9.1.1.1<br>Figure 1<br>Table 4 |
| Revised total number of expected screened subjects from 2100 to 2800 | To reflect current screen failure rate | Synopsis – Number of<br>Subjects<br>Section 9.3 |
| Revised inclusion (#6) requirement for ISI at both V1 and V3 from "\ge 15" to "\ge 13". | To more accurately target<br>study population (those with<br>chief complaint of sleep<br>maintenance insomnia) for<br>inclusion | Synopsis – Inclusion<br>Criteria<br>Section 9.3.1 |
| Revised inclusion (#9) requirements for time spent in bed requirement from ">9 hours on more than 2 nights per week" to ">10 hours on more than 2 nights per week. | To permit broader inclusion of appropriate subjects | Synopsis – Inclusion<br>Criteria<br>Section 9.3.1 |
| Revised inclusion (#13) to eliminate the need for sleep efficiency component | For consistency throughout protocol | Synopsis – Inclusion<br>Criteria<br>Section 9.3.1 |
| Revised exclusion (#1) for<br>ESS score ">10" to ">15" as<br>an indicator of excessive<br>daytime sleepiness and | Based on ESS data in<br>Study 304 to date, to record<br>excessive sleepiness in<br>medical history instead of | Synopsis – Exclusion<br>Criteria<br>Section 9.3.2<br>Section 9.5.1.2.1 |
| required that scores of 11-15 require excessive daytime sleepiness to be recorded in subject's Medical History) | excluding subjects | |
| Revised exclusion (#3) for MUPS such that endorsing | To allow investigatory follow-up and clinical | Synopsis – Exclusion<br>Criteria |

Previous Version (Amendment 01): V4.0 Current Version (Amendment 02): V5.0 Date of Revisions: 16 Feb 2017

| Date of Revisions: 16 Feb 2017 | | |
|---|---|---|
| Change | Rationale | Affected Protocol Sections |
| item relating to a history of symptoms of Rapid Eye Movement (REM) Behavior Disorder or sleep related violent behavior is no longer automatically exclusionary and clarified requirements with regard to sleep-driving | judgment for subjects who<br>endorse the item regarding a<br>history of "acting out<br>dreams," rather than<br>automatically excluding<br>these subjects | Section 9.3.2 |
| Revised exclusion (#19) for suicidal behavior as per the C-SSRS from a "lifetime" to "in the past 10 years" | To facilitate enrollment and align with other protocols in the program | Synopsis – Exclusion<br>Criteria<br>Section 9.3.2 |
| Revised window around<br>Screening and Run-In Visits | To permit flexibility in scheduling of subjects | Synopsis – Study Design<br>Section 9.1.1.1<br>Section 9.1.1.2<br>Table 4 |
| Revised timing for CDR posture training from "during" for "before" Visit 2a | To permit training on the assessment at Visit 1 | Table 4 |
| Revised analyses for<br>Rebound Insomnia | To match final Study 303 protocol per VHP review | Synopsis – Statistical<br>Methods<br>Section 9.7.1.1.3<br>Section 9.7.1.6.3 |
| Revised the detailed<br>Inclusion/Exclusion Criteria<br>Schedule (Appendix 2) | For clarity | Appendix 2 |
| Revised List of Prohibited<br>Concomitant Medications<br>(Appendix 3) | To correct lists of strong and moderate CYP3A inhibitors and CYP3A inducers | Appendix 3 |
| Deleted Zolpidem Prescribing Information (Appendix 4) | To ensure sites always have<br>the most current approved<br>version (will be provided to<br>sites outside the protocol) | Section 9.4.1<br>Appendix 4 |
| Added the requirement for monitoring of seizures and falls | Per request of FDA | Synopsis – Study Methods<br>Section 9.2.5<br>Table 4 |
| Revised text regarding ECG interpretation categories | For clarity | Section 9.7.1.8.5 |

Previous Version (Amendment 01): V4.0 Current Version (Amendment 02): V5.0 Date of Revisions: 16 Feb 2017

| Change | Rationale | Affected Protocol Sections |
|---|---|---|
| Revised T-BWSQ | For clarity | Synopsis – Study |
| assessment description such | | Assessments |
| that scores above 20 will not | | Section 9.5.1.5.2 |
| be considered clinically | | |
| significant and that the | | |
| symptoms will no longer be | | |
| summarized separately from | | |
| all other AEs. | | |
| Revised Sponsor signature | To reflect current Eisai | Protocol Signature Page |
| page | personnel | |

Previous Version (Revised protocol): V3.0 Current Version (Corrected protocol): V4.0

Date of Revisions: 16 Jul 2016

| Change | Rationale | <b>Affected Protocol Sections</b> |
|---|---|---|
| Corrected typographical | For consistency and | Section 9.3.2 |
| errors in the list of exclusion | editorial quality. No | |
| criteria | changes to content. | |

Previous Version (Revised protocol): V2.0 Current Version (Amended protocol): V3.0 Date of Revisions: 24 Jun 2016

| Date of Revisions: 24 Jun 2016 | | |
|---|---|---|
| Change | Rationale | <b>Affected Protocol Sections</b> |
| Stated in all relevant places<br>in Study Design that<br>subjects will rate their<br>morning sleepiness at 1.5<br>hours after waketime, and<br>specified analysis methods<br>for this assessment | For consistency with<br>Schedule of Assessments<br>and completeness of<br>analysis methods | Synopsis – Study Design<br>Synopsis – Statistical<br>Methods<br>Section 9.1.2.1<br>Section 9.5.1.3.1<br>Section 9.7.1.1.3<br>Section 9.7.1.6.3 |
| Specified that exclusion criteria include current diagnosis of obstructive sleep apnea | Per VHP comment | Synopsis – Exclusion Criteria<br>Section 4<br>Section 9.3.2 |
| Revised STOPBang score cutoff for exclusion from study | To avoid low specificity of more stringent criterion | Synopsis – Exclusion Criteria<br>Section 9.3.2 |
| Revised Epworth Sleepiness<br>Scale score cutoff for<br>exclusion from study | To avoid low specificity of more stringent criterion | Synopsis – Exclusion Criteria<br>Section 9.3.2 |
| Deleted "on a screening questionnaire" from exclusion criterion pertaining to screening for narcolepsy symptoms | No formal screening questionnaire is being utilized | Synopsis – Exclusion Criteria<br>Section 9.3.2 |
| Provided examples of clinically significant disease that would exclude the subject from the study | Per VHP review; to specify conditions for which zolpidem is contraindicated | Synopsis—Exclusion Criteria<br>Section 9.3.2 |
| Stated that subjects taking sedating drugs that would interfere with occupation or activities will be excluded | Per VHP review; to exclude such individuals from the study for reasons of safety | Synopsis – Exclusion Criteria<br>Section 9.3.2 |
| Revised the washout interval between taking a prohibited medication, including treatment for insomnia, and the first dose of study medication | For consistency and to account for medications or insomnia treatments with long half-lives | Synopsis – Exclusion Criteria<br>Section 9.3.2<br>Section 9.4.7.2 |
| Prohibited strong CYP3A inhibitors from being used any time during study, even if intermittently | Per VHP review; based on known drug metabolism interactions with zolpidem | Synopsis – Concomitant Drug<br>Therapy<br>Section 9.3.2<br>Section 9.4.7.2 |

Previous Version (Revised protocol): V2.0 Current Version (Amended protocol): V3.0 Date of Revisions: 24 Jun 2016

| Date of Revisions: 24 Jun 2016 | | |
|---|---|---|
| Change | Rationale | Affected Protocol Sections |
| Clarified that the MUPS to be used is an adapted version | For accuracy | Synopsis – Assessments<br>Section 9.5.1.2.2 |
| Added sleep onset latency as a PSG variable | For completeness of PSG variable dataset | Synopsis – Assessments<br>Section 9.5.1.3.1 |
| Clarified definition of REM latency | For accuracy | Synopsis – Assessments<br>Section 9.5.1.3.1 |
| Changed wording such that sleep diary will ask, not determine, alcohol consumption | For accuracy | Synopsis – Assessments<br>Section 9.5.1.3.2 |
| Allowed flexibility for the means of documenting the time and date of 2 most recent doses before each blood sample for pharmacokinetic analyses | Time and date are being documented by means other than in the electronic Case Report Form | Synopsis – Assessments<br>Section 9.5.1.4.1 |
| Clarified details of the CDR posture assessment at screening | For accuracy | Synopsis Assessments<br>Section 9.5.1.4.2 |
| Deleted statement that all cognitive performance assessment batteries require Yes/No button response | For accuracy – some tasks<br>do not require a Yes/No<br>button response | Synopsis – Assessments<br>Section 9.5.1.4.2 |
| Revised the expected completion time for the full PAB | For accuracy | Synopsis – Assessments<br>Section 9.5.1.4.2 |
| Moved analysis of cognitive<br>PAB tasks from Exploratory<br>to Secondary Analyses | For accuracy | Synopsis – Statistical<br>Methods<br>Section 9.7.1.6.3 |
| Revised method for assessment of rebound insomnia | Per VHP review; to<br>emphasize assessment of<br>rebound insomnia at<br>individual subject level | Synopsis – Statistical<br>Methods<br>Section 9.7.1.6.3 |
| Provided that for applicable countries, the year of birth will be collected instead of the date of birth | To meet requirements in some countries regarding personally identifying information | Section 9.5.1.1 |
| Specified viral tests for hepatitis B and hepatitis C | To provide additional detail of screening assessments | Section 9.5.1.5.5<br>Table 4 (footnote "g") |

Previous Version (Revised protocol): V2.0 Current Version (Amended protocol): V3.0 Date of Revisions: 24 Jun 2016

| Change | Rationale | Affected Protocol Sections |
|---|---|---|
| Deleted alcohol and nicotine/ cotinine from screening for drugs of abuse | To correct an error, as these drugs are not being tested in the urine drug screen in this study | Section 9.5.1.5.5 |
| Corrected window of study days for Screening | To correct an error | Table 4 |
| Clarified interval for reporting of follow-up SAE, pregnancy, or breastfeeding information | Per VHP review; for accuracy | Section 9.5.4.1 |
| Added sentence<br>distinguishing between<br>definitions of "study<br>completer" per protocol<br>versus for statistical analysis<br>purposes | For clarity | Section 9.5.5 |
| Corrected statement referring to study visit at which randomization occurs | To correct an error | Section 9.5.5 |
| Deleted reference to examples of source documents that will not be used in this study | For accuracy | Section 11.3 |
| Deleted glucose-<br>metabolizing agents from<br>list of<br>prohibited/concomitant<br>medications | This prohibition is considered unnecessary. | Appendix 3 |
| Added Appendix 4 – Prescribing Information for Ambien CR® | For reference | Section 9.4.1<br>Appendix 4 |
| Revised signature sheet | Changes in corporate structure | Protocol signature page |

| <b>Revision History:</b> | | |
|---|---|---|
| Previous Version (Original protocol): V1.0 | | |
| Current Version (Revised protocol): V2.0 | | |
| Date of Revisions: 04 Apr 2010 | 6 | |
| Change Rationale Affected Protocol Section | | |
| Specify that an additional | The previous description of | Synopsis – Objectives |
| secondary objective will be | these comparisons did not | Section 8.2.2 |
| the determination of whether | make reference to | |
| LEM5 or LEM10 or both | superiority. | |
| LEM5 and LEM10 are | | |
| superior to ZOL with respect | | |
| to SE, WASO, TST, sSOL, | | |
| sSE, sWASO, and sTST at | | |
| defined time intervals. | | |
| Add an additional secondary | Previously, the comparison | Synopsis – Objectives |
| objective specifying the | of LEM5 and LEM10 to | Synopsis – Statistical |
| evaluation of whether LEM5 | ZOL on LPS was not a | Methods |
| or LEM10 or both LEM5 and | separate additional | Section 8.2.2 |
| LEM10 are superior to ZOL | secondary objective, and | Section 9.7.1.1.2 |
| with respect to LPS, | the previous description of | Section 9.7.1.6.2 |
| separately from comparisons | these comparisons with | |
| of drug effects on other sleep | regard to LPS did not make | |
| measures. | reference to superiority. | |
| Specify that an additional | The previous description of | Synopsis – Objectives |
| secondary objective will be | these comparisons did not | Section 8.2.2 |
| the evaluation of whether | make reference to | |
| LEM5 or LEM10 or both | superiority. | |
| LEM5 and LEM10 are | | |
| superior to ZOL with respect | | |
| to the proportions of sleep | | |
| onset and sleep maintenance | | |
| responders as defined by LPS, | | |
| WASO, sSOL, and sWASO. | | |
| Specify that an additional | The previous description of | Synopsis – Objectives |
| secondary objective will be | these comparisons did not | Section 8.2.2 |
| the evaluation of whether | make reference to | |
| LEM5 or LEM10 or both | superiority. | |
| LEM5 and LEM10 are | | |
| superior to ZOL and PBO | | |
| with respect to ISI and FSS | | |

Previous Version (Original protocol): V1.0 Current Version (Revised protocol): V2.0 Date of Revisions: 04 Apr 2016

| Change Rationale Affected Protocol Sections | | |
|---|---|---|
| Change Add an additional secondary | Previously, these | Synopsis – Objectives |
| objective specifying the | comparisons were an | Section 8.2.2 |
| evaluation of whether LEM5 | exploratory objective, and | Section 6.2.2 |
| or LEM10 or both LEM5 and | the previous description of | |
| LEM10 are superior to ZOL | these comparisons did not | |
| and PBO with respect to | make reference to | |
| cognitive performance the | superiority. | |
| morning after the first 2 nights | superiority. | |
| of treatment. | | |
| State as a separate additional | A separate additional | Synopsis—Statistical |
| secondary endpoint, the | secondary objective was | Methods |
| change of mean LPS from | added for the comparison | Wiethods |
| baseline on Days 1, 2, 29, and | of LEM versus ZOL on | |
| 30 of LEM5 and LEM10 | LPS. Previously this | |
| compared to ZOL | endpoint for LPS was | |
| | combined with other sleep | |
| | variables. | |
| Add the descriptor "potential" | For clarity. It is possible | Section 9.2.5 |
| before cases in the paragraph | that the Cataplexy | |
| describing the process to be | Adjudication Committee | |
| followed regarding the | may review cases that are | |
| Cataplexy Adjudication | adjudicated as events other | |
| Committee. | than cataplexy, but all | |
| | potential cases that may be | |
| | adjudicated as events of | |
| | cataplexy will be flagged | |
| | for review. | |

#### 1 TITLE PAGE



## **Clinical Study Protocol**

**Study Protocol** 

Number:

E2006-G000-304

**Study Protocol Title:** A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Active

> Comparator, Parallel-Group Study of the Efficacy and Safety of Lemborexant in Subjects 55 Years and Older with Insomnia Disorder

Sponsor: Eisai Inc. Eisai Ltd.

> 100 Tice Boulevard European Knowledge Centre

Mosquito Way Woodcliff Lake,

New Jersey 07677 Hatfield, Hertfordshire

AL10 9SN UK US

Investigational

E2006/lemborexant **Product Name:** 

**Indication:** Insomnia

3 Phase:

21 Mar 2016 (original protocol) **Approval Date:** V1.0

> V2.004 Apr 2016 (revised protocol) V3.024 Jun 2016 (per Amendment 01)

V4.0 16 Jul 2016 (per Amendment 01, editorial corrections)

V5.0 16 Feb 2017 (per Amendment 02) V6.0 16 Jun 2017 (per Amendment 03) V7.0 05 Feb 2018 (per Amendment 04)

111,871 **IND Number:** 

2015-004347-39 **EudraCT Number:** 

**GCP Statement:** This study is to be performed in full compliance with International

Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) and all applicable local Good Clinical Practice (GCP) and regulations. All required study documentation

will be archived as required by regulatory authorities.

Confidentiality

This document is confidential. It contains proprietary information of Eisai (the sponsor). Any viewing or disclosure of such information that is not **Statement:** 

authorized in writing by the sponsor is strictly prohibited. information may be used solely for the purpose of reviewing or performing

this study.

Confidential Eisai 

FINAL: (v7.0), 05 Feb 2018

## 2 CLINICAL PROTOCOL SYNOPSIS

Compound No.: E2006

Name of Active Ingredient: Lemborexant

#### **Study Protocol Title**

A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Active Comparator, Parallel-Group Study of the Efficacy and Safety of Lemborexant in Subjects 55 Years and Older with Insomnia Disorder

## Investigator(s)

To be determined

### Site(s)

Approximately 105 sites in North America and Europe (revised per Amendment 02)

#### **Study Period and Phase of Development**

Approximately 64 weeks

Phase 3

#### **Objectives**

### Primary Objective – US and Non-US (revised per Amendment 03)

• Demonstrate using polysomnography (PSG) that lemborexant (LEM10 and LEM5) is superior to placebo (PBO) on objective sleep onset as assessed by latency to persistent to sleep (LPS) after the last 2 nights of 1 month of treatment in subjects 55 years and older with insomnia disorder

## Key Secondary Objectives - US ONLY (revised per Amendment 03)

- Demonstrate that lemborexant (LEM10 and LEM5) is superior to PBO on sleep maintenance as assessed by sleep efficiency (SE) after the last 2 nights of treatment
- Demonstrate that lemborexant (LEM10 and LEM5) is superior to PBO on sleep maintenance as assessed by WASO after the last 2 nights of treatment (revised per Amendments 03 and 04)
- Demonstrate that lemborexant (LEM10 and LEM5) is superior to zolpdiem tartrate extended release 6.25 mg (Ambien CR®; ZOL) on wake after sleep onset in the second half of the night (WASO2H) after the last 2 nights of treatment

## **Key Secondary Objectives – Non-US ONLY (revised per Amendment 03)**

- Demonstrate that lemborexant (LEM10 and LEM5) is superior to PBO on sleep maintenance as assessed by SE after the last 2 nights of treatment
- Demonstrate that lemborexant (LEM10 and LEM5) is superior to PBO on wake after sleep onset (WASO) after the last 2 nights of treatment

## Additional Secondary Objectives - US and Non-US (revised per Amendment 03)

- Demonstrate that LEM5 or LEM10 or both LEM5 and LEM10 are superior to ZOL on postural stability in the morning after the first 2 nights of treatment
- Determine whether the efficacy of LEM5 or LEM10 or both LEM5 and LEM10 is superior to that of ZOL on selected PSG variables after the first 2 nights and the last 2 nights of treatment and on selected Sleep Diary variables over the first 7 nights and the last 7 nights of treatment
- Confirm the efficacy of LEM5 and LEM10 compared to placebo (PBO) on sleep as measured by PSG after the first 2 and last 2 nights of treatment and as measured by Sleep Diary over the first 7 and last 7 nights of treatment
- Evaluate the proportions of sleep onset and sleep maintenance responders to LEM5 and LEM10 and determine whether they are superior to that of ZOL and PBO as defined by response on PSG LPS and WASO and Sleep Diary subjective sleep onset latency (sSOL) and subjective wake after sleep onset (sWASO)
- Evaluate the safety and tolerability of lemborexant
- Determine whether the efficacy of LEM5 or LEM10 or both LEM5 and LEM10 is superior to that of ZOL and PBO on daytime functioning as assessed by the Insomnia Severity Index (ISI) and Fatigue Severity

Scale (FSS) at the end of treatment

• Determine whether the safety of LEM5 or LEM10 or both LEM5 and LEM10 is superior to that of ZOL and PBO as assessed by cognitive performance in the morning after the first 2 nights of treatment

## Exploratory Objectives – US and Non-US (revised per Amendment 03)

- Explore the effects of LEM5, LEM10, ZOL and PBO on:
  - o Subjective quality of sleep
  - o Postural stability in the morning after the last 2 nights of treatment
  - Cognitive performance after the last 2 nights of treatment
  - o Rebound insomnia in the 2 weeks following 30 days of treatment
  - o Subjective ratings of morning sleepiness during and following completion of treatment
  - o Sleep architecture parameters and other PSG variables
  - o Health outcomes on the Patient Global Impression Insomnia (PGI-Insomnia) and EQ-5D-3L
  - o Withdrawal symptoms after completion of treatment
- Summarize plasma concentrations of lemborexant and its metabolites M4, M9, and M10
- Conduct population pharmacokinetic (PK) modeling for lemborexant
- Explore PK/pharmacodynamic (PK/PD) relationships between lemborexant concentrations and efficacy and safety variables

### **Study Design**

E2006-G000-304 is a multicenter, randomized, double-blind, placebo-controlled, active comparator (ZOL), parallel-group study of 2 dose levels of lemborexant for 30 nights in approximately 950 subjects 55 years or older with insomnia disorder. Subjects will be males 65 years or older or females 55 years or older. Approximately 60% of the subjects will be age 65 years or older. (revised per Amendment 03)

The study will have 2 phases: The Prerandomization Phase and the Randomization Phase. The Prerandomization Phase will comprise 3 periods that will last up to a maximum of 35 days: a Screening Period, a Run-in Period, and a Baseline Period. The Randomization Phase will comprise a Treatment Period during which subjects are treated for 30 nights, and a minimum 14-day Follow-up Period before an End of Study (EOS) Visit. (revised per Amendment 02)

Throughout the Prerandomization Phase and the Randomization Phase, all subjects will undergo routine safety assessments at specified visits, including questioning regarding adverse events (AEs), 12-lead electrocardiograms (ECGs), vital signs, weight, height, clinical hematology and chemistry analysis and urinalysis, and suicidality.

## Screening Period

The Screening Period will begin no more than 35 days before the subject is randomized. At the first visit, informed consent will be obtained after the study has been fully explained to each subject and before the conduct of any screening procedures or assessments. A medical, psychiatric, and sleep history interview will be conducted, and will include confirmation that the subject meets diagnostic criteria for insomnia disorder, and further that the subject complains of difficulties with sleep maintenance and/or early morning awakening. Screening assessments will include the ISI, as well as the Epworth Sleepiness Scale (ESS), STOPBang, International Restless Legs Scale (IRLS), and Munich Parasomnia Scale (MUPS), collectively called the Sleep Disorders Screening Battery (SDSB). Other assessments administered will include the FSS and EQ-5D-3L. Additional eligibility criteria will be assessed and safety assessments including the electronic Columbia-Suicide Severity Rating Scale (eC-SSRS) will be conducted. (revised per Amendment 02)

Eligible subjects will be provided with an electronic device on which they will complete the Sleep Diary. Subjects will be trained in the use of this device. Site staff will instruct subjects to complete the diary each morning within 1 hour after morning waketime and will emphasize the importance of doing so. The Sleep Diary entries will be reviewed by site staff at least weekly throughout the study to ensure subject compliance with completion of the Sleep Diary and to ensure that study restrictions are met pertaining to duration of time spent in bed, and use of alcohol. Subjects will also be reminded of study restrictions pertaining to timing of meals and caffeine use.

After subjects have completed the Sleep Diary on at least 7 consecutive mornings, and provided that the Sleep

Diary entries indicate continued eligibility with regard to sleep timing, duration of time spent in bed, and frequency of nights with symptoms of insomnia, subjects will undergo the second screening visit. (Subjects who are not eligible based on Sleep Diary entries will return to the clinic for debriefing purposes and to return study equipment.) This visit must occur between Day -17 and Day -10. On this and all nights on which PSG is recorded, subjects will arrive at the clinic in the evening with sufficient time before bedtime to complete checkin procedures, any scheduled assessments, and preparations (eg, electrode montage placement) for the PSG recordings. In addition, at check-in before all visits at which PSG is to be recorded, subjects will undergo a urine drug test. (revised per Amendment 02)

After check-in has been completed, study personnel will familiarize subjects with the postural stability assessment (Cognitive Drug Research [CDR] posture assessment) and will also conduct a minimum of 2 training sessions for the cognitive performance assessment battery (PAB). Subjects will then undergo an 8-hour PSG recording, to start at the median habitual bedtime (MHB) as calculated from the Sleep Diary entries. The PSG recording will include channels in the electrode montage to screen for symptoms of sleep apnea and periodic limb movement disorder. Within 5 minutes of morning waketime, the CDR posture and PAB assessments will be administered under the same conditions (eg, timing of assessments relative to waketime, ambient lighting), as will be employed during the testing sessions. The CDR posture and PAB assessments at this time are for familiarization purposes only. At 1.5 hours after waketime, subjects will rate their morning sleepiness level. The PSG will be reviewed for exclusion criteria related to symptoms of sleep apnea and/or periodic limb movement disorder. Subjects who continue to meet the eligibility criteria will then be dispensed PBO tablets (single-blind) and will enter the Run-in Period.

#### Run-in Period

The Run-in Period will begin when eligible subjects are dispensed PBO tablets and will continue until the Baseline Period on Day 1. During the Run-in Period subjects will take PBO each night immediately (ie, within 5 minutes) before bedtime (defined as the time the subject intends to try to fall asleep). They will be reminded that they must remain in bed for at least 7 hours each night and maintain a regular bedtime and waketime throughout the study, according to the schedule determined by the study site and the subject. They will also be reminded that they must follow study restrictions with regard to timing of meals and use of caffeine and alcohol.

When subjects have completed the Sleep Diary on at least 7 consecutive mornings during the Run-in Period, the diary will be reviewed for continued eligibility with regard to whether the subject continues to report sWASO ≥60 minutes on at least 3 of the 7 nights, as well as the schedule and duration of time spent in bed. Subjects who are still eligible will return to the clinic for the first of 2 consecutive nights on which PSG will be recorded. The first of these 2 nights must be between Day -10 and Day -4. In the evening, before the PSG recording, the ISI, FSS, and EQ-5D-3L will be assessed. The ISI score will be reviewed for eligibility, and safety assessments will be conducted. Study personnel will administer study drug to subjects within 5 minutes before their scheduled bedtime, which will be at the same MHB as used for the second screening visit. Subjects will undergo an 8-hour PSG. The next morning, subjects will undergo assessments including the CDR posture and PAB assessments, will complete the Sleep Diary, and will rate their morning sleepiness level at 1.5 hours after waketime. (revised per Amendment 01) The PSG recording will be reviewed for continued eligibility and subjects may then leave the clinic only after the investigator determines that is safe for them to do so. (revised per Amendment 02)

Subjects will return to the clinic that evening. Study personnel will administer study drug to subjects within 5 minutes before the scheduled bedtime. A PSG will be recorded overnight. The following morning subjects will undergo postural stability and PAB assessments and will complete the Sleep Diary. At 1.5 hours after waketime, subjects will rate their morning sleepiness level. The PSG recording will be reviewed for continued eligibility, and both PSGs during the Run-in Period will also serve as the baseline for PSG-derived endpoints for subjects who are randomized. Subjects may then leave the clinic after the investigator determines that is safe for them to do so.

Subjects will continue to take study drug at home within 5 minutes before bedtime and they will continue to complete the Sleep Diary each morning within 1 hour after morning waketime. They will again be reminded that they must remain in bed for at least 7 hours each night, maintain a regular bedtime throughout the study, and follow study restrictions with regard to timing of meals and use of caffeine and alcohol.

#### **Baseline Period**

After a minimum of 2 nights following the baseline PSGs, the Run-in Period will end and the Baseline Period will take place. On Day 1, subjects will be admitted to the clinic and the ISI, FSS, and EQ-5D-3L will be administered. Blood and urine samples will be collected for routine safety assessments, an ECG will be performed, and vital signs and weight will be assessed. The eC-SSRS will be administered. Subjects who complete the Baseline Period and continue to meet the eligibility criteria will be randomized, and will begin the Treatment Period. (revised per Amendment 02)

#### Treatment Period

The Treatment Period will begin on Day 1 and will continue until Day 31. Subjects will be randomized in a double-blind manner, to receive LEM5, LEM10, ZOL, or PBO. (revised per Amendment 02)

Within 5 minutes before the subject's MHB, study drug will be administered and an 8-hour overnight PSG will be initiated. At completion of the PSG recording the following morning (Day 2), postural stability will be assessed and the PAB will be conducted immediately thereafter. Subjects will complete the Sleep Diary. At 1.5 hours after waketime, subjects will rate their morning sleepiness level. (revised per Amendment 01) They may leave the clinic after the investigator determines that is safe for them to do so.

On the evening of Day 2, subjects will return to the clinic. A PK blood sample will be collected predose and study drug will be administered within 5 minutes before the subject's MHB, followed by an overnight PSG. The next morning (Day 3), CDR posture and PAB assessments will be conducted and a PK sample will be obtained. Subjects will complete the Sleep Diary. The eC-SSRS will be administered. At 1.5 hours after waketime, subjects will rate their morning sleepiness level. Subjects may then leave the clinic after the investigator determines that is safe for them to do so. Study drug will be dispensed and subjects will be provided with instructions to continue completing the Sleep Diary each morning within 1 hour of waketime and taking study drug daily at home according to the same schedule and with the same instructions as during the Run-in Period.

On Day 29, subjects will return to the clinic. Study drug will be administered within 5 minutes before the subject's MHB, followed immediately by a PSG. On the morning of Day 30, CDR posture and PAB assessments will be conducted. At 1.5 hours after waketime, subjects will rate their morning sleepiness level. Subjects may leave the clinic after the investigator determines that is safe for them to do so.

On the evening of Day 30, subjects will return to the clinic. A PK blood sample will be collected predose and study drug will be administered within 5 minutes before the subject's MHB, followed by a PSG. On the morning of Day 31, CDR posture and PAB assessments will be conducted and a PK sample will be obtained. Then the ISI, FSS, EQ-5D-3L and PGI-Insomnia will be administered. Blood and urine samples will be collected for routine safety assessment. An ECG will be performed, and vital signs and weight will be assessed. The eC-SSRS will be administered. At 1.5 hours after waketime, subjects will rate their morning sleepiness level. Then, after the investigator determines that it is safe for them to do so, subjects will be discharged from the clinic.

#### Follow-up Period

The Follow-up Period will begin when the subjects leave the clinic at the end of the Treatment Period. Subjects will cease to take study drug but will continue to complete the Sleep Diary each morning until the EOS Visit.

At least 14 days but no more than 18 days after completion of the Treatment Period subjects will return to the clinic for the EOS Visit. The Tyrer Benzodiazepine Withdrawal Symptom Questionnaire (T-BWSQ) and eC-SSRS will be administered, and routine safety assessments will be conducted.

A subject who prematurely discontinues taking study drug should return to the clinic as soon as practicable after discontinuing study drug, to complete an Early Termination (ET) Visit. If the subject discontinues from the study due to an AE, the subject must complete an ET Visit and the AE must be followed to resolution or for 2 weeks, whichever comes first. In addition, subjects who withdraw due to an AE should undergo a urine drug test.

#### **Interim Analysis**

An interim analysis is planned to be conducted after approximately 50% of subjects (approximately 475 subjects) have been randomized and either completed Day 31 assessments or discontinued from the study, which is anticipated to occur by the end of July 2017. This interim analysis will be conducted for administrative reasons as detailed in the separate Interim Analysis charter. (revised per Amendment 03)

Adjudication Committee (revised per Amendment 02)

An independent Adjudication Committee will be employed at intervals to review, in a blinded manner, AEs that could potentially be considered cataplexy or seizure. A set of preferred terms constituting a customized Medical Dictionary for Regulatory Activities (MedDRA) query for cataplexy or seizure will be used to identify events for adjudication (including cataplexy, muscle fatigue, muscular weakness, muscle tone disorder, hypotonia, drop attacks, slurred speech, diplopia, falls, convulsions [SMQ narrow and broad], atypical migraine, loss of consciousness, decreased consciousness, myoclonus, syncope, transient global amnesia, lipothymia, and transient ischemic attack). To assist in the preparation of narratives about such events and to support the Committee's adjudication process, investigators and site personnel will be instructed to query subjects who report any of the above events for supplemental information about the events, using a questionnaire for events potentially related to cataplexy and the SAE form for any of the above events considered serious. (revised per Amendment 02)

#### End of Study

Estimates for End of Study are as follows:

- The study will begin in approximately April 2016
- The end of the study will be the date of the last study visit for the last subject in the study.

The estimated duration for each subject on study is anticipated to be a maximum of 81 days (11.5 weeks) consisting of the Screening Period plus Run-in Period plus Baseline Period maximum of 35 days plus Treatment Period plus Follow-up Period and EOS Visit maximum of 53 days. A subject who completes the Treatment Period (assessments through discharge from clinic on the morning of Day 31) will be considered to have completed the study. (revised per Amendment 02)

### **Number of Subjects**

Approximately 2800 subjects will be screened to provide approximately 950 randomized subjects. Subjects will be randomized to one of the following treatment arms: LEM5, LEM10, ZOL, or PBO, in an approximate 5:5:5:4 ratio (n=250:250:250:200). Randomization will be stratified by country and age group (55 to 64 years old; 65 years or older). Approximately 60% of the subjects will be age 65 years or older. (revised per Amendments 02 and 03)

#### **Inclusion Criteria**

- Male age 65 years or older or female age 55 years or older at the time of informed consent
- Meets the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition criteria for Insomnia Disorder, as follows:
  - Complains of dissatisfaction with nighttime sleep, in the form of difficulty staying asleep and/or awakening earlier in the morning than desired despite adequate opportunity for sleep (Note that if the complaint is limited to difficulty initiating sleep, the subject is not eligible)
  - Frequency of complaint  $\geq 3$  times per week
  - Duration of complaint ≥3 months
  - Associated with complaint of daytime impairment
- 3. At Screening: History of subjective WASO (sWASO) typically  $\geq 60$  minutes on at least 3 nights per week in the previous 4 weeks
- At Screening: Reports regular time spent in bed, either sleeping or trying to sleep, between 7 and 9 hours
- At Screening: Reports habitual bedtime, defined as the time the subject attempts to sleep, between 21:00 and 24:00 and habitual waketime between 05:00 and 09:00
- At Screening and at check-in before the first PSG during the Run-in Period: ISI score ≥13 (revised per Amendment 02)
- Confirmation of current insomnia symptoms as determined from responses on the Sleep Diary on the 7 most recent mornings (minimum 5 of 7 for eligibility) before the second screening visit, such that sWASO  $\geq$  60 minutes on at least 3 of the 7 nights
- 8. Confirmation of regular bedtime and waketime as determined from responses on the Sleep Diary on the 7 most recent mornings before the second screening visit, such that neither bedtime, (defined as the time the subject attempts to try to sleep), nor waketime (defined as the time the subject gets out of bed for the day) deviates more than 1 hour on more than 2 nights from the calculated MHB or median habitual waketime

Eisai  (MHW), respectively, from the screening Sleep Diary entries

- 9. Confirmation of sufficient duration of time spent in bed, as determined from responses on the Sleep Diary on the 7 most recent mornings before the second screening visit, such that there are no more than 2 nights with time spent in bed duration < 7 hours or > 10 hours (revised per Amendment 02)
- 10. During the Run-in Period: Reconfirmation of insomnia symptoms, as determined from responses on the Sleep Diary on the 7 most recent mornings before the first PSG during the Run-in Period, such that sWASO ≥ 60 minutes on at least 3 of the 7 nights
- 11. During the Run-in Period: Reconfirmation of regular bedtimes and waketimes as defined in Inclusion Criterion 8
- 12. During the Run-in Period: Reconfirmation of sufficient duration of time spent in bed as defined in Inclusion Criterion 9 (revised per Amendment 02)
- 13. During the Run-in Period: Objective (PSG) evidence of insomnia as follows: WASO average ≥ 60 minutes on the 2 consecutive PSGs, with neither night < 45 minutes (revised per Amendment 02)
- 14. Willing and able to comply with all aspects of the protocol, including staying in bed for at least 7 hours each night
- 15. Willing not to start a behavioral or other treatment program for the treatment of insomnia during the subject's participation in the study

#### **Exclusion Criteria**

- 1. A current diagnosis of sleep-related breathing disorder including obstructive sleep apnea (with or without continuous positive airway pressure [CPAP] treatment), periodic limb movement disorder, restless legs syndrome, circadian rhythm sleep disorder, or narcolepsy, or an exclusionary score on screening instruments to rule out individuals with symptoms of certain sleep disorders other than insomnia as follows: (revised per Amendment 01)
  - a. STOPBang score ≥5
  - b. International Restless Legs Scale score ≥16
  - c. Epworth Sleepiness Scale score >15 (Scores of 11-15 require excessive daytime sleepiness to be recorded in subject's Medical History) (revised per Amendments 01 and 02)
- 2. Reports symptoms potentially related to narcolepsy, that in the clinical opinion of the investigator indicates the need for referral for a diagnostic evaluation for the presence of narcolepsy
- 3. On the MUPS, endorsed the item that corresponds to a history of sleep-eating or reports a history of sleep-related violent behavior, sleep-driving, or symptoms of another parasomnia that in the investigator's opinion make the subject unsuitable for the study (revised per Amendment 02)
- 4. Apnea-Hypopnea Index > 15 or Periodic Limb Movement with Arousal Index > 15 as measured on the PSG at the second screening visit
- 5. Beck Depression Inventory II (BDI-II) score >19 at Screening
- 6. Beck Anxiety Index (BAI) score >15 at Screening
- 7. Habitually naps during the day more than 3 times per week
- 8. Is a female of childbearing potential
  - Note: All females will be considered to be of childbearing potential unless they are postmenopausal (defined as amenorrheic for at least 12 consecutive months, and are postmenopausal without other known or suspected cause), or have been sterilized surgically (ie, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing).
- 9. Excessive caffeine use that in the opinion of the investigator contributes to the subject's insomnia, or habitually consumes caffeine-containing beverages after 18:00 and is unwilling to forego caffeine after 18:00 for the duration of his/her participation in the study
- 10. History of drug or alcohol dependency or abuse within approximately the previous 2 years
- 11. Reports habitually consuming more than 14 drinks containing alcohol per week (females) or more than

Eisai  FINAL: (v7.0), 05 Feb 2018

- 21 drinks containing alcohol per week (males), or unwilling to limit alcohol intake to no more than 2 drinks per day or forego having alcohol within the 3 hours before bedtime for the duration of his/her participation in the study
- 12. Known to be positive for human immunodeficiency virus
- 13. Active viral hepatitis (B or C) as demonstrated by positive serology at Screening
- 14. A prolonged OT/OTcF interval (OTcF >450 ms) as demonstrated by a repeated ECG at Screening (repeated only if initial ECG indicates a OTcF interval >450 ms)
- 15. Current evidence of clinically significant disease (eg, cardiac; respiratory including chronic obstructive pulmonary disease, acute and/or severe respiratory depression; gastrointestinal; severe hepatic impairment; renal including severe renal impairment; neurological including myasthenia gravis; psychiatric disease; or malignancy within the past 5 years other than adequately treated basal cell carcinoma) or chronic pain that in the opinion of the investigator(s) could affect the subject's safety or interfere with the study assessments. including the ability to perform tasks on the cognitive PAB. Subjects for whom a sedating drug would be contraindicated for safety reasons because of the subject's occupation or activities are also excluded. (revised per Amendment 01)
- 16. Comorbid nocturia resulting in frequent need to get out of bed to use the bathroom during the night
- 17. Any history of a medical or psychiatric condition that in the opinion of the investigator(s) could affect the subject's safety or interfere with the study assessments, including the ability to perform the PAB.
- 18. Any suicidal ideation with intent with or without a plan, at the time of or within 6 months before the eC-SSRS administration during the Prerandomization Phase (ie, answering "Yes" to questions 4 or 5 on the Suicidal Ideation section of the eC-SSRS)
- 19. Any suicidal behavior in the past 10 years (per the Suicidal Behavior section of the eC-SSRS) (revised per Amendment 02)
- 20. Scheduled for surgery during the study
- 21. Used any prohibited prescription or over-the-counter concomitant medications within 1 week or 5 halflives, whichever is longer, before the first dose of study medication (Run-in Period). (A list of prohibited concomitant medications is presented in Appendix 3 of the protocol) (revised per Amendment 01)
- 22. Used any modality of treatment for insomnia, including cognitive behavioral therapy or marijuana within 1 week or 5 half-lives, whichever is longer, before the first dose of study medication (Run-in Period) (revised per Amendment 01)
- 23. Failed treatment with suvorexant (Belsomra®) (efficacy and/or safety) following treatment with an appropriate dose and of adequate duration in the opinion of the investigator
- 24. Transmeridian travel across more than 3 time zones in the 2 weeks before Screening, or between Screening and Baseline, or plans to travel across more than 3 time zones during the study
- 25. A positive drug test at Screening, Run-In, or Baseline, or unwilling to refrain from use of recreational drugs during the study
- 26. Hypersensitivity to lemborexant or zolpidem or to their excipients
- 27. Currently enrolled in another clinical trial or used any investigational drug or device within 30 days or 5× the half-life, whichever is longer preceding informed consent
- 28. Previously participated in any clinical trial of lemborexant

## Study Treatment(s)

#### Test drug

Lemborexant 5 mg or 10 mg, or lemborexant-matched placebo taken orally in tablet form each night for 30 consecutive nights immediately before the time the subject intends to try to sleep

### Comparator drug

Zolpidem tartrate extended release 6.25 mg or zolpidem-matched placebo taken orally in tablet form each night for 30 consecutive nights immediately before the time the subject intends to try to sleep

Run-in Period

Eisai  FINAL: (v7.0), 05 Feb 2018

All subjects will receive 1 lemborexant-matched placebo tablet and 1 zolpidem-matched PBO tablet in a single-blind manner during the Run-in Period

## **Treatment Period**

During the Treatment Period, all subjects will receive 2 tablets as described below according to the treatment arm to which the subject has been randomized:

LEM5: 1 zolpidem-matched placebo tablet and 1 lemborexant 5 mg tablet

LEM10: 1 zolpidem-matched placebo tablet and 1 lemborexant 10 mg tablet

ZOL: 1 zolpidem 6.25 mg tablet and 1 lemborexant-matched placebo tablet

PBO: 1 zolpidem-matched placebo tablet and 1 lemborexant-matched placebo tablet

#### **Duration of Treatment**

A maximum of approximately 7.5 weeks: Up to 17 days of PBO during the Run-in Period and up to 35 days of randomized treatment

## Concomitant Drug/Therapy

Caffeine will be permitted in limited quantities during the study. Subjects will be advised to limit caffeine consumption to  $\leq 4$  cups of caffeinated beverages per day, or  $\leq 400$  mg caffeine per day. They will be instructed to avoid caffeine after 13:00 on days when they are scheduled for a PSG recording and after 18:00 on all other days during the study.

Alcohol will be permitted in limited quantities during the study. Subjects may consume a maximum of 2 alcoholic drinks on any day during the study, but will be instructed not to consume any alcohol within 3 hours before bedtime. They must not consume any alcohol on days when they are scheduled for a PSG recording. Compliance with these restrictions will be monitored by specific questions on the Sleep Diary.

Prohibited medications include strong and moderate CYP3A inhibitors and all CYP3A inducers. Prohibited therapies also include any treatment for insomnia disorder, including any drugs or non-pharmacological treatment such as cognitive behavioral therapy; medications that are used for the purpose of inducing sleep (hypnotics) or inducing wakefulness (stimulants; except caffeine; see above) and medications that have known sedating effects or alerting effects. The prohibition applies even if the entire class to which that medication belongs is not prohibited (eg, anticonvulsants).

If a medication is not on the list of prohibited medications but in the opinion of the investigator causes or exacerbates the subject's insomnia, it must not be used throughout the study. If a medication is not specified as prohibited but is in the same class as a medication that is listed in Appendix 3 of the protocol, and if the investigator is uncertain whether the medication has known sedating or alerting effects, the Medical Monitor must be consulted.

If a subject starts any prohibited medication or therapy during the study, he/she must discontinue from the study, with the exception that certain prohibited medications may be used for a short duration (not to exceed 2 weeks) to treat an acute condition if this is agreed with the Medical Monitor. Note that strong CYP3A inhibitors will not be permitted at any time for any duration during the study. (revised per Amendment 01)

#### Assessments

## Screening Assessments (administered only at first screening visit)

Sleep Disorders Screening Battery

The SDSB will include the:

- StopBANG: a list of eight questions to be answered Yes or No, which screens subjects for obstructive sleep apnea
- IRLS: a subjective scale comprising ten questions, which measures severity of symptoms of restless legs syndrome
- ESS: a questionnaire that asks the subject to rate their probability of falling asleep, on a scale of increasing probability from 0 to 3 for eight different situations that most people engage in during their daily lives, which assesses the severity of daytime sleepiness
- MUPS (adapted version): a scale comprising 21 questions asking whether the subject has experienced

phenomena related to the International Classification of Sleep Disorders Version 2 classified parasomnias (eg, enuresis, sleepwalking, sleep paralysis) along with a time frame for occurrence of these experiences ranging from within past month to lifetime and frequency within the time frame ranging from occasionally to almost every night. (revised per Amendment 01)

## Beck Depression Inventory – II

The BDI-II is a 21-question multiple-choice self-report questionnaire that subjects will use to rate the presence, frequency, and severity of symptoms of depression using a 4-point Likert scale. Scores on the BDI-II may range from 0 to 63, with higher scores indicating higher levels of depressive symptoms. Subjects with BDI-II scores greater than 19 will be excluded from participation.

## **Beck Anxiety Inventory**

The BAI is a 21-question multiple-choice self-report inventory that subjects will use to rate the presence, frequency, and severity of symptoms of anxiety using a 4-point Likert scale. Scores on the BAI may range from 0 to 63, with higher scores indicating higher levels of anxiety symptoms. Subjects with scores on the BAI greater than 15 will be excluded from participation.

#### **Efficacy Assessments**

## Polysomnography (PSG)

Each PSG recording will include an electrode montage with electroencephalography (EEG), electromyography (EMG), electrooculography, and ECG channels, for scoring of sleep parameters and sleep architecture via standard sleep scoring criteria. In addition, the first PSG will include channels for assessment of symptoms of sleep apnea and periodic limb movement disorder.

Trained PSG scorers will score PSG records in 30-second epochs according to standard criteria. The PSG at the second screening visit will be used only to calculate the Apnea-Hypopnea Index and the Periodic Limb Movements with Arousal Index for evaluation of eligibility criteria; sleep parameters and sleep architecture will not be evaluated from this PSG. The 2 PSGs obtained during the Run-in Period will be used to a) determine eligibility and b) derive baseline PSG parameters for those subjects who are randomized.

All PSG parameters will be obtained separately for each PSG recording and averaged across the pairs of consecutive PSG nights.

The following parameters will be derived from all PSGs:

- LPS: minutes from lights off to the first epoch of 20 consecutive epochs of non-wakefulness
- SE: proportion of time spent asleep per time in bed (TIB), calculated as TST/interval from lights off until lights on
- WASO: minutes of wake from the onset of persistent sleep until lights on
- WASO2H: minutes of wake during the interval from 240 minutes after lights off until lights on
- TST: minutes of sleep from sleep onset until terminal awakening
- Mean duration of long awakenings (DurLongAw): average duration of all long awakenings (with long awakening defined as 10 or more consecutive epochs [ie, 5 minutes or longer] scored as wake or N1, initiated with at least one epoch of wake, after onset of persistent sleep, and including any terminal awakening)

Additional sleep architecture parameters will also be calculated from each PSG, including:

- Sleep onset latency: minutes from lights off to the first epoch of any stage of sleep (N1, N2, N3, REM) (revised per Amendment 01)
- Number of awakenings after persistent sleep, with an awakening defined as at least 2 consecutive epochs of wakefulness; an awakening cannot be interrupted by stage N1, but must be interrupted by stage N2, N3, or REM
- Number of long awakenings
- WASO1H (wake after sleep onset in the first half of the night): minutes of wake during the interval from onset of persistent sleep until 240 minutes after lights off (revised per Amendment 03)
- Percentage of sleep stages per TIB: wake, non-REM (NREM) sleep (stages N1, N2, N3 separately and

## combined), REM sleep

- Minutes of sleep stages per TIB: wake, NREM sleep (stages N1, N2, N3), REM sleep
- Percentage of sleep stages per TST: wake, NREM sleep (stages N1, N2, N3 separately and combined), REM sleep
- Minutes of sleep stages per TST: wake, NREM sleep (stages N1, N2, N3), REM sleep
- REM episode frequency and duration
- Mean REM/NREM cycle duration
- REM latency: minutes from first epoch of sleep (N1, N2, N3) to first epoch of REM (revised per Amendment 01)

Each of these PSG-derived variables, with the exceptions of SE, REM episode frequency and duration, mean REM/NREM cycle duration, and REM latency, will also be calculated by hour and half of the 8-hour TIB.

## Electronic Sleep Diary

The Sleep Diary will be completed within an hour of morning waketime on each morning of the study from Screening through the end of the study. Sleep Diary entries may be maintained in paper format as a backup to the electronic Sleep Diary, if necessary. This Sleep Diary will yield several self-reported measures of sleep that will be used to determine eligibility, as well as to assess efficacy and safety. In addition, the Sleep Diary will include questions that relate to morning sleepiness and to alcohol consumption. (revised per Amendment 02)

#### Sleep parameters:

- Subjective Sleep Onset Latency (sSOL): estimated minutes from the time that the subject attempts to sleep until sleep onset
- Subjective Wake After Sleep Onset (sWASO): sum of estimated minutes of wake during the night after initial sleep onset until the time that the subject stopped trying to sleep for the night
- Subjective Total Sleep Time (sTST): derived minutes of sleep from sleep onset until the time the subject stopped trying to sleep for the night
- Subjective Sleep Efficiency (sSE): proportion of sTST per subjective time spent in bed, calculated as the interval from the time the subject reported attempting to sleep until the time the subject stopped trying to sleep for the night, and time spent asleep derived from subjective time spent in bed minus sWASO

#### *Quality of Sleep:*

The Sleep Diary will also be used to assess the subject's perception of the quality of sleep on the previous night with the following question, "How would you rate the quality of your sleep last night?" Subjects will rate the quality of their sleep on a scale from 1 to 9 with 1 being extremely poor and 9 being extremely good.

#### Morning Sleepiness:

The Sleep Diary will also be used to assess subjective ratings of morning sleepiness with the following question: "How sleepy/alert do you feel this morning?" Subjects will rate their sleepiness/alertness level on a scale from 1 to 9, with 1 being extremely sleepy, and 9 being extremely alert.

The morning sleepiness question that is part of the electronic Sleep Diary will also be asked verbatim, using a paper-and-pencil format, at 1.5 hours after waketime each morning the subject is in the clinic following a PSG recording. The rating on this question will be taken into consideration by the investigator when making the determination about whether it is safe for the subject to be discharged from the clinic.

#### Alcohol Consumption:

The Sleep Diary will include questions to ask whether the subject consumed alcohol the previous day within 3 hours before bedtime, or exceeded the daily maximum of 2 alcoholic drinks, or both. (revised per Amendment 01)

### Insomnia Severity Index

The ISI is a 7-item self-report questionnaire assessing the nature, severity and impact of insomnia. The dimensions evaluated are severity of sleep onset, sleep maintenance, early-morning awakening problems; sleep dissatisfaction; interference of sleep difficulties with daytime functioning, noticeability of the sleep problems by others; and distress caused by the sleep difficulties. A 5-point Likert scale is used to rate each item (from 0 = no problem to 4 = very severe problem, yielding a total score from 0 to 28.

Confidential Eisai  FINAL: (v7.0), 05 Feb 2018

#### Fatigue Severity Scale

The FSS is a self-report scale on which subjects are instructed to choose a number from 1 to 7 that indicates their degree of agreement with each of 9 statements about their fatigue where "1" indicates strongly disagree and "7", strongly agree. The FSS score is the sum of all responses to the 9 questions. Higher scores indicate greater fatigue.

#### **Pharmacokinetic Assessments**

A single blood sample for plasma concentrations of lemborexant and its metabolites M4, M9 and M10 or zolpidem will be taken at predefined visits. The time and date of the 2 most recent doses before each sample will be documented.

## Pharmacodynamic Assessments

#### Postural Stability using the CDR Posture Assessment

Postural stability will be assessed using an apparatus similar to the Wright ataxiameter, and referred to as the CDR posture device. The CDR posture device measures directional trunk movements (ie, body sway) through a cord placed around the subject's waist and connected to the ataxiameter. On the evening of the Screening PSG visit, subjects will be introduced to the CDR posture assessment. Subjects will stand on a firm surface with feet comfortably apart, either barefoot or wearing socks. The standing position (inside heel-to-inside heel distance) and barefoot/socks conditions will be documented to ensure they remain the same for a given subject at each postural stability assessment timepoint. They will be instructed to stand as still as possible with eyes closed for 1 minute. (revised per Amendment 01) On the morning after the Screening PSG, subjects will complete a CDR posture assessment session for familiarization purposes only; no data from this session will be used for analyses. This session must be conducted under the same conditions (eg, starting within 5 minutes of morning waketime, at bedside) as during the testing sessions at subsequent visits.

Body sway is detected through the cable around the subject's waist by the ataxiameter and these data are transmitted to a laptop. Body sway is measured in units of  $1/3^{\circ}$  of the angle of arc. For ease in reporting these will be called arbitrary units, with a higher number indicating more body sway (less postural stability).

### Cognitive Performance Assessment Battery

A computerized PAB will be administered on a laptop computer after the postural stability test. (revised per Amendment 01) While completing the PAB, subjects will be in bed and ambient lighting will be maintained at a level of 80 – 100 lux at the subject's eye level. On the evening of the Screening PSG visit, before bedtime, subjects will be introduced to the PAB tasks and will undergo a minimum of 2 training sessions. If subjects cannot adequately perform the tasks during the training sessions, they will be excluded from further participation. On the morning after the Screening PSG, subjects will complete a session of the cognitive PAB for familiarization purposes only; no data from this session will be used for analyses. This session must be conducted under the same conditions (eg, lighting, subject in bed) as during the testing sessions at subsequent visits

The PAB comprises 9 tasks including Simple Reaction Time, Choice Reaction Time, Digit Vigilance, Immediate Word Recall, Delayed Word Recall, Numerical Working Memory, Spatial Working Memory, Word Recognition, and Picture Recognition. The full PAB will take approximately 18 to 30 minutes to complete. Four composite domain factor scores are calculated by combining outcome variables from the various tests. The four domain factor scores are Power of Attention, Continuity of Attention, Quality of Memory, and Speed of Memory Retrieval.

- Power of Attention
  - o A composite score from the speed scores of 3 tests of attention
  - Reflects the ability to focus attention and process information
- Continuity of Attention
  - A composite score created by combining the accuracy scores from the tests of attention
  - o Reflects the ability to sustain attention (vigilance)
- Quality of Memory
  - A composite score created by combining the accuracy measures from the two tests of working memory and the four tests of episodic memory

Eisai 

- Reflects the ability to store information in memory and subsequently retrieve it
- Speed of Memory Retrieval
  - A composite score created by combining the reaction time scores from the two working memory tests and the two episodic recognition tests
  - Reflects time taken to retrieve information held in both working and episodic memory

#### **Safety Assessments**

Safety assessments will consist of monitoring and recording all AEs; regular laboratory evaluation for hematology, blood chemistry, and urine values; periodic measurement of vital signs, weight and ECGs; and the performance of physical examinations. Safety will be assessed at every clinic visit throughout the study, and at the EOS Visit.

## Columbia - Suicidality Severity Rating Scale

Suicidality will be assessed using a self-rated electronic version of the C-SSRS (eC-SSRS). The eC-SSRS assesses an individual's degree of suicidality, including both suicidal ideation and suicidal behavior.

## Tyrer Benzodiazepine Withdrawal Symptom Questionnaire

An assessment of withdrawal symptoms will be made using the T-BWSQ completed at the EOS Visit. Subjects will be asked about the presence/absence and severity of the symptoms listed in the questionnaire. For each listed symptom, the subject is to respond "No" (Score = 0), "Yes -moderate" (Score = 1) or "Yes - severe" (Score = 2). The sum of responses will be the subject's score. (revised per Amendment 02)

#### **Other Assessments**

#### EO-5D-3L

The EO-5D-3L is a generic instrument that can be used in the clinical and economic evaluation of health care. and to collect data on quality of life and preferences/utility. The instrument comprises questions on mobility, self-care, usual activities, pain/discomfort and anxiety/depression, and a visual analogue scale from 0 ("Worst imaginable health state") to 100 ("Best imaginable health state").

## Patient Global Impression – Insomnia

The PGI-Insomnia is a self-report assessment asking about subjects' perceptions of the effects of the study medication on their sleep relative to their sleep before entering in the study. As such, the PGI-Insomnia does not have a baseline and the outcome is not change from baseline, but rather the global impression of the study medication's effects at the end of treatment. The PGI-Insomnia has 3 items related to study medication effects (a) helped/worsened sleep, (b) decreased/increased time to fall asleep, (c) increased/decreased total sleep time, and 1 item related to perceived appropriateness of study medication strength. The first 3 items are answered on a 3-point scale (1=positive medication effect, 2=neutral medication effect, 3=negative medication effect) and the last item on a different 3-point scale (medication: 1=too strong, 2=just right, 3=too weak).

#### **Bioanalytical Methods**

Plasma concentrations of lemborexant and its metabolites (M4, M9, and M10) and zolpidem (as needed), will be measured using validated liquid chromatography-tandem mass spectrometry assay methods.

#### Statistical Methods

All statistical tests will be based on the 5% level of significance (2-sided).

## **Study Endpoints**

## **Primary Endpoint(s)**

The primary endpoint is:

Change from baseline of mean LPS on Days 29 and 30 of LEM10 and LEM5 compared to PBO (revised per Amendment 03)

## Secondary Endpoint(s)

#### **Key Secondary Endpoints: US ONLY (revised per Amendment 03)**

- Change from baseline of mean SE on Days 29 and 30 of LEM10 and LEM5 compared to PBO
- Change from baseline of mean WASO on Days 29 and 30 of LEM10 and LEM5 compared to PBO (revised per Amendment 04)

Eisai  Change from baseline of mean WASO2H on Days 29 and 30 of LEM10 and LEM5 compared to ZOL

#### **Key Secondary Endpoint(s): Non-US ONLY (revised per Amendment 03)**

- Change from baseline of mean SE on Days 29 and 30 of LEM10 and LEM5 compared to PBO
- Change from baseline of mean WASO on Days 29 and 30 of LEM10 and LEM5 compared to PBO

## Additional Secondary Endpoints: US and Non-US (revised per Amendment 03)

- Change from baseline on the postural stability test of mean units of body sway on Days 2 and 3 of LEM5 and LEM10 compared to ZOL
- Change from baseline of mean LPS, WASO, and TST on Days 1 and 2 and Days 29 and 30 of LEM5 and LEM10 compared to ZOL
- Change from baseline mean of subjective Sleep Diary variables including sSOL, sWASO, sSE and sTST over the first 7 and last 7 nights of the Treatment Period of LEM5 and LEM10 compared to ZOL
- Change from baseline of mean LPS, SE, WASO, WASO2H, and TST on Days 1 and 2 of LEM5 and LEM10 compared to PBO
- Change from baseline of mean WASO2H and TST on Days 29 and 30 of LEM5 and LEM10 compared to PBO
- Change from baseline mean of subjective Sleep Diary variables including sSOL, sWASO, sSE and sTST over the first 7 and last 7 nights of the Treatment Period of LEM5 and LEM10 compared to PBO
- Proportion of responders after Days 1 and 2 and Days 29 and 30 (PSG), and over the first 7 nights and last 7 nights of treatment (Sleep Diary), to LEM5 and LEM10 compared to ZOL and PBO, such that:
  - Objective sleep onset response is defined as LPS ≤ 20 minutes (provided mean baseline LPS was > 30 minutes)
  - Subjective sleep onset response is defined as  $sSOL \le 20$  minutes (provided mean baseline sSOL was > 30 minutes)
  - Objective sleep maintenance response is defined as WASO ≤ 60 minutes (provided mean baseline WASO was > 60 minutes and is reduced by > 10 minutes compared to baseline)
  - Subjective sleep maintenance response is defined as  $sWASO \le 60$  minutes (provided mean WASO was > 60 minutes and is reduced by > 10 minutes compared to baseline)
- Safety and tolerability of LEM
- Change from baseline of the score from items 4 to 7 on the ISI at Day 31 of LEM5 and LEM10 compared to ZOL and PBO
- Change from baseline on the FSS score at Day 31 of LEM5 and LEM10 compared to ZOL and PBO
- Change from baseline of mean power of attention, mean continuity of attention, mean quality of memory, and mean speed of memory retrieval on Days 2 and 3

## **Exploratory Endpoints**

The change from baseline of WASO2H for LEM5 and LEM10 compared to ZOL will be considered as exploratory for all non-US submissions. The following endpoints will also be explored for LEM5 and LEM10. Except for PK endpoints, comparisons to ZOL and PBO will be made. (revised per Amendment 03)

- Change from baseline of the mean rating on the Quality of Sleep question from the Sleep Diary of the first 7 days and last 7 days of the Treatment Period
- Change from baseline of mean power of attention, mean continuity of attention, mean quality of memory, and mean speed of memory retrieval on Days 30 and 31
- From the postural stability test, change from baseline of mean units of body sway after the first 2 nights of the Treatment Period compared to PBO and the last 2 nights of the Treatment Period compared to ZOL and PBO
- Rebound insomnia endpoints as assessed from the Sleep Diary during the Follow-up Period
  - O Change from baseline of sSOL at the following timepoints during the Follow-up Period: each of the first 3 nights, mean of the first 3 nights, mean of the first 7 nights, mean of the second 7 nights(revised per Amendment 03)

Eisai 

- Change from baseline of sWASO at the following timepoints during the Follow-up Period: each of the first 3 nights, mean of the first 3 nights, mean of the first 7, mean of the second 7 nights (revised per Amendment 03)
- Proportion of subjects whose sSOL is longer than at Screening at the following timepintgs during the the Follow-up Period: each of the first 3 nights, mean of the first 3 nights, mean for first 7 nights, mean of the second 7 nights (revised per Amendments 02 and 03)
- Proportion of subjects whose sWASO is higher than at Screening at the following timepoints during the Follow-up Period: each of the first 3 nights, mean of the first 3 nights, mean for the first 7 nights, for the second 7 nights (revised per Amendments 02 and 03)
- Mean rating on the morning sleepiness item of the Sleep Diary on the first 7 mornings and last 7 mornings of the Treatment Period
- Mean rating on the morning sleepiness item of the Sleep Diary on the first 7 mornings and second 7 mornings of the Follow-up Period
- Change from baseline of mean morning sleepiness ratings assessed at 1.5 hours after waketime when subjects are in clinic on Days 1 and 2, and Days 29 and 30 (revised per Amendment 01)
- Change from baseline of mean minutes and mean percentage (a) per TIB and (b) per TST of sleep stage N1, N2, N3 (separately and combined) and REM on Days 1 and 2 and Days 29 and 30
- Change from baseline of mean REM latency, mean number of awakenings, and mean number of long awakenings on Days 1 and 2 and Days 29 and 30 (revised per Amendment 03)
- Number and percentage of subjects with a rating of a positive medication effect on each PGI-Insomnia item at Day 31
- Change from baseline on the EQ-5D-3L at Day 31
- Mean score on the T-BWSO of LEM5 and LEM10 compared to ZOL and PBO at end of study
- Proportion of subjects who score ≥ 3 on the T-BWSQ of LEM5 and LEM10 compared to ZOL and PBO at end of study
- PK of lemborexant and its metabolites M4, M9, and M10
- Relationships between lemborexant PK, efficacy, and/or safety variables using PK/PD modeling

### **Analysis Sets**

The Safety Analysis Set is the group of randomized subjects who received at least 1 dose of randomized study drug and had at least 1 postdose safety assessment.

The Full Analysis Set (FAS) is the group of randomized subjects who received at least 1 dose of randomized study drug and had at least 1 postdose primary efficacy measurement.

The Per Protocol (PP) Analysis Set is the group of subjects who sufficiently complied with the protocol. Details of the evaluability criteria will be determined before database lock and treatment unblinding and will be specified in the Statistical Analysis Plan (SAP).

The PK Analysis Set is the group of subjects who have at least one quantifiable plasma concentration of lemborexant or its metabolites, or zolpidem, with adequately documented dosing history.

The PK/PD Analysis Set is the group of subjects receiving either lemborexant or placebo who have efficacy or safety data with documented dosing history. In addition, subjects receiving lemborexant should have at least one quantifiable lemborexant concentration data point as per the PK Analysis Set.

### **Efficacy Analyses**

#### **Definitions of Baseline**

Baseline is defined as the means from the 2 PSGs during the Run-in Period for PSG-derived variables and the mean of the last 7 mornings before the first baseline PSG during the Run-in Period for Sleep Diary variables. For other endpoints, baseline data are captured during the Run-in Period and Baseline Period. Details will be specified in the SAP.

## **Control of Type I Error (revised per Amendment 03)**

A sequential gate-keeping procedure will be used for the primary and the key secondary endpoint comparisons to control for the overall type I error at the 0.05 significance level. The first endpoint comparison will be tested

Confidential Eisai  at the 0.05 significance level. If the testing is found to be statistically significant, then proceed to the next endpoint testing at significance level of 0.05, otherwise stop testing.

The primary endpoints will be tested in the following order:

- Change from baseline of the mean LPS of Days 29 and 30 of LEM10 compared to PBO
- Change from baseline of the mean LPS of Days 29 and 30 of LEM5 compared to PBO

The key secondary endpoints will only be tested if both primary analyses are statistically significant at the 0.05 level. The key secondary endpoints will be tested in the following order:

#### US Only

- Change from baseline of the mean SE of Days 29 and 30 of LEM10 compared to PBO
- Change from baseline of the mean SE of Days 29 and 30 of LEM5 compared to PBO
- Change from baseline of the mean WASO of Days 29 and 30 of LEM10 compared to PBO (revised per Amendment 04)
- Change from baseline of the mean WASO2H of Days 29 and 30 of LEM10 compared to ZOL
- Change from baseline of the mean WASO on Days 29 and 30 of LEM5 compared to PBO (revised per Amendment 04)
- Change from baseline of the mean WASO2H on Days 29 and 30 of LEM5 compared to ZOL

#### Non-US Only

- Change from baseline of the mean SE of Days 29 and 30 of LEM10 compared to PBO
- Change from baseline of the mean SE of Days 29 and 30 of LEM5 compared to PBO
- Change from baseline of the mean WASO of Days 29 and 30 of LEM10 compared to PBO
- Change from baseline of the mean WASO on Days 29 and 30 of LEM5 compared to PBO

No multiplicity adjustment will be done on other efficacy analyses.

#### **Analysis for the Primary Endpoint**

<u>Null Hypothesis</u>: No difference exists in the mean change from baseline of the mean LPS of Days 29 and 30 for treatment with LEM10 (or LEM5) as compared with PBO. (revised per Amendment 03)

<u>Alternative Hypothesis</u>: A difference exists in the mean change from baseline of the mean LPS of Days 29 and 30 for LEM10 (or LEM5) compared to PBO. (revised per Amendment 03)

The LPS change from baseline (the mean of Days 1 and 2, and the mean of Days 29 and 30) will be analyzed using the mixed effect model repeated measurement analysis (MMRM) on the FAS. The model will include all data and will be adjusted for the corresponding baseline value (the means from the 2 PSG recordings during the Run-in Period), region, age group (55 – <65 years; 65 years or older), treatment, time (Days 1/2, and Days 29/30), and the interaction of treatment by time (revised per Amendment 04). Since LPS is known to be non-normally distributed, a log-transformation will be used in the analysis. An unstructured covariance matrix will be used, and if the model fails to converge, then an autoregressive matrix will be used. The missing values will be imputed using a pattern mixture model utilizing multiple imputations (MI) assuming the missing values are missing not at random (MNAR) utilizing the complete case missing value pattern (CCMV - subjects who completed primary efficacy assessments without missing values) (revised per Amendment 04). The missing values for a given visit will be imputed using all available values including the retrieved measurement from the post-discontinuation data. The treatment comparison will be performed using contrasts. The p-value, least square (LS) means and the 95% confidence interval (CI) for the treatment difference will also be provided. (revised per Amendment 03)

Subgroup analyses and additional sensitivity analysis will be performed as appropriate.

The following analyses will be considered as sensitivity analyses:

- PP analysis: The same primary efficacy analyses described above will be repeated based on PP analysis set.
- Completer analysis: The same primary efficacy analyses described above will be repeated on subjects who completed all efficacy assessments and have no missing values.
- As-treated analysis: The same primary efficacy analyses (MMRM analysis with MI for missing value imputation) will be repeated based on the actual treatment the subject received regardless of randomization.

Eisai 

- MMRM analysis assuming missing at random (MAR): The same primary endpoint analysis described above will be analyzed using MMRM assuming the missing values are MAR.
- MI Imputation assuming MNAR utilizing CCMV-4: The same MMRM method used in the primary analysis will be applied utilizing CCMV-4 (ie, up to 4 monotone missing patterns will be used for missing value imputation as follows): (revised per Amendment 04)

| Study days where results are available | 1 | 2 | 29 | 30 |
|----------------------------------------|---|---|----|----|
| Pattern 1 | X | X | X | X |
| Pattern 2 | X | X | X | • |
| Pattern 3 | X | X | | • |
| Pattern 4 | x | | | |
| x = result present; . = result missing | • | | | |

Tipping point analysis: A range of shifts will be used in the multiple imputation of missing data assuming MNAR to identify the specific shift and treatment effect that will tip the results from statistically significant to non-significant. (revised per Amendment 04)

## Secondary Efficacy Analyses

### Key Secondary Efficacy Analysis (revised per Amendments 03 and 04)

Changes from baseline of mean SE, WASO2H, and WASO of Days 1 and 2 and the mean of Days 29 and 30 will be analyzed using a pattern mixture model utilizing MI assuming MNAR. The treatment comparison will be performed using contrasts. The p-value, LS means and the 95% CI of the treatment differences will also be provided. The comparison of LEM10 and LEM5 to ZOL on WASO2H will be considered as exploratory for all non-US submissions. (revised per Amendment 03)

#### Other Secondary Efficacy Analyses (revised per Amendment 03)

The other secondary efficacy endpoints (change from baseline of the mean of the following endpoints: LPS, SE, WASO2H, and WASO of the mean of Days 1 and 2; TST of the mean of Days 1 and 2 and of the mean of Days 29 and 30; sSOL, sWASO, sSE, and sTST for the mean of the first 7 and last 7 days of the Treatment Period) will be analyzed using MMRM assuming MAR. (revised per Amendment 03)

The proportion of responders will be analyzed using the Cochran-Mantel-Haenszel test, controlled for region and age group, for each dose of lemborexant compared to PBO and ZOL. The analysis will be similarly repeated for responder analysis based on Sleep Diary variables (sSOL and sWASO) over the first 7 and last 7 nights of treatment. (revised per Amendment 03)

The change from baseline of the ISI total of four items on daytime functioning at Day 31 and the FSS score at Day 31 will be analyzed using analysis of covariance (ANCOVA), adjusted for the corresponding baseline value, age group, region, and treatment. (revised per Amendment 03)

Changes from baseline in mean power of attention, mean continuity of attention, mean quality of memory, and mean speed of memory retrieval for the PAB tasks will be analyzed using MMRM assuming MAR. (revised per Amendments 01 and 03)

Secondary endpoints may also be presented graphically or analyzed by modeling methods if warranted. (revised per Amendment 03)

No multiplicity adjustment or missing values imputation is planned for other secondary analyses. (revised per Amendment 03)

## **Exploratory and Pharmacodynamic Analyses**

The change from baseline mean score of the quality of sleep item on the Sleep Diary for the means of the first 7 days and last 7 days of the Treatment Period will be analyzed using MMRM assuming MAR. (revised per Amendment 03)

Rebound insomnia is defined as worsened sleep relative to Screening after study drug treatment is completed. Sleep Diary data from the Follow-up Period will be compared to Sleep Diary data from the Screening Period to assess whether subjects experience rebound insomnia. Specifically, a higher value for sSOL or sWASO during

Confidential Eisai  the Follow-up Period compared to the mean sSOL or sWASO value during the Screening Period will be considered worsened sleep. (revised per Amendment 02)

To assess rebound insomnia, both categorical analysis at the subject level and continuous analysis at the group mean level will be performed. For each of the first 3 nights, the mean of the first 3 nights, and the mean of each of the 2 weeks of the Follow-up Period the proportion of subjects whose corresponding value for sSOL or sWASO exceeds the corresponding Screening Period value by 5 minutes will be summarized by treatment group and compared to placebo. The percentage of 'rebounders' between each treatment and placebo group will be analyzed using a CMH test. (revised per Amendments 01, 02, and 03)

To assess statistical significance using the continuous data at the group mean level, the data will be analyzed using ANCOVA, adjusted for region, age group and treatment. The LS mean of each of the first 3 nights and each week of the Follow-up Period will be compared to the Screening Period between each treatment group and placebo. If the lower bound of the 95% CI of sSOL or sWASO for each of the first 3 nights and the mean of each week of the Follow-Up Period exceeds the upper bound of a 95% CI for the values during the Screening Period in the given treatment group, it will be considered strong evidence for rebound insomnia. If the LS means for sSOL and sWASO for the Follow-up Period are all lower than for the Screening Period, then no rebound insomnia is suggested. (revised per Amendments 01 and 03)

To evaluate morning residual sleepiness during study treatment and following completion of treatment, the change from baseline of the mean of morning sleepiness item on the Sleep Diary for the first 7 mornings of the Treatment Period, the last 7 mornings of the Treatment Period, as well as the means of the first 7 days and second 7 days of the Follow-up Period will be analyzed using MMRM assuming MAR. Change from baseline of the mean morning sleepiness ratings assessed at 1.5 hours after waketime when subjects are in clinic on days 1 and 2 and days 29 and 30 will be similarly analyzed using MMRM assuming MAR. (revised per Amendments 01 and 03)

The change from baseline of the mean of Days 1 and 2 and of the mean of Days 29 and 30 for the sleep architecture and other PSG endpoints (WASO1H minutes and percentage [a] per TIB and [b] per TST of sleep stage N1, N2, N3, total NREM and REM; REM latency, DurLongAW, number of awakenings, number of long awakenings, REM episode frequency and duration, and mean REM/NREM cycle duration) will be summarized. (revised per Amendment 03)

Each item on the PGI-Insomnia at Day 31 will be analyzed separately by calculating the number and percentages of subjects for each response category (eg, negative [3], neutral [2], positive [1] medication effect). The percentage of positive responses will be compared between treatment groups using the chi-square test, and repeated for age subgroups.

The change from baseline in the EQ-5D-3L score at Day 31 will be analyzed using ANCOVA, adjusted for region, age group and treatment. (revised per Amendment 03)

No multiplicity adjustment or missing value imputation is planned for exploratory and pharmocodynamic analyses. (revised per Amendment 03)

#### Pharmacokinetic Analysis

The Safety Analysis Set will be used for individual lemborexant and its metabolites M4, M9, and M10, as well as zolpidem plasma concentration listings. The PK Analysis Set will be used for summaries of lemborexant and its metabolites M4, M9, and M10, as well as zolpidem plasma concentrations by dose, time, and day.

A population PK approach will be used to characterize the PK of lemborexant. For this approach, PK analysis data from this study will be pooled with relevant data from Phase 1 and 2 studies, and other Phase 3 studies if available. The effect of covariates (ie, demographics) on the PK of lemborexant will be evaluated. The PK model will be parameterized for apparent total clearance following extravascular administration (CL/F) and volumes of distribution. Derived exposure parameters such as area under the concentration-time curve (AUC), maximum lemborexant plasma concentration ( $C_{max}$ ) and any other relevant parameters will be calculated from the model using the individual posterior estimate of CL/F and dosing history.

#### Pharmacodynamic Analysis

These analyses are described in the Secondary Efficacy Analyses, and Exploratory and Pharmacodynamic Analyses sections (above).

#### Pharmacokinetic/Pharmacodynamic Analysis

The PK/PD relationship between exposure to lemborexant and efficacy variables including but not limited to

Eisai 

LPS and WASO, and safety variables including but not limited to morning sleepiness and frequently occurring treatment-emergent adverse events (TEAEs), will be explored graphically. Any emergent PK/PD relationships will be evaluated by population PK/PD modeling. The population PK/PD analysis plan will be described and results will be reported in a separate document.

Population PK and PK/PD analyses will be performed using NONMEM version 7.2 or later.

## **Safety Analyses**

Evaluations of safety will be performed on the relevant Safety Analysis Set. The incidence of AEs, out-of-normal-range laboratory safety test variables, abnormal ECG findings, out-of-range vital signs and weight, suicidality (eC-SSRS), and T-BWSQ (including frequency and percentage of subjects with T-BWSQ score ≥3), along with change from baseline in laboratory safety test variables, ECGs, and vital sign and weight measurements, will be summarized by treatment group using descriptive statistics.

#### Other Analyses

Secondary and exploratory endpoints may be additionally presented graphically or analyzed by modeling methods if warranted.

Although ZOL is included in the study as an active comparator, comparison of ZOL to PBO, and comparison between LEM10 and LEM5 may be made to facilitate evaluation of study results.

## **Interim Analyses**

An interim analysis is planned to be conducted after approximately 50% of subjects (approximately n=475 subjects) have been randomized and either completed Day 31 assessments or discontinued from the study. This interim analysis will be conducted for administrative reasons as detailed in the separate Interim Analysis charter. When the specified number of subjects has completed the Day 31 assessments, an independent statistician external to the Sponsor will be provided with the relevant PSG dataset and will be unblinded to the primary endpoint, ie, change from baseline in WASO2H for the mean of Days 29 and 30. A conditional power will be calculated to predict the probability that the trial will achieve a significant treatment effect for WASO2H in the LEM10 versus ZOL arms at the end of the study, given what is observed at the time of interim analysis. The interim analysis will be limited to the comparison of LEM10 versus ZOL on the change from baseline in WASO2H for the mean of Days 29 and 30. No other endpoints, dose groups, or timepoints will be analyzed at the interim analysis. The study will not be terminated for either futility or efficacy. Therefore no impact to the type I error rate is expected.

The method of calculating the conditional power will be detailed in the Interim Analysis charter, along with operational procedures, unblinding procedures, procedures for communicating the results of the conditional power calculation and recipients of this information. To preclude potential influence on the conduct of the remainder of the study, disclosure of the conditional power will be limited to a prespecified set of executive-level individuals at the sponsor and sponsor's co-development partner. No individuals involved with the conduct of the study will have access to the interim data or the results of the interim analysis (i.e., the conditional power of LEM10 versus ZOL on the change from baseline in WASO2H for the mean of Days 29 and 30).

Enrollment of subjects will not be stopped during the interval during which the interim analysis is conducted. The interim analysis may be waived or otherwise not conducted, for reasons including but not limited to a higher than anticipated enrollment rate which would make the interim analysis unnecessary as the majority of subjects would have been enrolled by the time the interim analysis was concluded.

## Sample Size Rationale

The sample size was estimated for each comparison of LEM10 vs. PBO, and LEM5 vs PBO with respect to the mean change from baseline of LPS at Month 1, on the basis of a 2-sided t-test at the  $0.05~\alpha$ -level for each treatment comparison. (revised per Amendment 03)

On the basis of the dose finding study E2006-G000-201 (Study 201), across various lemborexant doses (1 to 25 mg) at Days 14 and 15, the standard deviation (SD) of change from baseline for log-transformed LPS is assumed to be 0.9. The LS mean treatment difference at Days 14/15 from Study 201 for log-transformed LPS of LEM10 and LEM5 compared with PBO was 0.75 and -1.15, respectively. Therefore, a sample size of 250 subjects for LEM5, 250 subjects for LEM10, and 200 subjects for PBO has at least 95% power for each treatment comparison, LEM10 with PBO, and LEM5 with PBO, based on 2-sided, 2-sample t-test at 5% significance level. (revised per Amendment 03)

Power is also estimated for the key secondary objectives, the comparison of LEM10 and LEM5 to PBO on

change from baseline of SE and WASO, and LEM10 and LEM5 to ZOL on WASO2H. A sample size of 250 subjects each for LEM5, LEM10, and ZOL, and 200 subjects for PBO has at least 95% power for detecting a statistically significant difference between LEM and PBO for change from baseline in SE, at least 80% power for detecting a statistically significant difference between LEM10 and ZOL/PBO for change from baseline in WASO/WASO2H based on 2-sided 2-sample t-test at 5% significance level. (revised per Amendments 03 and 04)

| Endpoint (Test) | Estimated Treatment Difference | Estimated SD | Power |
|---|---|---|---|
| Log(LPS) (LEM5 vs PBO) | -0.75 | 0.9 | >95% |
| Log(LPS) (LEM10 vs PBO) | -1.15 | 0.9 | >95% |
| SE (LEM5 vs PBO) | 5% | 14% | >95% |
| SE (LEM10 vs PBO) | 7% | 14% | >95% |
| WASO (LEM5 vs PBO) | -10 min | 55 min | 48% |
| WASO (LEM10 vs PBO) | -15 min | 55 min | 81% |
| WASO2H (LEM5 vs ZOL) | -8 min | 38 min | 65% |
| WASO2H (LEM10 vs ZOL) | -11 min | 38 min | 89% |

Estimated treatment difference and SD are based on Study 201.

# 3 TABLE OF CONTENTS

| 1 | TITLE PAGE | 1 |
|---|---|---|
| 2 | CLINICAL PROTOCOL SYNOPSIS | 2 |
| 3 | TABLE OF CONTENTS | 21 |
| 4 | LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS | 26 |
| 5 | ETHICS | 29 |
| | 5.1 Institutional Review Boards/Independent Ethics Committees | 29 |
| | 5.2 Ethical Conduct of the Study | 29 |
| | 5.3 Subject Information and Informed Consent | 30 |
| 6 | INVESTIGATORS AND STUDY PERSONNEL | 31 |
| 7 | INTRODUCTION | 32 |
| | 7.1 Indication | 32 |
| | 7.1.1 Current Therapeutic Options | 32 |
| | 7.1.2 Lemborexant (E2006) | 32 |
| | 7.1.2.1 Mechanism of Action | 32 |
| | 7.1.2.2 Clinical Experience with Lemborexant | 32 |
| | 7.1.2.2.1 Phase 1 | 32 |
| | 7.1.2.2.2 Phase 2 | 34 |
| | 7.2 Study Rationale | 34 |
| 8 | STUDY OBJECTIVES | 36 |
| | 8.1 Primary Objective – US and Non-US (revised per Amendment 03) | |
| | 8.2 Secondary Objectives | 36 |
| | 8.2.1 Key Secondary Objectives – US ONLY (revised per Amendment 03) | 36 |
| | 8.2.2 Key Secondary Objectives – Non-US ONLY (revised per Amendment 03) | 36 |
| | 8.2.3 Additional Secondary Objectives – US and Non-US (revised per | |
| | Amendment 03) | 36 |
| | 8.3 Exploratory Objectives – US and Non-US (revised per Amendment 03) | 37 |
| 9 | INVESTIGATIONAL PLAN | 38 |
| | 9.1 Overall Study Design and Plan | 38 |
| | 9.1.1 Prerandomization Phase | 40 |
| | 9.1.1.1 Screening Period | |
| | 9.1.1.2 Run-in Period | 41 |
| | 9.1.1.3 Baseline Period | 42 |
| | 9.1.2 Randomization Phase | 42 |
| | 9.1.2.1 Treatment Period | 42 |
| | 9.1.2.2 Follow-up Period | |
| | 9.2 Discussion of Study Design, Including Choice of Control Groups | 43 |

| 9.2.1 | Randomization | 43 |
|---|---|---|
| 9.2.2 | Run-In | 43 |
| 9.2.3 | Efficacy Assessments | 44 |
| 9.2.4 | Morning Residual Effects on Postural Stability and Cognitive Performance | 44 |
| 9.2.5 | Adjudication Committee (revised per Amendment 02) | |
| 9.2.6 | Study Duration | |
| 9.2.7 | Age Group | |
| 9.2.8 | Time of Dosing | |
| 9.2.9 | Interim Analysis | |
| 9.3 Sel | ection of Study Population | 47 |
| 9.3.1 | Inclusion Criteria | |
| 9.3.2 | Exclusion Criteria | 48 |
| 9.3.3 | Removal of Subjects From Therapy or Assessment | 50 |
| 9.4 Tre | atment(s) | |
| 9.4.1 | Treatment(s) Administered | |
| 9.4.2 | Identity of Investigational Product(s) | 51 |
| 9.4. | 2.1 Chemical Name, Structural Formula of E2006/Lemborexant | 52 |
| 9.4. | 2.2 Comparator Drug | 52 |
| 9.4. | 2.3 Labeling for Study Drug | 52 |
| 9.4. | 2.4 Storage Conditions | 52 |
| 9.4.3 | Method of Assigning Subjects to Treatment Groups | 53 |
| 9.4.4 | Selection of Doses in the Study | 53 |
| 9.4.5 | Selection and Timing of Dose for Each Subject | 54 |
| 9.4.6 | Blinding. | 54 |
| 9.4.7 | Prior and Concomitant Therapy | 54 |
| 9.4. | 7.1 Drug-Drug Interactions | 54 |
| 9.4. | 7.2 Prohibited Concomitant Therapies and Drugs | 54 |
| 9.4.8 | Treatment Compliance | 55 |
| 9.4.9 | Drug Supplies and Accountability | 56 |
| 9.5 Stu | dy Assessments | 57 |
| 9.5.1 | Assessments | 57 |
| 9.5. | 1.1 Demography | 57 |
| 9.5. | 1.2 Baseline Assessments | 58 |
| Ģ | 9.5.1.2.1 Medical History and Physical Examinations | 58 |
| Ģ | 9.5.1.2.2 Sleep Disorders History and Screening Battery | 58 |
| Ģ | 9.5.1.2.3 Beck Depression Inventory - II | 58 |
| | 9.5.1.2.4 Beck Anxiety Inventory | 59 |

| 9.5.1.3 | Efficacy Assessments | 59 |
|---|---|---|
| 9.5.1.3.1 | Polysomnography | 59 |
| 9.5.1.3.2 | 2 Electronic Sleep Diary | 60 |
| 9.5.1.3.3 | 3 Insomnia Severity Index | 61 |
| 9.5.1.3.4 | Fatigue Severity Scale | 62 |
| | Pharmacokinetic, Pharmacodynamic, Pharmacogenomic, and Other Biomarker Assessments | 62 |
| 9.5.1.4.1 | Pharmacokinetic Assessments | 62 |
| 9.5.1.4.2 | Pharmacodynamic Assessments | 62 |
| 9.5.1.4.3 | B Pharmacogenomic Assessments | 63 |
| 9.5.1.4.4 | 4 Other Biomarker Assessments | 63 |
| 9.5.1.5 | Safety Assessments | 64 |
| 9.5.1.5.1 | Columbia-Suicide Severity Rating Scale | 64 |
| 9.5.1.5.2 | 2 Tyrer Benzodiazepine Withdrawal Symptom Questionnaire | 64 |
| 9.5.1.5.3 | 3 Adverse Events | 64 |
| 9.5.1.5.4 | Serious Adverse Events and Events Associated With Special Situations | 66 |
| 9.5.1.5.5 | 5 Laboratory Measurements | 67 |
| 9.5.1.5.0 | Vital Signs and Weight Measurements | 69 |
| 9.5.1.5.7 | 7 Physical Examinations | 69 |
| 9.5.1.5.8 | B Electrocardiograms | 69 |
| 9.5.1.5.9 | Other Assessments | 70 |
| 9.5.2 Sche | dule of Procedures/Assessments | 70 |
| 9.5.2.1 | Schedule of Procedures/Assessments | 70 |
| 9.5.2.2 | Description of Procedures/Assessments Schedule | 75 |
| 9.5.3 Appr | opriateness of Measurements | 75 |
| 9.5.4 Repo | orting of Serious Adverse Events, Pregnancy, and Events ciated with Special Situations | 75 |
| 9.5.4.1 | Reporting of Serious Adverse Events | 75 |
| | Reporting of Pregnancy and Exposure to Study Drug Through Breastfeeding | 76 |
| 9.5.4.3 | Reporting of Events Associated with Special Situations | 77 |
| 9.5.4.4 | Expedited Reporting | 77 |
| 9.5.4.5 | Breaking the Blind | 78 |
| 9.5.4.6 | Regulatory Reporting of Adverse Events | 78 |
| 9.5.5 Com | pletion/Discontinuation of Subjects | 78 |
| 9.5.6 Abus | se or Diversion of Study Drug | 79 |
| 9.5.7 Conf | irmation of Medical Care by Another Physician | 79 |
| Data Quali | ty Assurance | 79 |

9.6

| 9.6.1 Data Collection | 79 |
|---|---|
| 9.6.2 Clinical Data Management | 80 |
| 9.7 Statistical Methods | 80 |
| 9.7.1 Statistical and Analytical Plans | 80 |
| 9.7.1.1 Study Endpoints | 80 |
| 9.7.1.1.1 Primary Endpoint(s) | 80 |
| 9.7.1.1.2 Secondary Endpoint(s) | 80 |
| 9.7.1.1.3 Exploratory Endpoint(s) – US and Non-US (revised per Amendment 03) | 82 |
| 9.7.1.2 Definitions of Analysis Sets | |
| 9.7.1.3 Subject Disposition | |
| 9.7.1.4 Demographic and Other Baseline Characteristics | |
| 9.7.1.5 Prior and Concomitant Therapy | |
| 9.7.1.6 Efficacy Analyses | |
| 9.7.1.6.1 Primary Efficacy Analysis | |
| 9.7.1.6.2 Secondary Efficacy Analyses | |
| 9.7.1.6.3 Exploratory Efficacy and Pharmacodynamic Analyses | 89 |
| 9.7.1.7 Pharmacokinetic, Pharmacodynamic, Pharmacogenomic, and | |
| Other Biomarker Analyses | 90 |
| 9.7.1.7.1 Pharmacokinetic Analyses | |
| 9.7.1.7.2 Pharmacodynamic, Pharmacogenomic, and Other Biomarke Analyses | |
| 9.7.1.8 Safety Analyses | |
| 9.7.1.8.1 Extent of Exposure | 91 |
| 9.7.1.8.2 Adverse Events | 91 |
| 9.7.1.8.3 Clinical Laboratory Values | 92 |
| 9.7.1.8.4 Vital Signs, Height, and Weight | 93 |
| 9.7.1.8.5 Electrocardiograms | 93 |
| 9.7.1.8.6 Other Safety Analyses | 94 |
| 9.7.1.9 Other Analyses | 94 |
| 9.7.2 Determination of Sample Size | 94 |
| 9.7.3 Interim Analysis | 95 |
| 9.7.4 Procedure for Revising the Statistical Analysis Plan | |
| 10 REFERENCE LIST | 97 |
| 11 PROCEDURES AND INSTRUCTIONS (ADMINISTRATIVE PROCEDURES) | 99 |
| 11.1 Changes to the Protocol | 99 |
| 11.2 Adherence to the Protocol | 99 |
| 11.3 Monitoring Procedures | 99 |
| 11.4 Recording of Data | 100 |

| 11.5 Ide | ntification of Source Data | 100 |
|---|---|---|
| 11.6 Ret | ention of Records | 100 |
| 11.7 Au | diting Procedures and Inspection | 101 |
| 11.8 Hai | ndling of Study Drug | 101 |
| 11.9 Pub | olication of Results | 101 |
| 11.10 Dis | closure and Confidentiality | 102 |
| 11.11 Dis | continuation of Study | 102 |
| 11.12 Sub | eject Insurance and Indemnity | 102 |
| 12 APPEND | ICES | 103 |
| LIST OF IN | -TEXT TABLES | |
| Table 1 | Treatment Effect for Lemborexant versus Placebo (Study 201) | 46 |
| Table 2 | Clinical Laboratory Tests | 68 |
| Table 3 | Blood Sampling Schedule for All Laboratory and Pharmacokinetic Assessments | 68 |
| Table 4 | Schedule of Procedures/Assessments in Study E2006-G000-304 | 71 |
| Table 5 | Vital Sign Criteria | 93 |
| Table 6: | Power and Sample Size Calculation for Change from Baseline of LPS, SE, WASO2H, and WASO | |
| LIST OF IN | -TEXT FIGURES | |
| Figure 1 | Schematic Diagram of E2006-G000-304 Study Design | 39 |
| Figure 2 | Flow Chart of Gate Keeping Testing Procedure – Study E2006-G000-304 (revised per Amendment 04) | |
| LIST OF AI | PPENDICES | |
| Appendix | Sponsor's Grading for Laboratory Values | 104 |
| Appendix 2 | | |
| Appendix 3 | | |
# 4 LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

**Abbreviation** Term

AE adverse event

ALT alanine aminotransferase
ANCOVA analysis of covariance

AST aspartate aminotransferase

AUC area under the concentration-time curve

AUC<sub>(0-inf)</sub> area under the concentration-time curve extrapolated from zero time to infinite

time

BAI Beck Anxiety Inventory

BDI-II Beck Depression Inventory - II

BMI body mass index
BP blood pressure

CDR Cognitive Drug Research
CFR Code of Federal Regulations

CI confidence interval CL total clearance

CL/F apparent total clearance following extravascular administration
CPAP continuous positive airway pressure (revised per Amendment 01)

C<sub>max</sub> maximum observed concentration

CPMP Committee for Proprietary Medicinal Products,

CRA clinical research associate

CRF case report form

CRO Contract Research Organization

DORA dual orexin receptor antagonist

EASS events associated with special situations

ECG electrocardiogram

eCRF electronic case report form

eC-SSRS electronic Columbia-Suicide Severity Rating Scale

EEG electroencephalogram
EMG electromyography

EOS end of study

ESS Epworth Sleepiness Scale

ET early termination
EU European Union
FAS Full Analysis Set

| Abbreviation | Term |
|---|---|
| FDA | Food and Drug Administration |
| FSS | Fatigue Severity Scale |
| GCP | Good Clinical Practice |
| ICF | informed consent form |
| ICH | International Conference on Harmonisation |
| IEC | Institutional Ethics Committee |
| IR | immediate release |
| IRB | Institutional Review Board |
| IRLS | International Restless Legs Scale |
| ISI | Insomnia Severity Index |
| IxRS | an interactive voice and web response system |
| KSS | Karolinska Sleepiness Scale |
| LDA | longitudinal data analysis |
| LEM5 | lemborexant, 5-mg dose |
| LEM10 | lemborexant, 10-mg dose |
| LNH | low-normal-high |
| LPS | latency to persistent sleep |
| LS | least square |
| MAR | missing at random |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MHB | median habitual sleep time |
| MI | multiple imputations |
| M-MSLT | modified multiple sleep onset latency test |
| MNAR | missing not at random |
| MUPS | Munich Parasomnia Scale |
| NREM | non-REM sleep |
| PAB | performance assessment battery |
| PBO | placebo |
| PD | pharmacodynamic(s) |
| PGI | Patient Global Impression |
| PI | principal investigator |
| PK | pharmacokinetic(s) |
| PSG | polysomnography |
| PT | preferred term |
| QTcF | QT interval corrected for heart rate by Fridericia's formula |

| Abbreviation | Term |
|--------------|---------------------------------------------------------|
| RBC | red blood cells |
| REM | rapid eye movement (sleep stage) |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SDSB | Sleep Disorders Screening Battery |
| SE | sleep efficiency |
| SOC | system organ class |
| sSE | subjective sleep efficiency |
| sSOL | subjective sleep onset latency |
| sTST | subjective total sleep time |
| sWASO | subjective wake after sleep onset |
| T-BWSQ | Tyrer Benzodiazepine Withdrawal Symptom Questionnaire |
| TEAE | treatment-emergent adverse event |
| TIB | time in bed |
| TST | total sleep time |
| US | United States |
| WASO | wake after sleep onset |
| WASO1H | wake after sleep onset in the first half of the night |
| WASO2H | wake after sleep onset in the second half of the night |
| WBC | white blood cells |
| ZOL | zolpidem tartrate extended release 6.25 mg (Ambien CR®) |

## 5 ETHICS

## 5.1 Institutional Review Boards/Independent Ethics Committees

The protocol, informed consent form (ICF), and appropriate related documents must be reviewed and approved by an Institutional Review Board (IRB) or Independent Ethics Committee (IEC) constituted and functioning in accordance with International Conference on Harmonisation (ICH) E6 (Good Clinical Practice; GCP), Section 3, and any local regulations. Any protocol amendment or revision to the ICF will be resubmitted to the IRB/IEC for review and approval, except for changes involving only logistical or administrative aspects of the study (eg, change in clinical research associates [CRAs], change of telephone number[s]). Documentation of IRB/IEC compliance with the ICH E6 and any local regulations regarding constitution and review conduct will be provided to the sponsor.

A signed letter of study approval from the IRB/IEC chairman must be sent to the principal investigator (PI) (or if regionally required, the head of the medical institution) with a copy to the sponsor before study start and the release of any study drug to the site by the sponsor or its designee (ICH E6, Section 4.4). If the IRB/IEC decides to suspend or terminate the study, the investigator (or if regionally required, the head of the medical institution) will immediately send the notice of study suspension or termination by the IRB/IEC to the sponsor.

Study progress is to be reported to IRB/IECs annually (or as required) by the investigator or sponsor, depending on local regulatory obligations. If the investigator is required to report to the IRB/IEC, he/she will forward a copy to the sponsor at the time of each periodic report. The investigator(s) or the sponsor will submit, depending on local regulations, periodic reports and inform the IRB/IEC (or if regionally required, the investigator and the relevant IRB via the head of the medical institution) of any reportable adverse events (AEs) per ICH guidelines and local IRB/IEC standards of practice. Upon completion of the study, the investigator will provide the IRB/IEC with a brief report of the outcome of the study, if required.

At the end of the study, the sponsor should notify the IRB/IEC and Competent Authority within 90 days. The end of the study will be the date of the last study visit for the last subject in the study. The sponsor should also provide the IRB/IEC with a summary of the study's outcome.

In the case of early termination/temporary halt of the study, the investigator should notify the IRB/IEC and Competent Authority within 15 calendar days, and a detailed written explanation of the reasons for the termination/halt should be given.

# 5.2 Ethical Conduct of the Study

This study will be conducted in accordance with standard operating procedures of the sponsor (or designee), which are designed to ensure adherence to GCP guidelines as required by the following:

Eisai 

- o Principles of the World Medical Association Declaration of Helsinki
- o ICH E6 Guideline for GCP (CPMP/ICH/135/95) of the European Agency for the Evaluation of Medicinal Products, Committee for Proprietary Medicinal Products, International Conference on Harmonisation of Pharmaceuticals for Human Use
- Title 21 of the United States (US) Code of Federal Regulations (US 21 CFR) regarding clinical studies, including Part 50 and Part 56 concerning informed subject consent and IRB regulations and applicable sections of US 21 CFR Part 312
- European Good Clinical Practice Directive 2005/28/EC and Clinical Trial Directive 2001/20/EC for studies conducted within any European Union (EU) country. All suspected unexpected serious adverse reactions (SUSARs) will be reported, as required, to the Competent Authorities of all involved EU member states.
- Other applicable regulatory authorities' requirements or directives

# 5.3 Subject Information and Informed Consent

As part of administering the informed consent document, the investigator (or designee) must explain to each subject the nature of the study, its purpose, the procedures involved, the expected duration, the potential risks and benefits involved, any potential discomfort, potential alternative procedure(s) or course(s) of treatment available to the subject, and the extent of maintaining confidentiality of the subject's records. Each subject must be informed that participation in the study is voluntary, that he/she may withdraw from the study at any time, and that withdrawal of consent will not affect his/her subsequent medical treatment or relationship with the treating physician.

This informed consent should be given by means of a standard written statement, written in nontechnical language. The subject should understand the statement before signing and dating it and will be given a copy of the signed document. After the ICF and any other written information to be provided to subjects is read and explained to the subject, and after the subject has orally consented to the subject's participation in the study and, if capable of doing so, has signed and personally dated the ICF, the witness should sign and personally date the consent form. The subject will be asked to sign an ICF before any study-specific procedures are performed. No subject can enter the study before his/her informed consent has been obtained.

An unsigned copy of an IRB/IEC-approved ICF must be prepared in accordance with ICH E6, Section 4, and all applicable local regulations. The form must be signed and dated by the appropriate parties. The original, signed ICF for each subject will be verified by the sponsor and kept on file according to local procedures at the site.

The subject should be informed in a timely manner if new information becomes available that may be relevant to the subject's willingness to continue participation in the study. The communication of this information should be documented.

Eisai 

## **6 INVESTIGATORS AND STUDY PERSONNEL**

This study will be conducted by qualified investigators under the sponsorship of Eisai (the sponsor) at approximately 105 investigational sites in North America and Europe. (revised per Amendment 02)

The name and telephone and fax numbers of the Medical Monitor and other contact personnel at the sponsor and of the contract research organization(s) (CRO[s]) are listed in the Investigator Study File provided to each site.

## 7 INTRODUCTION

#### 7.1 Indication

## 7.1.1 Current Therapeutic Options

Insomnia is a sleep disorder characterized by difficulties with sleep onset, sleep maintenance, or early morning awakening, in association with a complaint of impairment during the daytime. Insomnia is a widespread problem in industrialized nations, with approximately 30% of the population having symptoms and at least 6% meeting diagnostic criteria for insomnia meriting treatment. Currently available pharmacological treatments used for insomnia include benzodiazepines, non-benzodiazepine γ-aminobutyric acid (GABA) receptor agonists (GABAergics), a recently approved dual orexin receptor antagonist (DORA), sedating antidepressants, melatonin and melatonin agonists, antihistamines, and other prescription and non-prescription medications with sedative properties.

The current commercial environment is generic, with the non-benzodiazepine, zolpidem (Ambien®), leading in prescriptions in the US. Other so-called "z-drugs" including zaleplon and eszopiclone, contribute substantially to market share as well. However, there are efficacy and safety concerns associated with the use of z-drugs, particularly zolpidem, particularly in older patients. This limited efficacy is characteristic of short-acting non-benzodiazepine hypnotics and represents an important unmet medical need, as sleep maintenance insomnia is the most prevalent type of insomnia experienced in aging. Up to 50% of individuals over age 55 report difficulty maintaining sleep. The recently approved DORA, suvorexant, was shown in clinical trials to significantly improve sleep maintenance insomnia, but at the starting dose approved for use, showed suboptimal efficacy.

## 7.1.2 Lemborexant (E2006)

#### 7.1.2.1 Mechanism of Action

Lemborexant, E2006, (1*R*,2*S*)-2-{[(2,4-dimethylpyrimidin-5-yl)oxy]methyl}-2-(3-fluorophenyl)-*N*-(5-fluoropyridin-2-yl)cyclopropanecarboxamide belongs to the pharmacologic class of orexin receptor antagonists.

Orexin neuropeptides (orexin-A and orexin-B) have been recognized as critical upstream controllers of most wake-promoting neurotransmitters via two G protein-coupled receptors, the orexin-1 receptor and the orexin-2 receptor. Small-molecule antagonists of orexin receptors, such as suvorexant, have recently emerged as a new class of chemical compounds that represents a novel alternative approach to treat insomnia disorder.

## 7.1.2.2 Clinical Experience with Lemborexant

#### 7.1.2.2.1 PHASE 1

E2006-A001-001 (Study 001): single ascending dose study. This study included healthy subjects and otherwise healthy subjects with primary insomnia. In addition to determining

Eisai 

the safety and tolerability of single doses, the study provided preliminary evidence of efficacy in the target patient population.

E2006-A001-002 (Study 002): multiple ascending dose study. This study enrolled healthy adult and elderly subjects, each of whom was dosed with lemborexant or placebo at night. In addition to determining the safety and tolerability of multiple doses, the study also provided preliminary evidence of a lack of important differences in exposure between adult and elderly subjects.

E2006-A001-003 (Study 003): A multiple dose study to bridge pharmacokinetics (PK), pharmacodynamics (PD), safety and tolerability between Japanese and white healthy subjects. This study provided evidence of a lack of important differences in exposure and safety between Japanese and white subjects.

E2006-A001-004 (Study 004): metabolism-based inducer/inhibitor study. This study provided data demonstrating (1) strong inhibitors of CYP3A lead to higher plasma concentrations of lemborexant; and (2) strong inducers of CYP3A lead to notably lower plasma concentrations of lemborexant. The study also demonstrated a weak effect of lemborexant on CYP2B6 activity and no effect on CYP3A activity.

E2006-A001-005 (Study 005): relative bioavailability study of capsules vs tablet formulations. This study demonstrated that the capsules and tablets provided similar exposure (maximum observed concentration  $[C_{max}]$  and area under the concentration-time curve [AUC]), thus allowing the tablet formulation to be used in future clinical trials.

E2006-A001-007 (Study 007): human mass balance absorption, distribution, metabolism, and excretion study to characterize the route and extent of excretion of lemborexant. This study demonstrated that elimination takes place by fecal (57%) and urinary excretion (29%) based on total recovery (86.5%) of radioactivity following a single dose of radiolabeled lemborexant. In addition, there were no human-specific metabolites and the only major (12%) metabolite was M10. The blood-to-plasma ratio was approximately 0.65.

E2006-A001-008 (Study 008): food effect study. This study demonstrated a mild food effect. The  $C_{max}$  was decreased by 23% and the area under the concentration-time curve from zero time extrapolated to infinite time (AUC<sub>[0-inf]</sub>) was increased by 18% following consumption of a high fat meal.

E2006-A001-107 (Study 107): This Phase 1 study was conducted to evaluate the effects of the 5 and 10 mg doses on next-morning residual sleepiness in subjects with insomnia disorder. The study design was randomized, double-blind, and placebo (PBO)-controlled with a 3-way crossover. Next-morning residual sleepiness was measured on a modified multiple sleep onset latency test (M-MSLT). An active comparator, flurazepam 30 mg, was included to confirm assay sensitivity. Results showed that for neither 5 mg nor 10 mg was the lower bound of the 95% confidence interval (CI) of the treatment difference in change from baseline of average sleep onset latency on the M-MSLT more than -6 minutes, which was the prespecified criterion defining clinically meaningful next-morning residual sleepiness. That is, neither dose level of E2006 resulted in a clinically meaningful reduction

in average time to sleep onset in the morning hours, supporting the safety of these doses and their use in Phase 3 studies.

#### 7.1.2.2.2 PHASE 2

A dose-finding study (E2006-G000-201; Study 201) was conducted in subjects who had insomnia disorder, with the primary objectives of identifying doses that resulted in efficacy but did not result in significant next-day residual sleepiness. The doses evaluated were 1, 2.5, 5, 10, 15, and 25 mg, administered once daily for 15 days. The study was stopped early for efficacy after the prespecified success criterion for sleep efficiency (SE) was achieved without unacceptable next-day residual sleepiness as evaluated by the Karolinska Sleepiness Scale (KSS).

As measured by polysomnography (PSG), improvements in sleep were also demonstrated by statistically significant increases from baseline in SE, and by decreases from baseline in mean latency to persistent sleep (LPS) and wake after sleep onset (WASO). These changes were largely maintained over 15 days of treatment with lemborexant as compared with Subjective measures derived from sleep diary entries yielded results largely comparable to PSG-derived results. Further, there was no evidence of rebound insomnia after treatment was completed, as measured either by PSG or Sleep Diary.

At doses up to 10 mg, changes from baseline in next-day sleepiness, as measured by the KSS, did not differ from those after placebo. At the highest doses of 15 and 25 mg, the increase in KSS from baseline was statistically significantly different from placebo at some time points, but the increases in KSS were of small magnitude (ie, less than 1 unit on average). Although there was approximately a two-fold accumulation of lemborexant in plasma over the 15-day Treatment Period, next-day sleepiness did not increase from the beginning to the end of treatment.

Overall, data from the clinical program to date have shown an acceptable safety and tolerability profile of lemborexant, and efficacy on both objective and subjective measures of sleep onset and sleep maintenance.

#### 7.2 Study Rationale

The purpose of this study is to provide important information to begin to improve on the current treatment paradigm for older patients with sleep maintenance insomnia. The study will help establish the efficacy of lemborexant for the treatment of sleep onset and sleep maintenance difficulties, by comparing change from baseline in these parameters to placebo. With respect to comparisons to existing therapies, the current market leader, zolpidem has been shown to improve sleep onset insomnia. The immediate release (IR) formulation of zolpidem is not, however, indicated for sleep-maintenance insomnia. The extended release formulation, zolpidem tartrate extended release 6.25 mg (Ambien CR®; ZOL), was approved by the Food and Drug Administration (FDA) for the treatment of sleep maintenance symptoms as well as for sleep onset difficulties. However, 2 studies, one using 12.5 mg in adults and the other studying 6.25 mg in elderly patients, reported that effects on WASO after nights 1 and 2 of treatment were only statistically significantly different from placebo

Eisai  FINAL: (v7.0), 05 Feb 2018

for the first 6 hours (adults) or first 5 hours (elderly) of the 8-hour sleep period. After 2 weeks of treatment, WASO was significantly decreased for only the first 5 hours (adults) and first 4 hours (elderly) of the 8-hour sleep period. Given that this is the time of night when most sleep maintenance difficulties are experienced, particularly by elderly individuals, there is an unmet need that has not been effectively addressed with ZOL. In brief, while ZOL improves sleep maintenance more than the IR formulation, it does not sufficiently decrease WASO in the second half of the night (WASO2H). Nonetheless, ZOL was approved based on data for the first 6 hours of the sleep period. It should be noted that the pivotal studies for ZOL were based on data from 3-week trials analyzed for Nights 1/2 and 15/16. A comparison of lemborexant with ZOL, especially with respect to sleep maintenance, would provide clinically meaningful information for clinicians and patients. (revised per Amendment 03)

## 8 STUDY OBJECTIVES

# 8.1 Primary Objective – US and Non-US (revised per Amendment 03)

Demonstrate using PSG that lemborexant (LEM10 and LEM5) is superior to PBO on objective sleep onset as assessed by LPS after the last 2 nights of 1 month of treatment in subjects 55 years and older with insomnia disorder.

# 8.2 Secondary Objectives

- 8.2.1 Key Secondary Objectives US ONLY (revised per Amendment 03)
- Demonstrate that lemborexant (LEM10 and LEM5) is superior to PBO on sleep maintenance as assessed by sleep efficiency (SE) after the last 2 nights of treatment
- Demonstrate that lemborexant (LEM10) and LEM5) is superior to PBO on sleep maintenance as assessed by WASO after the last 2 nights of treatment (revised per Amendment 04)
- Demonstrate that lemborexant (LEM10 and LEM5) is superior to ZOL on WASO2H after the last 2 nights of treatment
- 8.2.2 Key Secondary Objectives Non-US ONLY (revised per Amendment 03)
- Demonstrate that lemborexant (LEM10 and LEM5) is superior to PBO on sleep maintenance as assessed by SE after the last 2 nights of treatment
- Demonstrate that lemborexant (LEM10 and LEM5) are superior to PBO on WASO after the last 2 nights of treatment
- 8.2.3 Additional Secondary Objectives US and Non-US (revised per Amendment 03)
- Demonstrate that LEM5 or LEM10 or both LEM5 and LEM10 are superior to ZOL on postural stability in the morning after the first 2 nights of treatment
- Determine whether the efficacy of LEM5 or LEM10, or both LEM5 and LEM10, is superior to that of ZOL on selected PSG variables after the first 2 nights and the last 2 nights of treatment and on selected Sleep Diary variables over the first 7 nights and last 7 nights of treatment.
- Confirm the efficacy of LEM5 and LEM10 compared to PBO on sleep as measured by PSG after the first 2 and last 2 nights of treatment and as measured by Sleep Diary over the first 7 and last 7 nights of treatment
- Evaluate the proportions of sleep onset and sleep maintenance responders to LEM5 and LEM10 and determine whether they are superior to those for ZOL and PBO as defined by response on PSG LPS and WASO and Sleep Diary subjective sleep onset latency (sSOL) and subjective wake after sleep onset (sWASO)
- Evaluate the safety and tolerability of lemborexant

- Determine whether the efficacy of LEM5 or LEM10, or both LEM5 and LEM10, is superior to that of ZOL and PBO on daytime functioning as assessed by the Insomnia Severity Index (ISI) and Fatigue Severity Scale (FSS) at the end of treatment
- Determine whether the safety of LEM5 or LEM10, or both LEM5 and LEM10, is superior to that of ZOL and PBO as assessed by cognitive performance in the morning after the first 2 nights of treatment

# 8.3 Exploratory Objectives – US and Non-US (revised per Amendment 03)

- Explore the effects of LEM5, LEM10, ZOL and PBO on:
  - Subjective quality of sleep
  - o Postural stability in the morning after the last 2 nights of treatment
  - o Cognitive performance after the last 2 nights of treatment
  - Rebound insomnia in the 2 weeks following 30 days of treatment
  - Subjective ratings of morning sleepiness during and following completion of treatment
  - Sleep architecture parameters and other PSG variables
  - Health outcomes on the Patient Global Impression Insomnia (Patient Global Impression [PGI]-Insomnia) and EQ-5D-3L
  - Withdrawal symptoms after completion of treatment
- Summarize plasma concentrations of lemborexant and its metabolites M4, M9, and M10
- Conduct population PK modeling for lemborexant
- Explore PK/PD relationships between lemborexant concentrations and efficacy and safety variables

### 9 INVESTIGATIONAL PLAN

# 9.1 Overall Study Design and Plan

E2006-G000-304 is a multicenter, randomized, double-blind, placebo-controlled, active comparator (ie, ZOL), parallel-group study of 2 dose levels of lemborexant for 30 nights in approximately 950 subjects 55 years or older with insomnia disorder. Subjects will be males 65 years or older or females 55 years or older. Approximately 60% of the population will be age 65 years or older. (revised per Amendment 03)

The study will have 2 phases, the Prerandomization Phase and the Randomization Phase. The Prerandomization Phase will comprise 3 periods that will last up to a maximum of 35 days: a Screening Period, a Run-in Period, and a Baseline Period. The Randomization Phase will comprise a Treatment Period during which subjects are treated for 30 nights followed by a minimum 14-day interval before an End of Study (EOS) Visit. (revised per Amendment 02)

Throughout the Prerandomization Phase and the Randomization Phase, all subjects will undergo routine safety assessments at specified visits, including questioning regarding AEs, 12-lead electrocardiograms (ECGs), vital signs, weight, height, clinical hematology and chemistry analysis and urinalysis, and suicidality.

Estimates for End of study are as follows:

- The study will begin in approximately Apr 2016
- o The end of the study will be the date of the last study visit for the last subject in the study.
- The estimated duration for each subject on study is anticipated to be a maximum of 81 days / 11.5 weeks (Screening Period plus Run-in Period plus Baseline Period maximum of 35 days plus Treatment Period plus Follow-up Period and EOS Visit maximum of 53 days). A subject who completes the Treatment Period (assessments through discharge from clinic on the morning of Day 31) will be considered to have completed the study. (revised per Amendment 02)

The study design is shown in Figure 1.



# = CDR Posture and cognitive PAB assessments in the morning following the PSG assessment.

a: All PSG visits will require an overnight stay in the clinic. At least 2 nights must intervene between the second BL PSG and BL (D1).

## Figure 1 Schematic Diagram of E2006-G000-304 Study Design

"D" refers to the study day.

BL = baseline, CDR = Cognitive Drug Research, LEM5 = lemborexant 5 mg, LEM10 = lemborexant 10 mg, PAB = performance assessment battery, PBO = placebo, PSG = polysomnography, ZOL = zolpidem tartrate extended release 6.25 mg.

Eisai 

#### 9.1.1 Prerandomization Phase

## 9.1.1.1 Screening Period

The Screening Period will begin no more than 35 days before the subject is randomized. At the first screening visit (Visit 1), informed consent will be obtained after the study has been fully explained to each subject and before the conduct of any screening procedures or assessments. A medical, psychiatric, and sleep history interview will be conducted, and will include confirmation that the subject meets diagnostic criteria for insomnia disorder, and further that the subject complains of difficulties with sleep maintenance or early morning awakening, or both. Screening assessments will include the ISI, as well as the Epworth Sleepiness Scale (ESS), the STOPBang, the International Restless Legs Scale (IRLS), and the Munich Parasomnia Scale (MUPS), collectively called the Sleep Disorders Screening Battery (SDSB). Additional eligibility criteria will be assessed and safety assessments will be conducted as described in Section 9.5.1.5 and summarized in Table 4. (revised per Amendment 02)

Subjects will be provided with an electronic device on which they will complete the Sleep Diary and will be trained in the use of this device. Site staff will instruct subjects to complete the diary each morning within 1 hour after morning waketime and will emphasize the importance of doing so. The Sleep Diary entries will be reviewed by site staff at least weekly throughout the study to ensure subject compliance with completion of the Sleep Diary and to ensure that study restrictions are met pertaining to duration of time spent in bed, and use of alcohol.

After subjects have completed the Sleep Diary on at least 7 consecutive mornings, and provided that the Sleep Diary entries indicate continued eligibility with regard to sleep timing, duration of time spent in bed, and frequency of nights with symptoms of insomnia, subjects will undergo the second screening visit. (Subjects who are not eligible on the basis of Sleep Diary entries will return to the clinic for debriefing purposes and to return study equipment.) This visit must occur between Day -17 and Day -10. On this and all nights on which PSG is to be recorded, subjects will arrive at the clinic in the evening with sufficient time before bedtime to complete check-in procedures, any scheduled assessments, and preparations (eg, electrode montage placement) for the PSG recordings. In addition, at check-in before all visits at which PSG is to be recorded, subjects will undergo a urine drug test. (revised per Amendment 02)

After check-in has been completed, study personnel will familiarize subjects with the postural stability assessment (CDR posture assessment) and will also conduct a minimum of 2 training sessions for the cognitive performance assessment battery (PAB). Subjects will then undergo an 8-hour PSG recording, to start at the median habitual bedtime (MHB) as calculated from the Sleep Diary entries. The PSG recording will include channels in the electrode montage to screen for symptoms of sleep apnea and periodic limb movement disorder. Within 5 minutes of morning waketime, the CDR posture and PAB assessments will be administered under the same conditions (eg, timing of assessments relative to waketime, ambient lighting), as will be employed during the testing sessions. The CDR

Eisai 

posture and PAB assessments at this time are for familiarization purposes only. At 1.5 hours after waketime, subjects will rate their morning sleepiness level. The PSG will be reviewed for exclusion criteria related to absence of symptoms of sleep apnea and/or periodic limb movement disorder, subjects who continue to meet the eligibility criteria will then be dispensed PBO tablets (single-blind) and will enter the Run-in Period.

#### 9.1.1.2 Run-in Period

The Run-in Period will begin when eligible subjects are dispensed PBO tablets and will continue until the Baseline Period on Day 1. During the Run-in Period, subjects will take PBO each night immediately (ie, within 5 minutes) before bedtime (defined as the time the subject intends to try to fall asleep). They will be reminded that they must remain in bed for at least 7 hours each night and maintain a regular bedtime throughout the study according to the schedule determined by the study site and the subject. They will also be reminded that they must follow study restrictions with regard to timing of meals and use of caffeine and alcohol.

When subjects have completed the Sleep Diary on at least 7 consecutive mornings during the Run-In Period, the diary will be reviewed for continued eligibility with regard to whether the subject continues to report sWASO ≥60 minutes on at least 3 of the 7 nights, as well as the schedule and duration of time spent in bed. Subjects who are still eligible will return to the clinic for the first of two consecutive nights on which PSG will be recorded. (Subjects who are not eligible on the basis of Sleep Diary entries will return to the clinic for debriefing purposes and to return study equipment.) The first of these 2 nights must be between Day -10 and Day -4. In the evening before the PSG recording, the ISI, the FSS, and the EQ-5D-3L will be assessed. The ISI score will be reviewed for eligibility and safety assessments will be conducted. Study personnel will administer study drug to subjects within 5 minutes before their scheduled bedtime, which will be at the same MHB as used for the second screening visit. Subjects will then undergo an 8-hour PSG. The next morning, subjects will undergo assessments including the CDR posture and PAB assessments and will complete the Sleep Diary. At 1.5 hours after waketime, subjects will rate their morning sleepiness level. The PSG recording will be reviewed for continued eligibility and subjects may then leave the clinic only after the investigator determines that is safe for them to do so. (revised per Amendment 02)

Subjects will return to the clinic that evening. Study personnel will administer study drug to subjects within 5 minutes before the scheduled bedtime. A PSG will be recorded overnight. The following morning subjects will undergo postural stability and PAB assessments and will complete the Sleep Diary. At 1.5 hours after waketime, subjects will rate their morning sleepiness level. The PSG recording will be reviewed for continued eligibility, and both PSGs during the Run-in Period will also serve as the baseline for PSG-derived endpoints for subjects who are randomized. Subjects may then leave the clinic only after the investigator determines that is safe for them to do so.

Subjects will continue to take study drug at home within 5 minutes before bedtime and they will continue to complete the Sleep Diary each morning within 1 hour after morning waketime. They will again be reminded that they must remain in bed for at least 7 hours

Eisai 

each night maintain a regular bedtime throughout the study, and follow study restrictions with regard to timing of meals and use of caffeine and alcohol.

#### 9.1.1.3 Baseline Period

After a minimum of 2 nights following the baseline PSGs, the Run-in Period will end and the Baseline Period will take place. On Day 1 subjects will be admitted to the clinic and the ISI, FSS, and EQ-5D-3L will be administered. Blood and urine samples will be collected for routine safety assessments, ECG will be performed, and vital signs and weight will be assessed. The electronic Columbia-Suicide Severity Rating Scale (C-SSRS) will be administered. Subjects who complete the Baseline Period and continue to meet the eligibility criteria will be randomized and will begin the Treatment Period. (revised per Amendment 02)

#### 9.1.2 Randomization Phase

#### 9.1.2.1 Treatment Period

The Treatment Period will begin on Day 1, and will continue until Day 31. Subjects will be randomized in a double-blind manner, to receive LEM5, LEM10, ZOL, or PBO. (revised per Amendment 02)

Within 5 minutes before the subject's MHB, study drug will be administered and an overnight PSG will be initiated. At completion of the PSG recording the following morning (Day 2), postural stability will be assessed and the PAB will be conducted immediately thereafter. Subjects will complete the Sleep Diary. At 1.5 hours after waketime, subjects will rate their morning sleepiness level. (revised per Amendment 01) They may then leave the clinic after the investigator determines that is safe for them to do so.

On the evening of Day 2, subjects will return to the clinic. A PK blood sample will be collected predose and study drug will be administered within 5 minutes before the subject's MHB, followed by an overnight PSG. The next morning (Day 3), the CDR posture and PAB assessments will be conducted and a PK blood sample will be obtained.

Subjects will complete the Sleep Diary. The electronic Columbia-Suicide Severity Rating Scale (eC-SSRS) will be administered. At 1.5 hours after waketime, subjects will rate their morning sleepiness level. Subjects may then leave the clinic after the investigator determines that is safe for them to do so. Study drug will be dispensed, and subjects will be provided with instructions to continue to complete the Sleep Diary each morning within 1 hour of waketime and to take study drug daily at home according to the same schedule and with the same instructions as during the Run-in Period.

On Day 29, subjects will return to the clinic. Study drug will be administered within 5 minutes before the subject's MHB, followed immediately by a PSG. On the morning of Day 30, postural stability will be assessed and the PAB will be conducted. At 1.5 hours after waketime, subjects will rate their morning sleepiness level. Subjects may leave the clinic after the investigator determines that is safe for them to do so.

Eisai 

On the evening of Day 30, subjects will return to the clinic. A PK blood sample will be collected predose and study drug will be administered within 5 minutes before the subject's MHB, followed by a PSG. On the morning of Day 31, postural stability and PAB assessments will be conducted and a PK sample will be obtained. Then the ISI, FSS, EQ-5D-3L and PGI-Insomnia will be administered. Blood and urine samples will be collected for routine safety assessment. An ECG will be performed, and vital signs and weight will be assessed. The eC-SSRS will be administered. At 1.5 hours after waketime, subjects will rate their morning sleepiness level. Then, after the investigator determines that it is safe for them to do so, subjects will be discharged from the clinic.

## 9.1.2.2 Follow-up Period

The Follow-up Period will begin when the subjects leave the clinic at the end of the Treatment Period. Subjects will cease to take study drug but will continue to complete the Sleep Diary each morning until the EOS Visit.

At least 14 days but no more than 18 days after completion of the Treatment Period, subjects will return to the clinic for the EOS Visit. The Tyrer Benzodiazepine Withdrawal Symptom Questionnaire (T-BWSQ) and eC-SSRS will be administered, and routine safety assessments will be conducted.

A subject who prematurely discontinues taking study drug should return to the clinic as soon as practicable after discontinuing study drug, to complete an Early Termination (ET) Visit. If the subject discontinues from the study due to an AE, the subject must complete an ET Visit and the AE must be followed to resolution or for 2 weeks, whichever comes first. In addition, subjects who withdraw due to an AE should undergo a urine drug test.

# 9.2 Discussion of Study Design, Including Choice of Control Groups

#### 9.2.1 Randomization

Randomization will be used in this study to avoid bias in the assignment of subjects to treatment, to increase the likelihood that known and unknown subject attributes (eg, demographics and baseline characteristics) are balanced across treatment groups, and to ensure the validity of statistical comparisons across treatment groups. Blinding to treatment will be used to reduce potential bias during data collection and evaluation of endpoints.

#### 9.2.2 Run-In

Insomnia trials are associated with large placebo effects. This study will include a placebo Run-in Period to exclude subjects who show a response to placebo. (revised per Amendment 03)

The Run-in Period will also help to identify and exclude subjects who are not compliant with the Sleep Diary instructions, duration of time spent in bed, or restrictions on alcohol use. In this regard, it is necessary for the subjects to be taking PBO and to obtain Sleep Diary data for a minimum of 1 week to adequately evaluate whether there is a PBO response and

Eisai 

compliance with the alcohol-related study restrictions. After this minimum 7 nights of treatment, eligible subjects will have PSG recordings on 2 consecutive nights. These recordings will be used to further screen for eligibility, and will serve as baseline values for those subjects who continue to randomization.

## 9.2.3 Efficacy Assessments

The study uses objective (PSG) as well as subjective (Sleep Diary) assessments of efficacy. Both assessments have been widely used in registration trials evaluating treatments for insomnia disorder. While PSG indicates that a measurable physiological effect of the study drug has occurred, Sleep Diary outcomes indicate the magnitude of the effect for the patient. (revised per Amendment 03)

Another focus of this study is on WASO2H, a measure of sleep maintenance in the second half of the night. The rationale for the selection of this endpoint is based on the loss of effect of ZOL on sleep maintenance at the end of the sleep period. However, any benefit on WASO2H observed with lemborexant must not be due to a worsening of sleep latency or continuity at the beginning of the night. Therefore, analyses of both LPS and total WASO as well as other PSG variables (eg, total sleep time [TST], number and duration of awakenings) will be conducted to confirm the efficacy of lemborexant on sleep onset and sleep maintenance. (revised per Amendment 03)

## 9.2.4 Morning Residual Effects on Postural Stability and Cognitive Performance

Non-benzodiazepine sleep-inducing agents such as zolpidem have been associated with motor and cognitive impairment, and laboratory studies have evaluated these impairments both during the middle of the night several hours postdose, and in the morning hours shortly after awakening. Of clinical importance is that the elderly are particularly sensitive to effects of zolpidem on postural stability, which is especially problematic given the increased risk of falls in the elderly.

Moderate to large treatment effects versus placebo on measures of postural stability and cognitive performance have been reported for both 5 mg and 10 mg doses of the IR formulation of zolpidem (Allain, et al., 2003, Mets, et al., 2010, and Boyle, et al., 2009; reviewed in Stranks and Crowe, 2014). Larger impairments are observed near the  $C_{max}$  of the zolpidem IR formulation at approximately 1.5 hours postdose than at later timepoints relative to dosing, but there remains a moderate impairing effect of zolpidem even the next morning on certain cognitive domains including attention and memory (Stranks and Crowe, 2014).

With regard to postural stability as measured in this study, zolpidem is assumed to have the same effect on body sway as alcohol at 4.5 hours after dosing (Wesnes, et al., 2000). Further, there is consistent evidence that the effects on postural stability of hypnotic drugs are larger after the first one or two nights of dosing and dissipate thereafter, which has been explained as due to behavioral tolerance (Mets, et al., 2010). For this reason, the key secondary objective for the current study is to compare the effects of lemborexant to those of zolpidem on postural stability at the beginning of treatment, in the morning shortly after waketime on Day 2 and Day 3. Whether there are differential effects of lemborexant and

Eisai 

zolpidem on postural stability at the end of treatment (Day 30 and Day 31) will be explored. Effects on cognitive performance in the morning shortly after waketime will be exploratory for both the beginning and end of treatment.

# 9.2.5 Adjudication Committee (revised per Amendment 02)

An independent Adjudication Committee will be employed at intervals to review, in a blinded manner, AEs that could potentially be considered cataplexy or seizure. A set of preferred terms constituting a customized Medical Dictionary for Regulatory Activities (MedDRA) query for cataplexy or seizure will be used to identify events for adjudication (including cataplexy, muscle fatigue, muscular weakness, muscle tone disorder, hypotonia, drop attacks, slurred speech, diplopia, falls, convulsions, atypical migraine, loss of consciousness, decreased consciousness, myoclonus, syncope, transient global amnesia, lipothymia and transient ischemic attack). To assist in the preparation of narratives about such events and to support the committee's adjudication process, investigators and site staff will be instructed to query subjects who report any of the above events for supplemental information about events of cataplexy or potential cataplexy events, using a questionnaire for events potential related to cataplexy and the SAE form for any of the above events considered serious. (revised per Amendment 02)

## 9.2.6 Study Duration

The registration trials for zolpidem were 3 weeks in duration, with analyses of PSG efficacy data conducted after the first 2 doses and at the end of 2 weeks of active treatment. As noted, treatment benefit of zolpidem declined over time such that WASO2H, particularly in the last 2 hours of the night, was not different from placebo on Nights 15/16 in the zolpidem registration trials. In contrast, when lemborexant was studied for 15 nights of treatment in Study 201, the treatment benefit was maintained such that there was no significant difference in LPS, WASO, or WASO2H between the first 2 and last 2 nights of treatment. Study 304 includes 30 days of active treatment. Based on the results of Study 201, it is expected that there will not be a loss of efficacy of lemborexant between 2 weeks and 4 weeks of treatment.

Moreover, as the beneficial effects of zolpidem on WASO2H did not persist for 2 weeks, it is not expected that there will be statistically or clinically significant effects of ZOL at the end of the 30 days of treatment.

## 9.2.7 Age Group

While the lower age is not the typical 65 years defining "elderly," it is physiologically meaningful, as insomnia incidence increases at middle age in both men and women, with a particularly steep increase in incidence in women at menopause. In addition, the homeostatic and circadian regulation of sleep are disturbed in many older individuals, which manifests most frequently as sleep maintenance insomnia in the second half of the night, and early morning awakening. The preponderance of sleep maintenance issues in the second half of the sleep period is clear from the literature as well as supported by analyses of data by age group from Study 201. (revised per Amendment 03)

Eisai 

When Study 201 data were analyzed separately for those aged 55 years and older, the apparent treatment effect of lemborexant versus placebo on WASO2H, as well as on WASO, was larger than for the full sample (all ages studied), suggesting that older individuals may be most likely to benefit from a treatment that reduced difficulties with both sleep onset and sleep maintenance. Table 1 shows the least square (LS) mean treatment difference between lemborexant and PBO for various dose groups and dose group combinations from Study 201 for the full sample and for those aged 55 and older. Caution must be exercised concerning the predictive ability of these data, however, since the observed variability in WASO2H was larger in the older subjects. For this reason, a conservative estimate of the expected treatment difference between lemborexant and PBO for WASO2H at the end of treatment was used for power analyses and sample size justification. Enrollment in this study is exclusively older subjects, aged 55 years and older. (revised per Amendment 03)

Table 1 Treatment Effect for Lemborexant versus Placebo (Study 201)

| | Treatment Effect in Minutes (95% CI) | | |
|---|---|---|---|
| | 5 mg | 10 mg | 5 and 10 mg<br>combined |
| Entire Subject Sample | -7.97 | -11.8 | -10.0 |
| | (-19.2, 3.23) | (-23.6, -0.05) | (-20.6, 0.55) |
| Aged 55 and Older | -23.9 | -14.8 | -20.2 |
| | (-43.8, -3.95) | (-36.9, 7.36) | (-40.1, -0.35) |

CI = confidence interval

# 9.2.8 Time of Dosing

The time of dosing of study drug will be within 5 minutes before bedtime on nights in the clinic. On nights at home, subjects will be instructed to take study drug just before they intend to try to fall asleep, but as consistently as possible with respect to the time across the study.

### 9.2.9 Interim Analysis

An interim analysis is planned to be conducted after 50% of the subjects (approximately 475 subjects) have been randomized and have either completed Day 31 assessments or discontinued from the study. The purpose of this analysis is to determine the conditional probability that a statistically significant difference between LEM10 and ZOL on WASO2H will emerge at the end of treatment. This interim analysis will be conducted by an independent statistician external to the Sponsor. The role of the independent statistician and procedures undertaken to preclude potential bias will be detailed in the statistical analysis plan (SAP) and in the Charter.

Eisai 

# 9.3 Selection of Study Population

Approximately 2800 subjects will be screened and approximately 950 subjects will be randomized at approximately 105 sites in North America and Europe. Subjects who do not meet all of the inclusion criteria or who meet any of the exclusion criteria will not be eligible to receive study drug. A table providing guidelines on the order in which criteria should be assessed and at what visits can be found in Appendix 2. (revised per Amendment 02)

### 9.3.1 Inclusion Criteria

- 1. Male age 65 years or older or female, age 55 years or older at the time of informed consent
- 2. Meets the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition criteria for Insomnia Disorder, as follows:
  - Complains of dissatisfaction with nighttime sleep, in the form of difficulty staying asleep and/or awakening earlier in the morning than desired despite adequate opportunity for sleep (Note that if the complaint is limited to difficulty initiating sleep, the subject is not eligible)
  - o Frequency of complaint  $\ge$  3 times per week
  - Duration of complaint  $\ge$  3 months
  - o Associated with complaint of daytime impairment
- 3. At Screening: History of subjective WASO (sWASO) typically  $\geq$  60 minutes on at least 3 nights per week in the previous 4 weeks
- 4. At Screening: Reports regular time spent in bed, either sleeping or trying to sleep, between 7 and 9 hours
- 5. At Screening: Reports habitual bedtime, defined as the time the subject attempts to sleep, between 21:00 and 24:00 and habitual waketime between 05:00 and 09:00
- 6. At Screening and at check-in before the first PSG during the Run-in Period: ISI score ≥13 (revised per Amendment 02)
- 7. Confirmation of current insomnia symptoms as determined from responses on the Sleep Diary on the 7 most recent mornings (minimum 5 of 7 for eligibility) before the second screening visit, such that sWASO ≥ 60 minutes on at least 3 of the 7 nights
- 8. Confirmation of regular bedtime and waketime as determined from responses on the Sleep Diary on the 7 most recent mornings before the second screening visit, such that neither bedtime, (defined as the time the subject attempts to try to sleep), nor waketime (defined as the time the subject gets out of bed for the day) deviates more than 1 hour on more than 2 nights from the calculated MHB or median habitual waketime, respectively, from the Screening Sleep Diary entries
- 9. Confirmation of sufficient duration of time spent in bed, as determined from responses on the Sleep Diary on the 7 most recent mornings before the second

Eisai 

- screening visit, such that there is not more than 2 nights with time spent in bed duration < 7 hours or > 10 hours (revised per Amendment 02)
- 10. During the Run-in Period: Reconfirmation of insomnia symptoms, as determined from responses on the Sleep Diary on the 7 most recent mornings before the first PSG during the Run-in Period, such that sWASO ≥ 60 minutes on at least 3 of the 7 nights
- 11. During the Run-in Period: Reconfirmation of regular bedtimes and waketimes as defined in Inclusion Criterion 8
- 12. During the Run-in Period: Reconfirmation of sufficient duration of time spent in bed as defined in Inclusion Criterion 9 (revised per Amendment 02)
- 13. During the Run-in Period: Objective (PSG) evidence of insomnia as follows: WASO average ≥ 60 minutes on the 2 consecutive PSGs, with neither night < 45 minutes (revised per Amendment 02)
- 14. Willing and able to comply with all aspects of the protocol, including staying in bed for at least 7 hours each night
- 15. Willing not to start a behavioral or other treatment program for the treatment of insomnia during the subject's participation in the study

#### 9.3.2 Exclusion Criteria

- 1. A current diagnosis of sleep-related breathing disorder (including obstructive sleep apnea with or without continuous positive airway pressure [CPAP] treatment), periodic limb movement disorder, restless legs syndrome, circadian rhythm sleep disorder, or narcolepsy, or an exclusionary score on screening instruments to rule out individuals with symptoms of certain sleep disorders other than insomnia as follows: (revised per Amendment 01)
  - a. STOPBang score ≥5
  - b. International Restless Legs Scale score ≥16
  - c. Epworth Sleepiness Scale score >15 (Scores of 11-15 require excessive daytime sleepiness to be recorded in subject's Medical History) (revised per Amendments 01 and 02)
- 2. Reports symptoms potentially related to narcolepsy that in the clinical opinion of the investigator indicates the need for referral for a diagnostic evaluation for the presence of narcolepsy (revised per Amendment 01)
- 3. On the MUPS, endorsed the item that corresponds to a history of sleep-eating or reports a history of sleep-related violent behavior, sleep-driving or symptoms of another parasomnia that in the investigator's opinion make the subject unsuitable for the study (revised per Amendment 02)
- 4. Apnea-Hypopnea Index > 15 or Periodic Limb Movement with Arousal Index > 15 as measured on the PSG at the second screening visit
- 5. Beck Depression Inventory II (BDI-II) score >19 at Screening

Eisai 

- 6. Beck Anxiety Inventory (BAI) score >15 at Screening
- 7. Habitually naps during the day more than 3 times per week
- 8. Is a female of childbearing potential
  - Note: All females will be considered to be of childbearing potential unless they are postmenopausal (defined as amenorrheic for at least 12 consecutive months, are in the appropriate age group, and are postmenopausal without other known or suspected cause), or have been sterilized surgically (ie, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing).
- 9. Excessive caffeine use that in the opinion of the investigator contributes to the subject's insomnia, or habitually consumes caffeine-containing beverages after 18:00 and is unwilling to forego caffeine after 18:00 for the duration of his/her participation in the study
- 10. History of drug or alcohol dependency or abuse within approximately the previous 2 years
- 11. Reports habitually consuming more than 14 drinks containing alcohol per week (females) or more than 21 drinks containing alcohol per week (males), or habitually consumes alcohol within the 3 hours before bedtime and unwilling to limit alcohol intake to no more than 2 drinks per day or forego having alcohol within the 3 hours before bedtime for the duration of his/her participation in the study
- 12. Known to be positive for human immunodeficiency virus
- 13. Active viral hepatitis (B or C) as demonstrated by positive serology at Screening
- 14. A prolonged QT/QTcF interval (QTcF > 450 ms) as demonstrated by a repeated ECG at Screening (repeated only if initial ECG indicates a QTcF interval >450 ms)
- 15. Current evidence of clinically significant disease (eg, cardiac; respiratory including chronic obstructive pulmonary disease, acute and/or severe respiratory depression; gastrointestinal including severe hepatic impairment; renal including severe renal impairment; neurological including myasthenia gravis; psychiatric disease; malignancy within the past 5 years other than adequately treated basal cell carcinoma) or chronic pain that in the opinion of the investigator(s) could affect the subject's safety or interfere with the study assessments, including the ability to perform tasks on the cognitive PAB. Subjects for whom a sedating drug would be contraindicated for safety reasons because of the subject's occupation or activities are also excluded. (revised per Amendment 01)
- 16. Comorbid nocturia resulting in frequent need to get out of bed to use the bathroom during the night
- 17. Any history of a medical or psychiatric condition that in the opinion of the investigator(s) could affect the subject's safety or interfere with the study assessments, including the ability to perform the PAB

Eisai 

- 18. Any suicidal ideation with intent with or without a plan, at the time of or within 6 months before the eC-SSRS administration during the Prerandomization Phase (ie, answering "Yes" to questions 4 or 5 on the Suicidal Ideation section of the eC-SSRS)
- 19. Any suicidal behavior in the past 10 years (per the Suicidal Behavior section of the eC-SSRS) (revised per Amendment 02)
- 20. Scheduled for surgery during the study
- 21. Used any prohibited prescription or over-the-counter concomitant medications within 1 week or 5 half-lives, whichever is longer, before the first dose of study medication (Run-in Period). (revised per Amendment 01) (A list of prohibited concomitant medications is presented in Appendix 3)
- 22. Used any modality of treatment for insomnia, including cognitive behavioral therapy or marijuana within 1 week or 5 half-lives, whichever is longer, before the first dose of study medication (Run-in Period) (revised per Amendment 01)
- 23. Failed treatment with suvorexant (Belsomra®) (efficacy and/or safety) following treatment with an appropriate dose and of adequate duration in the opinion of the investigator
- 24. Transmeridian travel across more than 3 time zones in the 2 weeks before Screening, or between Screening and Baseline, or plans to travel across more than 3 time zones during the study
- 25. A positive drug test at Screening, Run-In, or Baseline, or unwilling to refrain from use of recreational drugs during the study
- 26. Hypersensitivity to the study drugs (lemborexant or zolpidem) or to their excipients
- 27. Currently enrolled in another clinical trial or used any investigational drug or device within 30 days or 5× the half-life, whichever is longer preceding informed consent
- 28. Previously participated in any clinical trial of lemborexant

# 9.3.3 Removal of Subjects From Therapy or Assessment

The investigator may withdraw the subject from the study at any time for safety or administrative reasons. The subject may stop study drug or withdraw from the study at any time for any reason.

A subject who discontinues study treatment should return for an ET Visit as soon as possible. The primary reason for discontinuation and all other reason(s) contributing to the subject's discontinuation from study drug(s) should be collected on the Subject Disposition electronic case report form (eCRF). In addition, the date of last dose of study drug(s) will be recorded.

## 9.4 Treatment(s)

## 9.4.1 Treatment(s) Administered

## Test drug

Lemborexant 5 mg, lemborexant 10 mg or lemborexant-matched placebo will be taken orally in tablet form at home each night for 30 consecutive nights, immediately before the time the subject intends to try to sleep.

## Comparator drug

Zolpidem tartrate extended release 6.25 mg (Ambien CR®) or zolpidem-matched placebo will be taken orally in tablet form at home each night for 30 consecutive nights, immediately before the time the subject intends to try to sleep. The full Prescribing Information for Ambien CR will be provided to sites. (revised per Amendments 01 and 02)

#### Run-in Period

All subjects will receive 1 lemborexant-matched placebo tablet and 1 zolpidem-matched placebo tablet in a single-blind manner during the Run-in Period.

#### **Treatment Period**

During the Treatment Period, all subjects will receive 2 tablets as described below according to the treatment arm to which the subject has been randomized:

- LEM5: 1 zolpidem-matched placebo tablet and 1 lemborexant 5 mg tablet
- LEM10: 1 zolpidem-matched placebo tablet and 1 lemborexant 10 mg tablet
- ZOL: 1 zolpidem 6.25 mg tablet and 1 lemborexant-matched placebo tablet
- PBO: 1 zolpidem-matched placebo tablet and 1 lemborexant-matched placebo tablet

## 9.4.2 Identity of Investigational Product(s)

The sponsor will provide lemborexant tablets in strengths of 5 mg, 10 mg and lemborexant-matched placebo, identical in appearance. The comparator, zolpidem, will be obtained from commercial sources as zolpidem tartrate extended release 6.25 mg (Ambien CR 6.25) tablets, and the sponsor will provide placebo tablets identical in appearance to the zolpidem tablets. Tablets will be packaged in child-resistant blister cards in a double-blind manner.

Each subject will be dispensed a single card at the beginning of the Run-in Period and on Day 3. The subject will take 2 tablets a day; a single lemborexant or lemborexant-matched placebo tablet and a single zolpidem or zolpidem-matched placebo tablet. The placebo run-in card will contain a 17-day supply of lemborexant-matched placebo and zolpidem-matched placebo tablets per day. Each card for the Treatment Period will contain a 35-day supply of

Eisai 

tablets of either lemborexant or lemborexant-matched placebo and either zolpidem or zolpidem-matched placebo depending on the dose, in double-blind, double-dummy fashion.

#### 9.4.2.1 Chemical Name, Structural Formula of E2006/Lemborexant

• Test drug code: E2006

• Generic name: lemborexant

• Chemical name: (1R,2S)-2-{[(2,4-Dimethylpyrimidin-5-yl)oxy]methyl}-2-(3-fluorophenyl)-N-(5-fluoropyridin-2-yl)cyclopropanecarboxamide

• Molecular formula: C22H20F2N4O2

Molecular weight: 410.42

## 9.4.2.2 Comparator Drug

Zolpidem tartrate extended release 6.25 mg (Ambien CR 6.25)

Placebos to match lemborexant or zolpidem tartrate extended release 6.25 mg

## 9.4.2.3 Labeling for Study Drug

Lemborexant and zolpidem will be labeled in accordance with text that is in full regulatory compliance with each participating country and is translated into the required language(s) for each of those countries.

The following information has to be provided:

- For clinical trial use only
- Name and address of the sponsor
- Chemical name/drug identifier
- Lot number/batch number
- Storage conditions, expiration date if necessary

### 9.4.2.4 Storage Conditions

Study drug will be stored in accordance with the labeled storage conditions. Temperature monitoring is required at the storage location to ensure that the study drug is maintained within an established temperature range. The investigator is responsible for ensuring that the temperature is monitored throughout the total duration of the study and that records are maintained; the temperature should be monitored continuously by using either an in-house validated data acquisition system, a mechanical recording device, such as a calibrated chart recorder, or by manual means, such that minimum and maximum thermometric values over a specific time period can be recorded and retrieved as required.

## 9.4.3 Method of Assigning Subjects to Treatment Groups

At Baseline, subjects will be randomized, in a double-blind manner, to receive LEM5, LEM10, ZOL, or PBO in a 5:5:5:4 ratio. Randomization will be stratified by country and by age group (55 to 64 years; 65 years or older). Randomization to study treatments will be based on a computer-generated randomization scheme that will be reviewed and approved by an independent statistician. The randomization scheme and identification for each subject will be included in the final clinical study report for this study.

Randomization will be performed centrally by an interactive voice and web response system (IxRS). The IxRS or clinical supply vendor will generate the randomized blister card identification numbers. At enrollment (and after successful completion of study procedures the morning of Day 1), the investigator or designee will call the IxRS to register the subject information. At Randomization (morning of Day 1), the IxRS will assign each subject a unique 6-digit randomization number.

## 9.4.4 Selection of Doses in the Study

In Study 201, all doses studied met the first primary objective of balancing significant efficacy as measured by change from baseline in SE with sufficient safety measured by subjective sleepiness reported on the KSS. The second primary objective was also achieved, as there were no significant increases in the KSS at 1 hour after waketime at the end of treatment. However, there were dose-related increases in the KSS at both the beginning and end of treatment, and the rate of AEs of somnolence also increased with increasing dose level.

In Study 201, lemborexant 5 mg and 10 mg showed significant efficacy measured by SE, as well as decreases in sleep onset latency. These effects were maintained across the 15-day Treatment Period. For sleep maintenance, lemborexant 10 mg showed significant decreases, and while the magnitude of decreases in WASO was less for 5 mg, there was a significant proportion of subjects whose WASO decreased substantially, providing evidence for clinical benefit of 5 mg on sleep maintenance as well.

Because of the observed dose-related increases in subjective sleepiness and AEs of somnolence in Study 201, Study 107 was conducted to obtain additional information about the risk of clinically meaningful morning residual sleepiness. The study assessed average sleep onset latency on the M-MSLT after a single dose of LEM5 or LEM10 versus PBO. The results indicated that the pre-specified threshold for a clinically meaningful decrease in average sleep onset latency was not met by either the 5 mg or 10 mg dose level of lemborexant, supporting their use in the Phase 3 clinical trials. Taken together with the efficacy and safety results for lemborexant 5 mg and 10 mg in the Phase 2 study, these dose levels were selected for the current study.

Regarding ZOL, the FDA-approved doses of Ambien CR are 6.25 mg (recommended dose for women and elderly patients) and 12.5 mg (highest recommended dose for non-elderly patients). In the present study, only the 6.25 mg dose of ZOL will be administered. Of note is that a maximum of 40% of the study sample will be in the age range of 55 to 64 years old, and stratification by age will be implemented to ensure that approximately 60% will be

Eisai 

65 years or older. All of the subjects in the 55 to 64 years age group will be females. (revised per Amendment 03)

## 9.4.5 Selection and Timing of Dose for Each Subject

Throughout the Run-in Period and the Treatment Period, study drug will be taken immediately before the subject intends to sleep. When the subject is to sleep in the clinic for PSG, study personnel will administer study drug. On other nights, the subject will take study drug at home on as consistently a time schedule as possible. Subjects should not eat a meal within 3 hours before taking the study drug.

#### 9.4.6 Blinding

During the Run-in Period of the Prerandomization Phase, single blinding will be in effect such that the subject will be blinded to study treatment but study personnel will not be blinded. During the Randomization Phase, subjects and all personnel involved with the conduct and interpretation of the study, including investigators, site personnel, and sponsor staff will be blinded to the treatment codes. Randomization data will be kept strictly confidential, filed securely by an appropriate group with the sponsor or CRO and accessible only to authorized persons (eg, Eisai Global Safety) until the time of unblinding, per standard operating procedure.

A master list of all treatments and the subject numbers associated with them will be maintained in a sealed envelope by the clinical supply vendor, the IxRS vendor, and the sponsor. In the event that emergency conditions require knowledge of the study treatment given, the blind may be broken via the code breaker facility within the IxRS. Emergency procedures for revealing drug codes are given in Section 9.5.4.5. If possible, before breaking the blind, the investigator should consult with the sponsor to ascertain the necessity of breaking the code.

Disclosure of information from the interim analysis (Section 9.7.3) will be limited as detailed in the Interim Analysis charter. No individuals involved with the conduct of the study will have access to this information.

## 9.4.7 Prior and Concomitant Therapy

## 9.4.7.1 Drug-Drug Interactions

Not applicable

#### 9.4.7.2 Prohibited Concomitant Therapies and Drugs

Caffeine will be permitted in limited quantities during the study. Subjects will be advised to limit caffeine consumption to  $\leq 4$  cups of caffeinated beverages per day, or  $\leq 400$  mg caffeine per day. They will be instructed to avoid caffeine after 13:00 on days when they are scheduled for a PSG recording and after 18:00 on all other days during the study.

Eisai 

Alcohol will be permitted in limited quantities during the study. Subjects may consume a maximum of 2 alcoholic drinks on any day during the study, and will be advised not to consume any alcohol within 3 hours before bedtime. They must not consume alcohol on any days when they are scheduled for a PSG recording. Compliance with these restrictions will be monitored via questions on the Sleep Diary. If subjects cannot comply after an infraction and counseling, they may be discharged from the study.

Prohibited medications include strong and moderate CYP3A inhibitors and all CYP3A inducers. Prohibited therapies also include any treatment for insomnia disorder, including any drugs or non-pharmacological treatment such as cognitive behavioral therapy; medications that are used for the purpose of inducing sleep (hypnotics) or inducing wakefulness (stimulants; except caffeine; see above) and medications that have known sedating effects or alerting effects. This prohibition applies even if the entire class to which that medication belongs is not prohibited (eg, anticonvulsants).

A subject must discontinue any prohibited medication (Appendix 3) at least 1 week (or at least 5 half-lives, whichever is longer) before starting the Sleep Diary, ie, at least 2 weeks before the start of the Run-In Period.

Prohibited therapies include treatments for insomnia disorder (drugs or non-pharmacological treatment such as cognitive behavioral therapy) and any medication which, in the opinion of the investigator, causes or exacerbates the subject's insomnia. (revised per Amendment 01)

If a medication is not on the list of prohibited medications but in the opinion of the investigator causes or exacerbates the subject's insomnia, it must not be used throughout the study. If a medication is not specified as prohibited but is in the same class as a medication that is listed in Appendix 3, and if the investigator is uncertain whether the medication has known sedating or alerting effects, the Medical Monitor must be consulted.

If a subject starts any prohibited medication or therapy during the study, he/she must discontinue from the study, with the exception that certain prohibited medications may be used for a short duration (not to exceed 2 weeks) to treat an acute condition if this is agreed with the Medical Monitor. Note that strong CYP3A inhibitors will not be permitted at any time for any duration of use during the study. (revised per Amendment 01)

Any medication (including over-the-counter medications) or therapy administered to the subject within the last 3 months before Screening (ie, Prior Medications) or during the study, starting on the date of informed consent, will be recorded on the Prior and Concomitant Medication eCRF or Non-Pharmacological Procedures eCRF. The investigator will record on the Adverse Event eCRF any AE for which the concomitant medication/therapy was administered. If the concomitant medication/therapy is being administered for a medical condition present at the time of entry into the study, the investigator will record the medical condition on the Medical History and Current Medical Conditions eCRF.

## 9.4.8 Treatment Compliance

Compliance will be assessed for each study drug by examination of blister packs returned to the investigator at the end of the Run-in and Treatment Periods.

Eisai 

All subjects will be reminded of the importance of taking study medication as directed, ie, the correct number of tablets every night within 5 minutes before bedtime, and they will be reminded that their bedtime should be the same throughout the study. Subjects will be told that following these instructions about taking study medication is important for the treatment to be effective. Compliance will be monitored closely and determined at specific visits by tablet count. Tablets will be counted separately for tablets that are matched to lemborexant and tablets that are matched to zolpidem.

When subjects arrive for the first screening/baseline PSG during the Run-in Period, and the treatment compliance check indicates that a subject has missed any doses, the subject will be counseled by site personnel. If the subject has missed more than 1 dose, and given that the subject continues to meet eligibility criteria, the investigator must consult with the sponsor prior to the subject being randomized and come to a collaborative decision on whether the subject should continue in the study. When subjects arrive for Baseline, and the treatment compliance check indicates that a subject has missed any doses, the investigator must use clinical judgment to decide if the subject should continue in the study.

Records of treatment compliance for each subject will be kept during the study. Clinical research associates will review treatment compliance during site visits and at the completion of the study.

# 9.4.9 Drug Supplies and Accountability

In compliance with local regulatory requirements, drug supplies will not be sent to the investigator until the following documentation has been received by the sponsor:

- A signed and dated confidentiality agreement
- A copy of the final protocol signature page, signed and dated by both the sponsor and investigator
- Written proof of approval of the protocol, the ICFs, and any other information provided to the subjects by the IRB/IEC for the institution where the study is to be conducted
- A copy of the IRB/IEC-approved ICF and any other documentation provided to the subjects to be used in this study
- The IRB/IEC membership list and statutes or Health and Human Services Assurance number
- A copy of the certification and a table of the normal laboratory ranges for the reference laboratory conducting the clinical laboratory tests required by this protocol
- An investigator-signed and dated Form FDA 1572
- Financial Disclosure form(s) for the PI and all subinvestigators listed on Form FDA 1572
- A signed and dated curriculum vita of the PI including a copy of the PI's current medical license or medical registration number on the curriculum vitae
- A signed and dated clinical studies agreement
- A copy of the regulatory authority approval for the country in which the study is being conducted (if required), and the Import License (if required)

Eisai 

The investigator and the study staff will be responsible for the accountability of all study drugs (dispensing, inventory, and record keeping) following the sponsor's instructions and adherence to GCP guidelines as well as local or regional requirements.

Under no circumstances will the investigator allow the study drugs to be used other than as directed by this protocol. Study drugs will not be dispensed to any individual who is not enrolled in the study.

The site must maintain an accurate and timely record of the following receipt of all study drugs, dispensing of study drugs to the subject, collection and reconciliation of unused study drugs/ that are either returned by the subjects or shipped to site but not dispensed to subjects, and return of reconciled study drugs to the sponsor. This includes, but may not be limited to: (a) documentation of receipt of study drugs/, (b) study drugs, dispensing, and return reconciliation log, (c) study drug accountability log, (d) all shipping service receipts, (e) documentation of returns to the sponsor, and (f) certificates of destruction for any destruction of study drugs/ that occurs at the site. All forms will be provided by the sponsor. Any comparable forms that the site wishes to use must be approved by the sponsor.

The study drugs/ and inventory records must be made available, upon request, for inspection by a designated representative of the sponsor or a representative of a health authority (eg, FDA; Medicine and Healthcare products Regulatory Agency. As applicable, all unused study drugs/ and empty and partially empty containers from used study drugs/ are to be returned to the investigator (or if regionally required, the head of the medical institution or the designated pharmacist) by the subject and, together with unused study drugs/ that were shipped to the site but not dispensed to subjects, are to be returned to the sponsor's designated central or local depot(s) during the study or at the conclusion of the study. Upon completion of drug accountability and reconciliation procedures by the site's personnel and documentation procedures by the sponsor's personnel, study drugs/ that are to be returned to the sponsor's designated central or local depot(s) must be boxed, sealed, and shipped back to the central or local depot(s) following all local regulatory requirements. In some regions, study drugs/ may be removed from the site and hand delivered to the central or local depot by sponsor representatives.

Drug accountability will be reviewed during site visits and at the completion of the study.

Study sites are also responsible for tracking receipt, distribution, and return of all study equipment (eg, Sleep Diary devices) to the sponsor or designated entity.

# 9.5 Study Assessments

#### 9.5.1 Assessments

#### 9.5.1.1 Demography

Subject demographic information will be collected at the Screening Visit. Demographic information will include date of birth, sex, and race/ethnicity (where allowed). In applicable countries, to protect personal data, only the year of birth will be collected, and the month and

Eisai 

date of each subject's date of birth will be masked where necessary as January 1. (revised per Amendment 01)

#### 9.5.1.2 Baseline Assessments

#### 9.5.1.2.1 MEDICAL HISTORY AND PHYSICAL EXAMINATIONS

Sleep, medical, and psychiatric history and current medical conditions will be recorded at the Screening Visit. All sleep, medical, and psychiatric history within 5 years must be noted in the Medical History and Current Medical Conditions eCRF. If a subject has a score of 11-15 on the ESS at Screening, then the presence of excessive daytime sleepiness must be recorded in the subject's Medical History. Note that the presence of excessive daytime sleepiness in a subject's Medical History, combined with the definition of Adverse Event as specified in Section 9.5.1.5.3 means that only a worsening in daytime sleepiness during the study should be reported as an Adverse Event. (revised per Amendment 02)

Physical examinations (full or brief) will be performed as described in Section 9.5.1.5.7.

#### 9.5.1.2.2 SLEEP DISORDERS HISTORY AND SCREENING BATTERY

The SDSB will be administered only at the Screening Visit, and will include the:

- StopBANG: a list of eight questions to be answered Yes or No, which screens potential subjects for obstructive sleep apnea (Chung et al., 2008)
- IRLS: a subjective scale comprising ten questions, which measures disease of symptoms of restless legs syndrome (Abetz et al., 2006)
- ESS: a questionnaire that asks subjects to rate their probability of falling asleep, on a scale of increasing probability from 0 to 3 for eight different situations that most people engage in during their daily lives, which assesses the severity of daytime sleepiness (Johns, 1992)
- MUPS: a scale comprising 21 questions asking whether the subject has experienced phenomena related to International Classification of Sleep Disorders Version 2 classified parasomnias (eg, enuresis, sleepwalking, sleep paralysis) along with a time frame for occurrences of these experiences ranging from within past month to lifetime and frequency within the time frame ranging from occasionally to almost every night (Fulda et al., 2008). An adapted version will be used. (revised per Amendment 01)

#### 9.5.1.2.3 BECK DEPRESSION INVENTORY - II

The BDI-II is a 21-question multiple-choice self-report questionnaire that subjects will use to rate the presence, frequency, and severity of symptoms of depression using a 4-point Likert scale (Beck, et al., 1961). Scores on the BDI-II may range from 0 to 63, with higher scores indicating higher levels of depressive symptoms. Subjects with BDI-II scores greater than 19 will be excluded from participation.

Eisai 

#### 9.5.1.2.4 BECK ANXIETY INVENTORY

The BAI is a 21-question multiple-choice self-report inventory that subjects will use to rate the presence, frequency, and severity of symptoms of anxiety using a 4-point Likert scale (Beck, et al., 1988). Scores on the BAI may range from 0 to 63, with higher scores indicating higher levels of anxiety symptoms. Subjects with scores on the BAI greater than 15 will be excluded from participation.

#### 9.5.1.3 Efficacy Assessments

#### 9.5.1.3.1 POLYSOMNOGRAPHY

Each PSG recording will include an electrode montage with electroencephalography (EEG), electromyography (EMG), electrooculography, and ECG channels, for scoring of sleep parameters and sleep architecture via standard sleep scoring criteria. In addition, the screening PSG will include channels for assessment of symptoms of sleep apnea and periodic limb movement disorder.

Trained PSG scorers will score PSG records in 30-second epochs according to standard criteria. The PSG at the second screening visit will be used only to calculate the Apnea-Hypopnea Index and the Periodic Limb Movements with Arousal Index for evaluation of eligibility criteria; sleep parameters and sleep architecture will not be evaluated from this PSG. The 2 PSGs obtained during the Run-in Period will be used to a) determine eligibility and b) derive baseline PSG parameters for those subjects who are randomized.

All PSG parameters will be obtained separately for each PSG recording and averaged across the pairs of consecutive PSG nights.

The following parameters will be derived from all PSGs:

- LPS: minutes from lights off to the first epoch of 20 consecutive epochs of non-wakefulness
- SE: proportion of time spent asleep per TIB, calculated as TST/interval from "lights off" until "lights on"
- WASO: minutes of wake from the onset of persistent sleep until lights on
- WASO2H: minutes of wake during the interval from 240 minutes after lights off until lights on
- TST: minutes of sleep from sleep onset until terminal awakening
- Mean duration of long awakenings (DurLongAw): average duration of all long awakenings (with long awakening defined as 10 or more consecutive epochs [ie, 5 minutes or longer] scored as wake or N1, initiated with at least 1 epoch of wake, after onset of persistent sleep, and including any terminal awakening

Additional sleep architecture parameters will also be calculated from each PSG, including:

- Sleep onset latency: minutes from lights off to the first epoch of any stage of sleep (N1, N2, N3, REM) (revised per Amendment 01)
- Number of awakenings after persistent sleep, with an awakening defined as at least 2 consecutive epochs of wakefulness; an awakening cannot be interrupted by stage N1, but must be interrupted by stage N2, N3, or REM
- Number of long awakenings
- WASO1H (wake after sleep onset in the first half of the night): minutes of wake during the interval from onset of persistent sleep until 240 minutes after lights off (revised per Amendment 03)
- Percentage of sleep stages per TIB: wake, non-REM (NREM) sleep (stages N1, N2, N3 separately and combined), REM sleep
- Minutes of sleep stages per TIB: wake, NREM sleep (stages N1, N2, N3), REM sleep
- Percentage of sleep stages per TST: wake, NREM sleep (stages N1, N2, N3 separately and combined), REM sleep
- Minutes of sleep stages per TST: wake, NREM sleep (stages N1, N2, N3), REM sleep
- REM episode frequency and duration
- Mean REM/NREM cycle duration
- REM latency: minutes from first epoch of sleep (N1, N2, or N3) to first epoch of REM (revised per Amendment 01)

Each of these PSG-derived variables, with the exceptions of SE, REM episode frequency and duration, mean REM/NREM cycle duration, and REM latency, will also be calculated by hour and by half of the 8-hour time interval in bed.

#### 9.5.1.3.2 ELECTRONIC SLEEP DIARY

The Sleep Diary will be completed within an hour of morning waketime on each morning of the study from Screening through the end of the Follow-Up Period. Sleep Diary entries may be maintained in paper format as a backup to the electronic Sleep Diary, if necessary. This diary will yield several self-reported measures of sleep that will be used to determine eligibility, as well as to assess efficacy and safety. (revised per Amendment 02)

Subjects must comply with requirements for completion of the Sleep Diary. Failure to comply will require discussion with the Medical Monitor and may result in discontinuation of the subject from the study.

#### Sleep Parameters

- Subjective Sleep Onset Latency (sSOL): estimated minutes from the time that the subject attempts attempting to sleep until sleep onset
- Subjective Wake After Sleep Onset (sWASO): sum of estimated minutes of wake during the night after initial sleep onset until the time the subject stops trying to sleep for the night

Eisai 

- Subjective Total Sleep Time (sTST): derived minutes of sleep from sleep onset until the time the subject stops trying to sleep for the night
- Subjective Sleep Efficiency (sSE): proportion of sTST per subjective time spent in bed, calculated as the interval from the time that subject reports attempting to sleep until the time the subject stops trying to sleep for the night, and time spent asleep derived from subjective time spent in bed minus sWASO

## Quality of Sleep

The Sleep Diary will also include items assessing sleep quality and morning sleepiness/alertness.

The Sleep Diary will also be used to assess the subject's perception of the quality of sleep on the previous night with the following question: "How would you rate the quality of your sleep last night?" Subjects will rate the quality of their sleep on a scale from 1 to 9, with 1 being extremely poor and 9 being extremely good.

## Morning Sleepiness

The Sleep Diary will also be used to assess subjective ratings of morning sleepiness with the following question: "How alert/sleepy do you feel this morning?" Subjects will rate their sleepiness/alertness level on a scale from 1 to 9, with 1 being extremely sleepy and 9 being extremely alert. (revised per Amendment 03)

The morning sleepiness question that is part of the electronic Sleep Diary will also be asked verbatim, using a paper-and-pencil format, at 1.5 hours after waketime each morning the subjects is in the clinic following a PSG recording. The rating on this question will be taken into consideration by the investigator when making the determination about whether it is safe for the subject to be discharged from the clinic.

## **Alcohol Consumption**

The Sleep Diary will include questions that ask whether or not the subject consumed alcohol the previous day within 3 hours before bedtime or exceeded the daily maximum of 2 alcoholic drinks. (revised per Amendment 01)

#### 9.5.1.3.3 INSOMNIA SEVERITY INDEX

The ISI is a 7-item self-report questionnaire assessing the nature, severity and impact of insomnia (Bastien et al., 2001). The dimensions evaluated are: severity of sleep onset, sleep maintenance, early morning awakening problems; sleep dissatisfaction; interference of sleep difficulties with daytime functioning, noticeability of the sleep problems by others; and distress caused by the sleep difficulties. A 5-point Likert scale is used to rate each item (from 0 = 1 no problem to 0 = 1 no problem

Eisai 
#### 9.5.1.3.4 FATIGUE SEVERITY SCALE

The FSS is a self-report scale on which subjects are instructed to choose a number from 1 to 7 that indicates their degree of agreement with each of 9 statements about their fatigue where "1" indicates strongly disagree and "7", strongly agree. The FSS score is the sum of all responses to the 9 questions (Schwartz et al., 1993). Higher scores indicate greater fatigue.

# 9.5.1.4 Pharmacokinetic, Pharmacodynamic, Pharmacogenomic, and Other Biomarker Assessments

#### 9.5.1.4.1 PHARMACOKINETIC ASSESSMENTS

At predefined visits, a single, 4-mL blood sample per timepoint to determine plasma concentrations of lemborexant and its metabolites (M4, M9, and M10) or zolpidem will be taken and will be processed according to instructions in a laboratory manual to be provided to the study sites. Plasma concentrations will be using validated liquid chromatography-tandem mass spectrometry assay methods. Concentrations of zolpidem will be determined only on an as needed basis as determined by the Study Director or Medical Monitor. The time and date of the 2 most recent doses preceding the samples obtained on Day 2 and Day 30 will be documented. (revised per Amendment 01)

#### 9.5.1.4.2 PHARMACODYNAMIC ASSESSMENTS

# Postural Stability using the CDR Posture Assessment

Postural stability will be assessed using an apparatus similar to the Wright ataxiameter, and referred to as the CDR posture device. This device measures directional trunk movements (ie, body sway) through a cord placed around the subject's waist and connected to the ataxiameter. On the evening of the Screening PSG visit, subjects will be introduced to the CDR posture assessment. Subjects will stand on a firm surface with feet comfortably apart, either barefoot or wearing socks. The standing position (inside heel-to-inside heel distance) and barefoot/socks conditions will be documented to ensure they remain the same for a given subject at each postural stability assessment timepoint. They will be instructed to stand as still as possible with eyes closed for 1 minute. (revised per Amendment 01) On the morning after the Screening PSG, subjects will complete a CDR posture assessment session for familiarization purposes only; no data from this session will be used for analyses. This session must be conducted under the same conditions (eg, starting within 5 minutes of morning waketime, at bedside) as during the testing sessions at subsequent visits.

Body sway is detected through the cable around the subject's waist by the ataxiameter and these data are transmitted to a laptop. Body sway is measured in units of  $1/3^{\circ}$  of the angle of arc. For ease in reporting these will be called arbitrary units, with a higher number indicating more body sway (less postural stability).

Eisai 

# Cognitive Performance Assessment Battery

A computerized PAB will be administered on a laptop computer after the postural stability test. (revised per Amendment 01) While completing the PAB, subjects will be in bed and ambient lighting will be maintained at a level of 80 to 100 lux at the subject's eye level. On the evening of the Screening PSG visit, before bedtime, subjects will be introduced to the PAB tasks and will undergo a minimum of 2 training sessions. If subjects cannot adequately perform the tasks during the training sessions, they will be excluded from further participation. On the morning after the Screening PSG, subjects will complete a session of the cognitive PAB for familiarization purposes only; no data from this session will be used for analyses. This session must be conducted under the same conditions (eg, lighting, subject in bed) as during the testing sessions at subsequent visits.

The PAB comprises 9 tasks, including Simple Reaction Time, Choice Reaction Time, Digit Vigilance, Immediate Word Recall, Delayed Word Recall, Word Recognition, Picture Recognition, Numeric Working Memory, and Spatial Working Memory. The full PAB will take approximately 18 to 30 minutes to complete. Four composite domain factor scores are calculated by combining outcome variables from the various tests, as described below:

## • Power of Attention

- o A composite score from the speed scores of 3 tests of attention
- o Reflects the ability to focus attention and process information
- Continuity of Attention
  - A composite score created by combining the accuracy scores from the tests of attention
  - o Reflects the ability to sustain attention (vigilance)
- Quality of Memory
  - A composite score created by combining the accuracy measures from the two tests of working memory and the four tests of episodic memory
  - o Reflects the ability to store information in memory and subsequently retrieve it
- Speed of Memory Retrieval
  - A composite score created by combining the reaction time scores from the two working memory tests and the two episodic recognition tests
  - o Reflects time taken to retrieve information held in both working and episodic memory

#### 9.5.1.4.3 PHARMACOGENOMIC ASSESSMENTS

Not applicable

#### 9.5.1.4.4 OTHER BIOMARKER ASSESSMENTS

Not applicable.

# 9.5.1.5 Safety Assessments

Safety assessments will consist of monitoring and recording all AEs; regular laboratory evaluation for hematology, blood chemistry, and urine values; periodic measurement of vital signs, weight and ECGs; and the performance of physical examinations. Safety will be assessed at every clinic visit throughout the study, and at the EOS Visit.

## 9.5.1.5.1 COLUMBIA-SUICIDE SEVERITY RATING SCALE

Suicidality will be assessed using a self-rated electronic version of the eC-SSRS (Posner et al., 2011). The eC-SSRS assesses an individual's degree of suicidality, including both suicidal ideation and suicidal behavior. Qualified personnel must evaluate positive responses on the eC-SSRS and take appropriate action as detailed in the training and certification process for administering the eC-SSRS.

#### 9.5.1.5.2 Tyrer Benzodiazepine Withdrawal Symptom Questionnaire

An assessment of withdrawal symptoms will be made using the T-BWSQ (Tyrer et al., 1990) to be completed at the EOS Visit. Subjects will be asked about the presence/absence and severity of the symptoms listed in the questionnaire. For each listed symptom, the subject is to respond "No" (Score = 0), "Yes – moderate" (Score = 1) or "Yes – severe" (Score = 2). The sum of responses will be the subject's score. (revised per Amendment 02)

## 9.5.1.5.3 ADVERSE EVENTS

An AE is any untoward medical occurrence in a patient or clinical investigation subject administered an investigational product. An AE does not necessarily have a causal relationship with the medicinal product. For this study, the study drug is lemborexant.

The criteria for identifying AEs in this study are:

- Any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational product, whether or not considered related to the investigational product (Note: Every sign or symptom should not be listed as a separate AE if the applicable disease [diagnosis] is being reported as an AE)
- Any new disease or exacerbation of an existing disease
- Any deterioration in nonprotocol-required measurements of a laboratory value or other clinical test (eg, ECG or x-ray) that results in symptoms, a change in treatment, or discontinuation of study drug
- Recurrence of an intermittent medical condition (eg, headache) not present pretreatment (Baseline)

An abnormal laboratory test result should be considered an AE if the identified laboratory abnormality leads to any type of intervention, withdrawal of study drug, or withholding of study drug, whether prescribed in the protocol or not

Eisai 

All AEs observed during the study will be reported on the eCRF. All AEs, regardless of relationship to study drug or procedure, should be collected beginning from the time the subject signs the study ICF through the last visit. Serious adverse events (SAEs) will be collected for 28 days after the last dose.

Abnormal laboratory values should not be listed as separate AEs if they are considered to be part of the clinical syndrome that is being reported as an AE. It is the responsibility of the investigator to review all laboratory findings in all subjects and determine if they constitute an AE. Medical and scientific judgment should be exercised in deciding whether an isolated laboratory abnormality should be classified as an AE. Any laboratory abnormality considered to constitute an AE should be reported on the Adverse Event eCRF.

Abnormal ECG (QTcF) results, if not otherwise considered part of a clinical symptom that is being reported as an AE, should be considered an AE if the QTcF interval is more than 450 msec and there is an increase of more than 60 msec from baseline. Any ECG abnormality that the investigator considers as an AE should be reported as such.

It is the responsibility of the investigator to review the results of the eC-SSRS in all subjects and determine if any result constitutes an AE. Medical and scientific judgment should be exercised in deciding whether an isolated suicidality rating scale response should be classified as an AE (see Section 9.5.1.5 for a description of the eC-SSRS).

AEs in clinical investigation subjects include any change in the subject's condition. This includes symptoms, physical findings, or clinical syndromes. All AEs encountered during the clinical study will be reported on the eCRF.

All AEs must be followed for 28 days after the subject's last dose, or until resolution, whichever comes first.

Every effort must be made by the investigator to categorize each AE according to its severity and its relationship to the study treatment.

#### ASSESSING SEVERITY OF ADVERSE EVENTS

AEs will be graded on a 3-point scale (mild, moderate, severe) and reported in the detail indicated on the eCRF. The definitions are as follows:

Mild Discomfort noticed, but no disruption of normal daily activity

Moderate Discomfort sufficient to reduce or affect normal daily activity

Severe Incapacitating, with inability to work or to perform normal daily activity

The criteria for assessing severity are different than those used for seriousness (see Section 9.5.1.5.4) for the definition of an SAE).

#### ASSESSING RELATIONSHIP TO STUDY TREATMENT

Items to be considered when assessing the relationship of an AE to the study treatment are:

- Temporal relationship of the onset of the event to the initiation of the study treatment
- The course of the event, especially the effect of discontinuation of study treatment or reintroduction of study treatment, as applicable
- Whether the event is known to be associated with the study treatment or with other similar treatments
- The presence of risk factors in the study subject known to increase the occurrence of the event
- The presence of nonstudy, treatment-related factors that are known to be associated with the occurrence of the event

#### CLASSIFICATION OF CAUSALITY

The relationship of each AE to the study drug will be recorded on the eCRF in response to the following question:

Is there a reasonable possibility that the study drug caused the AE?

Yes (related) A causal relationship between the study drug and the AE is a reasonable possibility.

No (not related) A causal relationship between the study drug and the AE is not a reasonable possibility.

## 9.5.1.5.4 SERIOUS ADVERSE EVENTS AND EVENTS ASSOCIATED WITH SPECIAL SITUATIONS

An SAE is any untoward medical occurrence that at any dose:

- Results in death
- Is life-threatening (ie, the subject was at immediate risk of death from the AE as it occurred; this does not include an event that, had it occurred in a more severe form or was allowed to continue, might have caused death)
- Requires inpatient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity
- Is a congenital anomaly/birth defect (in the child of a subject who was exposed to the study drug)

Other important medical events that may not be immediately life-threatening or result in death or hospitalization but, when based on appropriate medical judgment, may jeopardize the subject or may require intervention to prevent one of the outcomes in the definition of

SAE listed above should also be considered SAEs. Medical and scientific judgment should be exercised in deciding whether expedited reporting is appropriate in such situations.

In addition to the above, events associated with special situations (EASS) include pregnancy or exposure to study drug through breastfeeding and AEs associated with study drug overdose, misuse, abuse, or medication error. These EASSs are to be captured using the SAE procedures but are to be considered as SAEs only if they meet one of the above criteria. All AEs associated with special situations are to be reported on the eCRF whether or not they meet the criteria for SAEs.

All SAEs must be followed to resolution or, if resolution is unlikely, to stabilization.

The following hospitalizations are not considered to be SAEs because there is no "AE" (ie, there is no untoward medical occurrence) associated with the hospitalization:

- Hospitalizations for respite care
- Planned hospitalizations required by the protocol
- Hospitalization planned before informed consent (where the condition requiring the hospitalization has not changed after study drug administration)
- Hospitalization for administration of study drug or insertion of access for administration of study drug
- Hospitalization for routine maintenance of a device (eg, battery replacement) that was in place before study entry

If possible, a blood sample for the measurement of study drug plasma concentration should be drawn at the first report of an SAE or a severe unexpected AE and at its resolution.

#### 9.5.1.5.5 LABORATORY MEASUREMENTS

Clinical laboratory tests are to be performed according to the schedule in Table 2. Blood and urine samples will be collected for the clinical laboratory tests as listed in Table 3. Subjects should be in a seated or supine position during blood collection.

Viral testing for hepatitis B and C will be conducted from a blood sample obtained at Screening. The specific test for hepatitis B is the surface antigen panel (HBsAg) with confirmation as needed. The specific tests for hepatitis C are the hepatitis C virus (HCV) antibody immunoglobulin G (IgG), with confirmation as needed using the HCV score. (revised per Amendment 01)

A 30-mL urine sample for assessment of drugs of abuse will be collected at designated time points as specified in the Schedule of Procedures/Assessments (Table 4). These samples will be tested for common drugs of use/abuse: eg, cocaine, cannabinoids, phencyclidine, opioids (as a group), benzodiazepines, barbiturates, and amphetamines. (revised per Amendment 01)

Eisai 

Table 2 Clinical Laboratory Tests

| Category | Parameters |
|---|---|
| Hematology | hematocrit, hemoglobin, platelets, RBC count, and WBC count with differential (bands, basophils, eosinophils, lymphocytes, monocytes, neutrophils) |
| Chemistry | |
| Electrolytes | bicarbonate, chloride, potassium, sodium |
| Liver function tests | alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, direct bilirubin, total bilirubin |
| Renal function parameters | blood urea/blood urea nitrogen, creatinine |
| Other | albumin, calcium, cholesterol, globulin, glucose, iron, lactate dehydrogenase, phosphorus, total protein, triglycerides, uric acid |
| Urinalysis | bacteria, casts, crystals, epithelial cells, glucose, ketones, occult blood, pH, protein, RBCs, specific gravity, WBCs |

RBC = red blood cell, WBC = white blood cell.

Table 3 Blood Sampling Schedule for All Laboratory and Pharmacokinetic Assessments

| | Volume per Sample<br>Collection<br>(mL) | Collection<br>Time Points | Window Around Time<br>Point | Volume<br>Collected<br>(mL) |
|---|---|---|---|---|
| Clinical laboratory tests | 12 <sup>a</sup> | Screening<br>Baseline<br>Day 31<br>EOS/ET | n/a | 48 |
| Viral tests | 6 <sup>a</sup> | Screening | n/a | 6 |
| PK sampling | 4 | Day 2 pm<br>Day 3 am<br>Day 30 pm<br>Day 31 am | pm: within 2 hours predose am: after PAB and within 1 hour after morning waketime | 16 |
| <b>Total Volume Collect</b> | cted | | | 70 |

EOS = end of study, ET = early termination, n/a = not applicable, PK = pharmacokinetic

Clinical laboratory tests during the study will be performed by a central laboratory. All blood and urine samples will be collected and sent to the central laboratory on the day of collection unless otherwise instructed. In cases of a safety concern, blood samples will be split (or two samples drawn) to allow a local laboratory analysis in addition to the central laboratory. Laboratory certification as available will be included in the final clinical study report for this study.

Eisai 

a. Estimated volume.

A laboratory abnormality may meet the criteria to qualify as an AE as described in this protocol (see Section 9.5.1.5.3) and the case report form (CRF) Completion Guidelines. In these instances, the AE corresponding to the laboratory abnormality will be recorded on the Adverse Event eCRF.

For laboratory abnormalities meeting the criteria of SAEs, the site must fax or email the SAE report including the laboratory report (as regionally required) to the sponsor using the SAE form (see Reporting of Serious Adverse Events, Section 9.5.4.1).

# 9.5.1.5.6 VITAL SIGNS AND WEIGHT MEASUREMENTS

Vital sign measurements (ie, systolic and diastolic blood pressure [BP] [mmHg], pulse [beats per minute], respiratory rate [per minute], and body temperature [in centigrade]) will be obtained at the visits designated in the Schedule of Procedures/Assessments (Table 4) by a validated method. Blood pressure and pulse will be measured after the subject has been in a sitting position for 5 minutes. All BP measurements should be performed on the same arm, preferably by the same person. Validated methods will be used for all vital sign measurements, and values will be recorded. Height (cm; once only) and weight (kg) will also be measured.

When vital signs are to be obtained concurrently with PK or other blood samples, the vital sign measurements will be performed before drawing blood samples in order to maximize the accuracy of blood sampling times while minimizing the potential effects of blood drawing on recordings obtained during safety assessments.

#### 9.5.1.5.7 PHYSICAL EXAMINATIONS

Physical examinations (full or brief) will be performed as designated in the Schedule of Procedures/Assessments Table 4). At Screening and at the end-of-study visit, a full physical examination will be conducted, including evaluation of the head, eyes, ears, nose, throat, neck, chest (including heart and lungs), abdomen, limbs, skin. The full physical examination will include a brief neurological examination to assess possible impairment in major functions (ie, motor, cerebellar, sensory, major pathological reflexes). A urogenital examination will only be required in the presence of clinical symptoms related to this region and at the discretion of the investigator. At other study visits as designated in Table 4, a brief physical examination will be conducted to assess health status by brief evaluation of the head, eyes, ears, nose, throat, heart, lungs, abdomen, and extremities, and other physical conditions of note. Documentation of the physical examinations, including the brief neurological examinations, will be included in the source documentation at the site. Only changes from screening physical examination findings that meet the definition of an AE will be recorded on the AE eCRF.

#### 9.5.1.5.8 ELECTROCARDIOGRAMS

Electrocardiograms will be obtained as designated in the Schedule of Procedures/Assessments (Table 4).

Eisai 

An ECG abnormality may meet the criteria of an AE as described in this protocol (see Section 9.5.1.5.3). In these instances, the AE corresponding to the ECG abnormality will be recorded on the Adverse Events eCRF.

For ECG abnormalities meeting criteria of an SAE (see Section 9.5.1.5.4), the site must fax or email the SAE report including the ECG report to the sponsor using the SAE form (see Reporting of Serious Adverse Events [Section 9.5.4.1]).

#### 9.5.1.5.9 OTHER ASSESSMENTS

## EQ-5D-3L

The EQ-5D-3L is a generic instrument that can be used in the clinical and economic evaluation of health care, and to collect data on quality of life and preferences/utility (Brooks et al., 1996). The instrument comprises questions on mobility, self-care, usual activities, pain/discomfort and anxiety/depression, and a visual analogue scale from 0 ("Worst imaginable health state") to 100 ("Best imaginable health state").

#### PATIENT GLOBAL IMPRESSION – INSOMNIA

The PGI-Insomnia questionnaire is a self-report assessment asking about a subject's perception of the effects of the study medication on their sleep relative to their sleep before entering in the study. As such, the PGI-Insomnia does not have a baseline and the outcome is not change from baseline, but rather the global impression of the study medication's effects at the end of treatment. The PGI-Insomnia has 3 items related to study medication effects (a: helped/worsened sleep, b: decreased/increased time to fall asleep, and c: increased/decreased TST) and 1 item related to perceived appropriateness of study medication strength. The first 3 items are answered on a 3-point scale (1=positive medication effect, 2=neutral medication effect, 3=negative medication effect) and the last item on a different 3-point scale (medication: 1=too strong, 2=just right, 3=too weak). Each item will be reported separately. This scale was used in studies of zolpidem (Roth et al., 2006; Walsh et al., 2008).

## 9.5.2 Schedule of Procedures/Assessments

#### 9.5.2.1 Schedule of Procedures/Assessments

Table 4 presents the schedule of procedures/assessments for this study.

Table 4 Schedule of Procedures/Assessments in Study E2006-G000-304

| Phase | Prerandomization | | | | | | | | Randomization | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Period | Scr | eening | Ţ, | | Ru | n-in | | BL | | | | Treat | tment | | | | Foll | low-Up ET <sup>e</sup> | | TINI |
| Visit | 1 | 2a | 2b | 3a | 3b | 4a <sup>a</sup> | 4b | 5a | 5b | 5c | 6a <sup>b</sup> | 6b | 7a | 7b | 8a <sup>c</sup> | 8b | | EOS <sup>d</sup> | E1 | UN |
| Target Study Day | -21 | -14 | -13 | -7 | -6 | -6 | -5 | 1 | 1 | 2 | 2 | 3 | 29 | 30 | 30 | 31 | | 44 | | |
| Window | -14/+4 | -3/ | +4 | -3/ | +3 | -3/ | +3 | | n/a | | n | /a | -2/ | +5 | -2/ | /+5 | | | | |
| Possible Study<br>Day(s) Given<br>Window | -35<br>to<br>-17 | -17<br>to<br>-10 | -16<br>to<br>-9 | -10<br>to<br>-4 | -9<br>am<br>to<br>-3<br>am | -9<br>pm<br>to<br>-3<br>pm | -8<br>to<br>-2 | 1 | 1<br>pm | 2<br>am | 2<br>pm | 3<br>am | 29<br>pm | 30<br>am | 30<br>pm | 31<br>am | 31<br>to<br>44 | 44 | | |
| Procedures/<br>Assessments | | | | | | | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | | | | | | |
| Informed consent | X | | | | | | | | | | | | | | | | | | | |
| Inclusion/exclusion criteria <sup>f</sup> | | | | | | | | > | | | | | | | | | | | | |
| Height | X | | | | | | | | | | | | | | | | | | | |
| Weight | X | | | | | | | X | | | | | | | | X | | X | X | |
| Clinical laboratory tests | X | | | | | | | X | | | | | | | | X | | X | X | X |
| Viral screening <sup>g</sup> | X | | | | | | | | | | | | | | | | | | | |
| Vital signs | X | | | | | | | X | | | | | | | | X | | X | X | X |
| 12-lead ECG | X | | | | | | | X | | | | | | | | X | | X | X | X |
| Sleep, medical, and psychiatric history | X | | | | | | | | | | | | | | | | | | | |
| ISI | X | | | X | | | | X | | | | | | | | X | | | | |
| $SDSB^h$ | X | | | | | | | | | | | | | | | | | | | |
| Physical exami | X | | | | | | | | | | | | | | | X | | X | X | X |
| Prior / concomitant | | | | | | | | | | | | | | | | | > | <u> </u> | | |

Eisai 

Table 4 Schedule of Procedures/Assessments in Study E2006-G000-304

| Phase | | | Prei | andon | nizatio | n | | | | | | | | Rand | lomiza | tion | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Period | Scr | eening | 5 | | Ru | n-in | | BL | | | | Trea | tment | | | | Fol | low-Up | ETe | UN |
| Visit | 1 | 2a | 2b | 3a | 3b | 4a <sup>a</sup> | 4b | 5a | 5b | 5c | 6a <sup>b</sup> | 6b | 7a | 7b | 8a <sup>c</sup> | 8b | | EOS <sup>d</sup> | L I | UN |
| Target Study Day | -21 | -14 | -13 | -7 | -6 | -6 | -5 | 1 | 1 | 2 | 2 | 3 | 29 | 30 | 30 | 31 | | 44 | | |
| Window | -14/+4 | -3/ | <b>/+4</b> | -3/ | <b>'+3</b> | -3/ | +3 | | n/a | | n | /a | -2/ | <b>/+5</b> | -2/ | /+5 | | | | |
| Possible Study<br>Day(s) Given<br>Window | -35<br>to<br>-17 | -17<br>to<br>-10 | -16<br>to<br>-9 | -10<br>to<br>-4 | -9<br>am<br>to<br>-3<br>am | -9<br>pm<br>to<br>-3<br>pm | -8<br>to<br>-2 | 1 | 1<br>pm | 2<br>am | 2<br>pm | 3<br>am | 29<br>pm | 30<br>am | 30<br>pm | 31<br>am | 31<br>to<br>44 | 44 | | |
| Procedures/<br>Assessments | | | | | | | | | | | | | | | | | | | | |
| medications | | | | | | | | | | | | | | | | | | | | |
| Beck Depression<br>Inventory II | X | | | | | | | | | | | | | | | | | | | |
| Beck Anxiety<br>Inventory | X | | | | | | | | | | | | | | | | | | | |
| Urine drug test | X | X | | X | | X | | X | | | X | | X | | X | | | | | X |
| Postural stability | | $X^{j}$ | $X^{\mathbf{k}}$ | | X | | X | | | X | | X | | X | | X | | | | |
| Cognitive PAB | | $X^{j}$ | $X^{\mathbf{k}}$ | | X | | X | | | X | | X | | X | | X | | | | |
| FSS | X | | | X | | | | X | | | | | | | | X | | | | |
| Morning Sleepiness | | | X | | X | | X | | | X | | X | | X | | X | | | | |
| Sleep Diary <sup>l</sup> | | | | | | | | | | | | | | | | | | <b>&gt;</b> | | |
| EQ-5D-3L | X | | | X | | | | X | | | | | | | | X | | | | |
| PK blood sampling <sup>m</sup> | | | | | | | | | | | X | X | | | X | X | | | | X |
| eC-SSRS | X | | | | | | | X | | | | X | | | | X | | X | X | X |
| Polysomnography <sup>n</sup> | | | X | | X | | X | | | X | | X | | X | | X | | | | |

Eisai 

Table 4 Schedule of Procedures/Assessments in Study E2006-G000-304

| Phase | | | Prei | andon | nizatio | n | | | Randomization | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Period | Scr | eening | 5 | | Ru | n-in | | BL | | | | Trea | tment | | | | Fol | low-Up ET <sup>e</sup> | | UN |
| Visit | 1 | 2a | 2b | 3a | 3b | 4a <sup>a</sup> | 4b | 5a | 5b | 5c | 6a <sup>b</sup> | 6b | 7a | 7b | 8a <sup>c</sup> | 8b | | EOS <sup>d</sup> | LI | UN |
| <b>Target Study Day</b> | -21 | -14 | -13 | -7 | -6 | -6 | -5 | 1 | 1 | 2 | 2 | 3 | 29 | 30 | 30 | 31 | | 44 | | |
| Window | -14/+4 | -3/ | <b>/+4</b> | -3/ | +3 | -3/ | +3 | | n/a | | n | /a | -2/ | <b>/+5</b> | -2/ | <b>/+5</b> | | | | |
| Possible Study<br>Day(s) Given<br>Window | -35<br>to<br>-17 | -17<br>to<br>-10 | -16<br>to<br>-9 | -10<br>to<br>-4 | -9<br>am<br>to<br>-3<br>am | -9<br>pm<br>to<br>-3<br>pm | -8<br>to<br>-2 | 1 | 1<br>pm | 2<br>am | 2<br>pm | 3<br>am | 29<br>pm | 30<br>am | 30<br>pm | 31<br>am | 31<br>to<br>44 | 44 | | |
| Procedures/<br>Assessments | | | | | | | | | | | | | | | | | | | | |
| Randomization | | | | | | | | | X | | | | | | | | | | | |
| PGI-Insomnia | | | | | | | | | | | | | | | | X | | | | |
| T-BWSQ | | | | | | | | | | | | | | | | | | X | X | |
| Dispense study drug | | | X | | | | | | | | | X | | | | | | | | |
| Study drug at bedtime <sup>o</sup> | | | - | | | | | | | | | | | | > | • | | | | |
| Retrieve unused study drug | | | | | | | | X | | | | | X | | | | | | | |
| Check study drug compliance <sup>p</sup> | | | | X | | | | X | | | | | X | | | | | | | |
| Admission to clinic | | X | | X | | X | | X | | | X | | X | | X | | | | | |
| Discharge from clinic | | | X | | X | | X | | | X | | X | | X | | X | | | | |
| Discharge from study | | | | | | | | | | | | | | | | | | X | X | |
| Adverse events <sup>q</sup> | | | | | | | | | | | | | | | | | | | : | <u> </u> |

Eisai 

E2006-G000-304

# (revised per Amendment 01)

# Table 4 Schedule of Procedures/Assessments in Study E2006-G000-304

BL = baseline, eC-SSRS = electronic Columbia-Suicide Severity Rating Scale, ECG = electrocardiogram, EMG = electromyography, EOS = end of study; ET = early termination, FSS = Fatigue Severity Scale, ISI = Insomnia Severity Index, PAB = performance assessment battery, PGI = Patient Global Impression, PK = pharmacokinetic, PSG = polysomnography, SDSB = Sleep Disorders Screening Battery, T-BWSQ = Tyrer Benzodiazepine Withdrawal Symptom Questionnaire; UN = unscheduled visit.

- a: Must be consecutive with Visit 3a.
- b: Must be consecutive with Visit 5b.
- c: Must be consecutive with Visit 7a.
- d: Must occur 14 18 days after Visit 8.
- e: Subjects who discontinue the study early for any reason after Randomization at Visit 5 should complete this visit.
- f: Inclusion and exclusion criteria to be evaluated at visits other than or in addition to Visit 1 are listed in Appendix 2.
- g: Viral screening for hepatitis B (HBsAg) and hepatitis C (HCV antibody IgG) will be conducted. (revised per Amendment 01)
- h: The Sleep Disorders Screening Battery includes: STOPBang, International Restless Legs Scale, Epworth Sleepiness Scale, and Munich Parasomnia Scale.
- i: Full physical examination (including a brief neurological exam) will be carried out at Screening and EOS and ET (if applicable). Brief physical examinations will be carried out at other visits.
- j: For training purposes only. Introduction to the CDR posture assessment and at least 2 training sessions of cognitive PAB to be completed before the end of Visit 2a. (revised per Amendment 02)
- k: For familiarization purposes only. The CDR posture and cognitive PAB assessments are to be completed at Visit 2b under the same conditions as for testing at subsequent visits.
- 1: Should be completed, within 1 hour of morning waketime, on every day of the study from Screening until the end of the study, and reviewed for eligibility before initiating any study assessments at Visit 2 and Visit 3.
- m: One PK blood sample (approximately 4 mL) will be obtained at the following timepoints: within 2 hours predose Day 2 and Day 30; within 1 hour after morning waketime on Day 3 and Day 31.
- n: PSG recordings will include a standard montage on all PSG nights. Diagnostic channels (respiratory effort, airflow, leg EMG) will be added to the standard montage on the PSG at Visit 2. All PSG visits will require an overnight stay in the clinic. At least 2 nights must intervene between the second BL PGG (Visit 4b) and BL (Visit 5a). (revised per Amendment 02)
- o: First dose of study drug is taken by the subject on the first night at home after Visit 2b. On the days that subjects are admitted to the clinic, study drug will be administered to the subject by clinical staff. The first dose of active study drug will be administered at Visit 5. On days that the subjects are not admitted to the clinic subjects will self-administer study drug. All study drug administration must be within 5 minutes of bedtime (defined as the time the subject attempts to sleep). (revised per Amendment 02)
- p: Subjects will be questioned about study drug compliance upon check-in at Visits 3a, 5a, and 7a. Tablet counts for study drug compliance will be done after end of Run-in Period and end of Treatment Period.
- q: At each visit, subjects will be asked whether they have had a fall since the previous visit. If yes, supplemental information must be obtained to support a narrative for the event, per Section 9.2.5 Adjudication Committee.

Eisai 

## 9.5.2.2 Description of Procedures/Assessments Schedule

The scheduling of study procedures and assessments is shown in Table 4.

# 9.5.3 Appropriateness of Measurements

Most of the clinical assessments are standard measurements commonly used in studies of drugs for the treatment of subjects with insomnia disorder.

Completion of sleep diaries by subjects is considered to be an appropriate method to measure changes in subjective sleep parameters, thereby allowing assessments of secondary efficacy in this study. The advantages of the electronic Sleep Diary to be used in this study include that the questions and instructional text have been adapted from sleep diaries that have were developed by clinicians and researchers with expertise in insomnia disorder, and have undergone linguistic validation and cognitive debriefing to optimize their use in this study. The Sleep Diary will include questions to assess the subject's rating of sleep quality each night and sleepiness/alertness level in the morning. The ISI has been widely used to evaluate the subjective impact of insomnia severity on psychosocial functioning, which is one type of davtime functioning impairment experienced by those with insomnia disorder. The FSS measures fatigue, which is another type of daytime impairment that is often a consequence of This scale has been employed primarily in clinical trials of cognitive and behavioral treatments for insomnia disorder. Because the objectives of this study include assessing the response to lemborexant of both nighttime sleep and daytime impairment complaints, the ISI and the FSS will be evaluated for changes from baseline. The PGI-Insomnia and EuroQoL assessment (version EQ-5D-3L) will also be employed. measures have been used in studies evaluating the impact of treatment for insomnia on the patients' global perceptions of sleep quality and quality of life. Together these measures will provide a broad evaluation of the effects of lemborexant on each patient's sleep, daytime functioning, and quality of life.

The CDR posture and cognitive PAB will assess whether there are residual effects of study drug on morning postural stability and cognition. There are documented effects of hypnotic drugs, including zolpidem, on postural stability and certain cognitive domains in the morning hours. These effects are associated with an increased risk of falling and other negative effects on functioning in the morning hours. The measures to be employed to evaluate the effects on postural stability and cognition have been widely used in clinical trials of drugs in older individuals, including clinical trials of treatments for insomnia disorder.

# 9.5.4 Reporting of Serious Adverse Events, Pregnancy, and Events Associated with Special Situations

## 9.5.4.1 Reporting of Serious Adverse Events

All SERIOUS ADVERSE EVENTS, regardless of their relationship to study treatment, must be reported on a completed SAE form by email or fax as soon as possible but no later than 24 hours from the time the investigator becomes aware of the event. (revised per Amendment 01)

Eisai 

Serious adverse events, regardless of causality assessment, must be collected through the last visit and for 28 days after the subject's last dose. All SAEs must be followed to resolution or, if resolution is unlikely, to stabilization. Any SAE judged by the investigator to be related to the study treatment or any protocol-required procedure should be reported to the sponsor regardless of the length of time that has passed since study completion.

The detailed contact information for reporting of SAEs is provided in the Investigator Study File.

**For urgent safety issues** please ensure all appropriate medical care is administered to the subject and contact the appropriate study team member listed in the Investigator Study File.

It is very important that the SAE report form be filled out as completely as possible at the time of the initial report. This includes the investigator's assessment of causality.

Any follow-up information received on SAEs should be forwarded within 24 hours of its receipt. (revised per Amendment 01) If the follow-up information changes the investigator's assessment of causality, this should also be noted on the follow-up SAE form.

Preliminary SAE reports should be followed as soon as possible by detailed descriptions including copies of hospital case reports, autopsy reports, and other documents requested by the sponsor.

The investigator must notify his/her IRB/IEC of the occurrence of the SAE in writing, if required by their institution. A copy of this communication must be forwarded to the sponsor or the responsible CRO, to be filed in the sponsor's Trial Master File.

# 9.5.4.2 Reporting of Pregnancy and Exposure to Study Drug Through Breastfeeding

Although the female subject population will be postmenopausal, in the event that a pregnancy does occur, investigators will capture and report such events.

Any pregnancy in which the estimated date of conception is either before the last visit or within 28 days of last study treatment, or any exposure to study drug through breastfeeding during study treatment or within 28 days of last study treatment, must be reported.

If an adverse outcome of a pregnancy is suspected to be related to study drug exposure, this should be reported regardless of the length of time that has passed since the exposure to study treatment.

A congenital anomaly, death during perinatal period, an induced abortion, or a spontaneous abortion are considered to be an SAE and should be reported in the same time frame and in the same format as all other SAEs (see Reporting of Serious Adverse Events [Section 9.5.4.1]).

Pregnancies or exposure to study drug through breastfeeding must be reported by fax or email as soon as possible but no later than 24 hours after the time the investigator becomes

Eisai  FINAL: (v7.0), 05 Feb 2018

aware of the pregnancy. (revised per Amendment 01) The contact information for the reporting of pregnancies and exposure to study drug through breastfeeding is provided in the Investigator Study File. The Pregnancy Report Form must be used for reporting. All pregnancies must be followed to outcome. The outcome of the pregnancy must be reported as soon as possible but no later than 24 hours after the time the investigator becomes aware of the outcome. (revised per Amendment 01)

A subject who becomes pregnant must be withdrawn from the study.

## 9.5.4.3 Reporting of Events Associated with Special Situations

Adverse events associated with study drug overdose, misuse, abuse, and medication error refer to AEs associated with uses of the study drug outside of that specified by the protocol. Overdose, misuse, abuse, and medication error are defined as follows:

Overdose Accidental or intentional use of the study drug in an amount higher

than the protocol-defined dose

Misuse Intentional and inappropriate use of study drug not in accordance with

the protocol

Abuse Sporadic or persistent intentional excessive use of study drug

accompanied by harmful physical or psychological effects

Medication error Any unintentional event that causes or leads to inappropriate study

drug use or subject harm while the study drug is in the control of site

personnel or the subject.

All AEs associated with overdose, misuse, abuse, or medication error should be captured on the Adverse Event CRF and also reported using the procedures detailed in Reporting of Serious Adverse Events (Section 9.5.4.1) even if the AEs do not meet serious criteria. Investigators should report whether one or both study drugs had been taken incorrectly. Abuse is always to be captured as an AE. If the AE associated with an overdose, misuse, abuse, or medication error does not meet serious criteria, it must still be reported using the SAE form and in an expedited manner but should be noted as nonserious on the SAE form and the Adverse Event eCRF.

## 9.5.4.4 Expedited Reporting

The sponsor must inform investigators (or as regionally required, the head of the medical institution) and regulatory authorities of reportable events, in compliance with applicable regulatory requirements, on an expedited basis (ie, within specific time frames). For this reason, it is imperative that sites provide complete SAE information in the manner described above.

## 9.5.4.5 Breaking the Blind

In the case of a medical emergency where the appropriate treatment of the subject requires knowledge of the study treatment given, the investigator may break the randomization code for an individual subject. In all such cases, the AE necessitating the emergency blind break will be handled as an SAE in accordance with the procedures indicated above. Any broken code will be clearly justified and documented. The Medical Monitor must be notified immediately of the blind break.

## 9.5.4.6 Regulatory Reporting of Adverse Events

Adverse events will be reported by the sponsor or a third party acting on behalf of the sponsor to regulatory authorities in compliance with local and regional law and established guidance. The format of these reports will be dictated by the local and regional requirements.

All studies that are conducted within any European country will comply with European Good Clinical Practice Directive 2005/28/EC and Clinical Trial Directive 2001/20/EC. All suspected unexpected serious adverse reactions will be reported, as required, to the competent authorities of all involved European member states.

# 9.5.5 Completion/Discontinuation of Subjects

For purposes of entering subject disposition in the eCRF, a subject will be considered to have completed the study per protocol after the End of Study visit has been completed. (revised per Amendment 01) For analysis purposes, a subject will be considered to have completed the study once the assessments on the morning after the last dose of study drug have been completed. All subjects will be required to return to the clinic at least 14, but not more than 18 days later for an End of Study (EOS) visit.

The investigator or subject may elect to discontinue the subject's participation in the study at any time for any reason. Subjects who discontinue study drug prematurely at any time after randomization at Visit 5 (Baseline) will be encouraged to return to the site as soon as possible (preferably within 7 days) to undergo an early termination (ET) Visit, as described in the Schedule of Procedures/Assessments (Table 4).

If the investigator or sponsor discontinues the study prematurely, the investigator will promptly explain to the subject involved that the study will be discontinued for that subject and will provide appropriate referral for medical treatment and other necessary measures for the subject. A subject who has ceased to return for visits will be followed up by mail, phone, or other means to gather information such as the reason for failure to return, the status of treatment compliance, the presence or absence of AEs, and clinical courses of signs and symptoms. This information will be recorded in the eCRF.

Subjects who discontinue early from the study will be discontinued for one of these primary reasons: AE(s), lost to follow-up, subject choice, lack of therapeutic effect, or administrative/other. Discontinuations due to non-compliance with study drug, time spent in

Eisai 

bed, or alcohol restrictions will be assigned to "administrative/other." In addition to the primary reason, the subject may indicate one or more of secondary reasons for discontinuation. Study disposition information will be collected on the Subject Disposition eCRF.

A subject removed from the study for any reason will not be replaced.

# 9.5.6 Abuse or Diversion of Study Drug

During the study, the investigator will report any concern about abuse or diversion of one or both study drugs.

Adverse events associated with abuse or diversion will be appropriately reported as AEs and monitored per Section 9.5.1.5.4. Abuse is always to be captured as an AE.

# 9.5.7 Confirmation of Medical Care by Another Physician

The investigator will instruct subjects to inform site personnel when they are planning to receive medical care by another physician. At each visit, the investigator will ask the subject whether he/she has received medical care by another physician since the last visit or is planning to do so in the future. When the subject is going to receive medical care by another physician, the investigator, with the consent of the subject, will inform the other physician that the subject is participating in the clinical study.

# 9.6 Data Quality Assurance

This study will be organized, performed, and reported in compliance with the protocol, SOPs, working practice documents, and applicable regulations and guidelines.

#### 9.6.1 Data Collection

Data required by the protocol will be collected on the eCRFs and entered into a validated data management system that is compliant with all regulatory requirements. As defined by ICH guidelines, the eCRF is a printed, optical, or electronic document designed to record all of the protocol-required information to be reported to the sponsor on each study subject.

Data collection on the eCRF must follow the instructions described in the eCRF Completion Guidelines. The investigator has ultimate responsibility for the collection and reporting of all clinical data entered on the eCRF. The investigator or designee as identified on Form FDA 1572 must sign the completed eCRF to attest to its accuracy, authenticity, and completeness.

Completed, original CRFs are the sole property of Eisai and should not be made available in any form to third parties without written permission from Eisai, except for authorized representatives of Eisai or appropriate regulatory authorities.

Eisai 

# 9.6.2 Clinical Data Management

All software applications used in the collection of data will be properly validated following standard computer system validation that is compliant with all regulatory requirements. All data, both eCRF and external data (eg, laboratory data), will be entered into a clinical system.

#### 9.7 Statistical Methods

# 9.7.1 Statistical and Analytical Plans

All statistical analyses will be performed by the sponsor or designee after the study is completed and the database is locked and released for unblinding. Statistical analyses will be performed using SAS software or other validated statistical software as required.

The statistical analyses are described in this section. Further details of the statistical analyses will be included in a separate SAP.

All statistical tests will be based on the 5% level of significance (2-sided). If statistical comparisons are not defined, all pairwise comparisons will be tested.

# 9.7.1.1 Study Endpoints

Unless otherwise stated, the time points for Sleep Diary endpoints refer to the mean of the final 7 nights before the visit.

## 9.7.1.1.1 PRIMARY ENDPOINT(S)

The primary endpoint is:

• Change from baseline of mean LPS on Days 29 and 30 of LEM10 and LEM5 compared to PBO (revised per Amendment 03)

#### 9.7.1.1.2 SECONDARY ENDPOINT(S)

## **Key Secondary Endpoints – US ONLY (revised per Amendment 03)**

- Change from baseline of mean SE on Days 29 and 30 of LEM10 and LEM5 compared to PBO
- Change from baseline of mean WASO on Days 29 and 30 of LEM10 and LEM5 compared to PBO (revised per Amendment 04)
- Change from baseline of mean WASO2H on Days 29 and 30 of LEM10 and LEM5 compared to ZOL

## **Key Secondary Endpoints – Non-US ONLY (revised per Amendment 03)**

 Change from baseline of mean SE on Days 29 and 30 of LEM10 and LEM5 compared to PBO

Eisai 

 Change from baseline of mean WASO on Days 29 and 30 of LEM10 and LEM5 compared to PBO

# Additional Secondary Endpoints – US and Non-US (revised per Amendment 03)

- Change from baseline on the postural stability test of mean units of body sway on Days 2 and 3 of LEM5 and LEM10 compared to ZOL
- Change from baseline of mean LPS, WASO, and TST on Days 1 and 2 and Days 29 and 30 of LEM5 and LEM10 compared to ZOL
- Change from baseline of mean subjective Sleep Diary variables including sSOL, sWASO, sSE and sTST over the first 7 and last 7 nights of the Treatment Period of LEM5 and LEM10 compared to ZOL
- Change from baseline of mean LPS, SE, WASO, WASO2H, and TST on Days 1 and 2 of LEM5 and LEM10 compared to PBO
- Change from baseline of mean WASO2H and TST on Days 29 and 30 of LEM5 and LEM10 compared to PBO
- Change from baseline mean of subjective Sleep Diary variables including sSOL, sWASO, sSE and sTST over the first 7 and last 7 nights of the Treatment Period of LEM5 and LEM10 compared to PBO
- Proportion of responders on Days 1 and 2 and Days 29 and 30 (PSG), and over the first 7 nights and last 7 nights of treatment (Sleep Diary), to LEM5 and LEM10 compared to ZOL and PBO, such that
  - o Objective sleep onset response is defined as LPS ≤ 20 minutes (provided mean baseline LPS was > 30 minutes)
  - o Subjective sleep onset response is defined as sSOL ≤ 20 minutes (provided mean baseline sSOL was > 30 minutes)
  - Objective sleep maintenance response is defined as WASO ≤ 60 minutes (provided mean baseline WASO was > 60 minutes and is reduced by > 10 minutes compared to baseline)
  - O Subjective sleep maintenance response is defined as  $sWASO \le 60$  minutes (provided mean WASO was > 60 minutes and is reduced by > 10 minutes compared to baseline)
- Safety and tolerability of LEM
- Change from baseline of the score from items 4-7 on the ISI at Day 31 of LEM5 and LEM10 compared to ZOL and PBO
- Change from baseline on the FSS score at Day 31 of LEM5 and LEM10 compared to ZOL and PBO
- Change from baseline of mean power of attention, mean continuity of attention, mean quality of memory, and mean speed of memory retrieval on Days 2 and 3

## 9.7.1.1.3 EXPLORATORY ENDPOINT(S) – US AND NON-US (REVISED PER AMENDMENT 03)

The change from baseline of WASO2H for LEM5 and LEM10 compared to ZOL will be considered as exploratory for non-US. The following endpoints will be also explored for LEM5 and LEM10. Except for PK endpoints, comparisons to ZOL and PBO will be made. (revised per Amendment 03)

- Change from baseline of the mean rating on the Quality of Sleep question from the Sleep Diary of the first 7 days and last 7 days of the Treatment Period
- Change from baseline of mean power of attention, mean continuity of attention, mean quality of memory, and mean speed of memory retrieval on Days 30 and 31
- From the postural stability test, change from baseline of mean units of body sway after the first 2 nights of the Treatment Period compared to PBO and the last 2 nights of the Treatment Period compared to ZOL and PBO
- Rebound insomnia endpoints as assessed from the Sleep Diary during the Follow-up Period
  - Change from baseline of sSOL at the following timepoints during the Follow-up Period: each of the first 3 nights, mean of the first 3 nights, mean of the first 7 nights, mean sSOL of the second 7 nights (revised per Amendment 03)
  - O Change from baseline of sWASO at the following timepoints during the Follow-up Period: each of the first 3 nights, mean of the first 3 nights, mean of the first 7, mean of the second 7 nights (revised per Amendment 03)
  - Proportion of subjects whose sSOL at the following timepoints during the Follow-up Period: each of the first 3 nights, mean of the first 3 nights, mean for first 7 nights, mean of the second 7 nights (revised per Amendments 02 and 03)
  - Proportion of subjects whose sWASO is higher at Screening at the following timepoints during the Follow-up Period: each of the first 3 nights, mean of the first 3 nights, mean for the first 7 nights, for thesecond 7 nights(revised per Amendments 02 and 03)
- Mean rating on the morning sleepiness item of the Sleep Diary on the first 7 mornings and last 7 mornings of the Treatment Period
- Mean rating on the morning sleepiness item of the Sleep Diary on the first 7 mornings and second 7 mornings of the Follow-up Period
- Change from baseline of mean morning sleepiness ratings assessed at 1.5 hours after waketime when subjects are in clinic on Days 1 and 2, and Days 29 and 30 (revised per Amendment 01)
- Change from baseline of mean minutes and mean percentage (a) per TIB and (b) per TST of sleep stage N1, N2, N3 (separately and combined) and REM on Days 1 and 2 and Days 29 and 30
- Change from baseline of mean REM latency, mean number of awakenings, and mean number of long awakenings at Days 1 and 2 and Days 29 and 30 (revised per Amendment 03)

- Number and percentage of subjects with a rating of a positive medication effect on each PGI-Insomnia item at Day 31
- Change from baseline on the EQ-5D-3L at Day 31
- Mean score on the T-BWSQ of LEM5 and LEM10 compared to ZOL and PBO at end of study
- Proportion of subjects who score ≥ 3 on the T-BWSQ of LEM5 and LEM10 compared to ZOL and PBO at end of study
- PK of lemborexant and its metabolites M4, M9, and M10
- Relationships between lemborexant PK, efficacy, and/or safety variables using PK/PD modeling

# 9.7.1.2 Definitions of Analysis Sets

The Safety Analysis Set is the group of randomized subjects who received at least 1 dose of randomized study drug and had at least 1 postdose safety assessment.

The Full Analysis Set (FAS) is the group of randomized subjects who received at least 1 dose of randomized study drug and had at least 1 postdose primary efficacy measurement.

The Per Protocol (PP) Analysis Set is the group of subjects who sufficiently complied with the protocol. Details of the evaluability criteria will be determined before database lock and treatment unblinding and will be specified in the SAP.

The PK Analysis Set is the group of subjects who have at least one quantifiable plasma concentration of lemborexant or its metabolites, or zolpidem, with adequately documented dosing history.

The PK/PD Analysis Set is the group of subjects receiving either lemborexant or placebo who have efficacy or safety data with documented dosing history. In addition, subjects receiving lemborexant should have at least one quantifiable lemborexant concentration data point as per the PK Analysis Set.

## 9.7.1.3 Subject Disposition

The number of subjects screened and the number failing screening (overall and by reason for failure) will be summarized. Screen failure data will be listed. The number of subjects randomized along with the number of subjects in each of the study populations will also be presented.

The number of subjects completing the study will be presented. Subjects who prematurely terminated their participation in the study will be summarized by their primary reason for study termination. Other reasons for study drug and study terminations will also be summarized. These tabulations will be produced for all randomized subjects by treatment group.

Eisai 

## 9.7.1.4 Demographic and Other Baseline Characteristics

Demographic and other baseline characteristics for the Safety Analysis Set will be summarized for each treatment group using descriptive statistics. Continuous demographic and baseline variables include age, height, weight, and BMI; categorical variables include sex, age group (55 – <65 years; 65 – <75 years; and 75 years or older), BMI group (less than 18.5, 18.5 to less than 25, 25 to 30, above 30), race and ethnicity. (revised per Amendments 03 and 04)

Characteristics of insomnia at Study Baseline will be summarized using Sleep Diary variables including sSOL, sWASO, sSE and sTST; PSG variables including LPS, WASO, SE, WASO2H and TST; ISI score and its individual question score, and FSS. The BDI-II and BAI scores will also be summarized at Study Baseline.

The above tables will be produced for the FAS if it differs from the Safety Analysis Set.

If sufficient numbers of subjects with a particular medical history (major depression, anxiety disorder, chronic pain, etc) are enrolled, demographic and other baseline characteristics will be summarized for each medical history group using descriptive statistics.

## 9.7.1.5 Prior and Concomitant Therapy

All investigator terms for medications recorded in the eCRF will be coded to an 11-digit code using the World Health Organization Drug Dictionary (Mar 2016 or latest version). The number (percentage) of subjects who take prior and concomitant medications will be summarized on the Safety Analysis Set by treatment group, Anatomical Therapeutic Chemical class, and World Health Organization Drug Dictionary-preferred term (PT). If the Safety Analysis Set and FAS differ substantially, then the prior and concomitant medication summaries will be repeated on the FAS.

Prior medications are defined as medications that stopped before the first dose of study drug, where study drug includes PBO during the Run-In Period.

Concomitant medications are defined as medications that (1) started before the first dose of randomized study drug and are continuing at the time of the first dose of study drug, or (2) started on or after the date of the first dose of randomized study drug to the last dose day plus 14 days. All medications will be presented in subject data listings. (revised per Amendment 02)

## 9.7.1.6 Efficacy Analyses

Where Sleep Diary endpoints are described, the first 7 nights of treatment refer to diary data entered on the first 7 mornings following the start of treatment; the last 7 nights of treatment refer to diary data entered on the last 7 mornings (up to and including the morning following the last PSG). Details of the handling of missing data for the various assessments will be addressed in the SAP.

Eisai 

Where PSG endpoints are described, Days 1 and 2 refer to the first two PSG recordings after start of treatment (scheduled on Visits 5 and 6), and Days 29 and 30 refer to the last two PSG recordings of the Treatment Period (scheduled on Visits 7 and 8).

## Definition of Baseline

Baseline is defined as the means from the 2 PSGs during the Run-in period for PSG-derived variables; and the mean of the last 7 mornings before the first Baseline PSG during the Run-In Period for Sleep Diary variables. For other endpoints, baseline data are captured during the Run-in Period and Baseline Period. Details will be specified in the SAP.

## Control of Type I Error (revised per Amendment 03)

A sequential gate-keeping procedure will be used for the primary and the key secondary endpoint comparisons to control for the overall type I error at the 0.05 significance level (Figure 2). The first endpoint comparison will be tested at the 0.05 significance level. If the testing is found to be statistically significant, then proceed to the next endpoint testing at significance level of 0.05, otherwise stop testing.

The primary endpoints will be tested in the following order:

- Change from baseline of the mean LPS of Days 29 and 30 of LEM10 compared to PBO
- Change from baseline of the mean LPS of Days 29 and 30 of LEM5 compared to PBO

The key secondary endpoints will only be tested if both primary analyses are statistically significant at the 0.05 level. The key secondary endpoints will be tested in the following order:

## **US Only**

- Change from baseline of the mean SE of Days 29 and 30 of LEM10 compared to PBO
- Change from baseline of the mean SE of Days 29 and 30 of LEM5 compared to PBO
- Change from baseline of the mean WASO of Days 29 and 30 of LEM10 compared to PBO (revised per Amendment 04)
- Change from baseline of the mean WASO2H of Days 29 and 30 of LEM10 compared to ZOL
- Change from baseline of the mean WASO on Days 29 and 30 of LEM5 compared to PBO (revised per Amendment 04)
- Change from baseline of the mean WASO2H on Days 29 and 30 of LEM5 compared to ZOL

## Non-US Only

- Change from baseline of the mean SE of Days 29 and 30 of LEM10 compared to PBO
- Change from baseline of the mean SE of Days 29 and 30 of LEM5 compared to PBO

- Change from baseline of the mean WASO of Days 29 and 30 of LEM10 compared to PBO
- Change from baseline of the mean WASO on Days 29 and 30 of LEM5 compared to PBO

No multiplicity adjustment will be done on other efficacy analyses.



Figure 2 Flow Chart of Gate Keeping Testing Procedure – Study E2006-G000-304 (revised per Amendment 04)

LEM5 = lemborexant 5 mg, LEM10 = lemborexant 10 mg, LPS = latency to persistent sleep, PBO = placebo, SE = sleep efficiency, US = Unites States, WASO = wake after sleep onset, WASO2H = wake after sleep onset in the second half of the night, ZOL = zolpidem tartrate extended release 6.25 mg.

## 9.7.1.6.1 PRIMARY EFFICACY ANALYSIS

Null Hypothesis: No difference exists in the mean change from baseline of the mean LPS of Days 29 and 30 for treatment with LEM10 (or LEM5) as compared with PBO. (revised per Amendment 03)

Alternative Hypothesis: A difference exists in the mean change from baseline of the mean LPS of Days 29 and 30 for LEM10 (or LEM5) compared to PBO. (revised per Amendment 03)

Eisai 

The LPS change from baseline (the mean of Days 1 and 2, and the mean of Days 29 and 30) will be analyzed using the mixed effect model repeated measurement analysis (MMRM) on the FAS. The model will include all data and will be adjusted for the corresponding baseline value (the means from the 2 PSG recordings during the Run-in Period), region, age group (55 – <65 years; 65 years or older), treatment, time (Days 1/2, and Days 29/30), and the interaction of treatment by time. Since LPS is known to be non-normally distributed, a logtransformation will be used in the analysis An unstructured covariance matrix will be used, and if the model fails to converge, then an autoregressive matrix will be used. The missing values will be imputed using a pattern mixture model utilizing multiple imputations (MI) assuming the missing values are missing not at random (MNAR) utilizing the complete case missing value pattern (CCMV - subjects who completed primary efficacy assessments without missing values). The missing values for a given visit will be imputed using all available values including the retrieved measurement from the post-discontinuation data. The treatment comparison will be performed using contrasts. The p-value, least square (LS) means and the 95% confidence interval (CI) for the treatment difference will also be provided. (revised per Amendments 03 and 04)

Subgroup analyses and additional sensitivity analysis will be performed as appropriate.

The following analyses will be considered as sensitivity analyses:

- PP analysis: The same primary efficacy analyses described above will be repeated based on PP analysis set.
- Completer analysis: The same primary efficacy analyses described above will be repeated on subjects who completed all efficacy assessments and have no missing values.
- As-treated analysis: The same primary efficacy analyses described in Section 5.4.1 (MMRM analysis with MI for missing value imputation) will be repeated based on the actual treatment the subject received regardless of randomization.
- MMRM analysis assuming missing at random (MAR): The same primary endpoint analysis described above will be analyzed using MMRM assuming the missing values are MAR. (revised per Amendment 03)
- MI Imputation assuming MNAR utilizing CCMV-4: The same MMRM method used in the primary analysis will be applied utilizing CCMV-4 (ie, up to 4 monotone missing patterns will be used for missing value imputation as follows): (revised per Amendment 04)

| Study days where results are available | 1 | 2 | 29 | 30 |
|----------------------------------------|---|---|----|----|
| Pattern 1 | X | X | X | X |
| Pattern 2 | X | X | X | • |
| Pattern 3 | X | X | | |
| Pattern 4 | X | | | • |
| x = result present; . = result missing | • | • | • | |

• Tipping point analysis: A range of shifts will be used in the multiple imputation of missing data assuming MNAR to identify the specific shift and treatment effect that will tip the results from statistically significant to non-significant. (revised per Amendment 04)

#### 9.7.1.6.2 SECONDARY EFFICACY ANALYSES

# **Key Secondary Efficacy Analysis (revised per Amendments 03 and 04)**

Changes from baseline of mean SE, WASO2H, and WASO of Days 1 and 2 and the mean of Days 29 and 30 will be analyzed using a pattern mixture model utilizing MI assuming MNAR. The treatment comparison will be performed using contrasts. The p-value, LS means and the 95% CI of the treatment differences will also be provided. The comparison of LEM10 and LEM5 to ZOL on WASO2H will be considered as exploratory for all non-US submissions. (revised per Amendment 03)

# Other Secondary Efficacy Analysis (revised per Amendment 03)

The other secondary efficacy endpoints (change from baseline of the mean of the following endpoints: LPS, SE, WASO2H, and WASO of the mean of Days 1 and 2; TST of the mean of Days 1 and 2 and of the mean of Days 29 and 30; sSOL, sWASO, sSE, and sTST for the mean of the first 7 and last 7 days of the Treatment Period) will be analyzed using MMRM assuming MAR. (revised per Amendment 03)

The proportion of responders will be analyzed using the Cochran-Mantel-Haenszel test, controlled for region and age group, for each dose of lemborexant compared to PBO and ZOL. The analysis will be similarly repeated for responder analysis based on Sleep Diary variables (sSOL and sWASO) over the first 7 and last 7 nights of treatment. (revised per Amendment 03)

The change from baseline of the ISI total of four items on daytime functioning at Day 31 and the FSS score at Day 31 will be analyzed using analysis of covariance (ANCOVA), adjusted for the corresponding baseline value, age group, region, and treatment. (revised per Amendment 03)

Changes from baseline in mean power of attention, mean continuity of attention, mean quality of memory, and mean speed of memory retrieval for the PAB tasks will be analyzed using MMRM assuming MAR. (revised per Amendments 01 and 03)

Secondary endpoints may also presented graphically or analyzed by modeling methods if warranted.

No multiplicity adjustment or missing value imputation is planned for other secondary analyses. (revised per Amendment 03)

#### 9.7.1.6.3 EXPLORATORY EFFICACY AND PHARMACODYNAMIC ANALYSES

The change from baseline mean score of the quality of sleep item on the Sleep Diary for the means of the first 7 days and last 7 days of the Treatment Period will be analyzed using MMRM assuming MAR. (revised per Amendment 03)

Rebound insomnia is defined as worsened sleep relative to Screening after study drug treatment is completed. Sleep Diary data from the Follow-up Period will be compared to Sleep Diary data from the Screening Period to assess whether subjects experience rebound insomnia. Specifically, a higher value for sSOL or sWASO during the Follow-up Period compared to the mean sSOL or sWASO value during the Screening Period will be considered worsened sleep. (revised per Amendments 01 and 02)

To assess rebound insomnia, both categorical analysis at the subject level and continuous analysis at the group mean level will be performed. For each of the first 3 nights, the mean of the first 3 nights, and the mean of each of the 2 weeks of the Follow-up Period the proportion of subjects whose corresponding value for sSOL or sWASO exceeds the corresponding Screening Period value by 5 minutes will be summarized by treatment group and compared to placebo. The percentage of 'rebounders' between each treatment and placebo group will be analyzed using a CMH test. (revised per Amendments 01, 02, and 03)

To assess statistical significance using the continuous data at the group mean level, the data will be analyzed using ANCOVA, adjusted for region, age group and treatment. The LS mean of each of the first 3 nights and each week of the Follow-up Period will be compared to the Screening Period between each treatment group and placebo. If the lower bound of the 95% CI of sSOL or sWASO for each of the first 3 nights and the mean of each week of the Follow-Up Period exceeds the upper bound of a 95% CI for the values during the Screening Period in the given treatment group, it will be considered strong evidence for rebound insomnia. If the LS means for sSOL and sWASO for the Follow-up Period are all lower than for the Screening Period, then no rebound insomnia is suggested. (revised per Amendments 01 and 03)

To evaluate morning residual sleepiness during study treatment and following completion of treatment, the change from baseline of the mean of morning sleepiness item on the Sleep Diary for the first 7 mornings of the Treatment Period, the last 7 mornings of the Treatment Period, as well as the means of the first 7 days and second 7 days of the Follow-up Period will be analyzed using MMRM assuming MAR. Change from baseline of the mean morning sleepiness ratings assessed at 1.5 hours after waketime when subjects are in clinic on days 1 and 2 and days 29 and 30 will be similarly analyzed using MMRM assuming MAR. (revised per Amendments 01 and 03)

The change from baseline of the mean of Days 1 and 2 and of the mean of Days 29 and 30 for the sleep architecture and other PSG endpoints (WASO1H, minutes and percentage [a] per TIB and [b] per TST of sleep stage N1, N2, N3, total NREM and REM; REM latency, DurLongAW, number of awakenings, number of long awakenings, REM episode frequency

and duration, and mean REM/NREM cycle duration) will be summarized. (revised per Amendment 03)

Each item on the PGI-Insomnia at Day 31 will be analyzed separately by calculating the number and percentages of subjects for each response category (eg, negative [3], neutral [2], positive [1] medication effect). The percentage of positive responses will be compared between treatment groups using the chi-square test, and repeated for age subgroups.

The change from baseline in the EQ-5D-3L score at Day 31 will be analyzed using ANCOVA, adjusted for region, age group and treatment. (revised per Amendment 03)

No multiplicity adjustment or missing value imputation is planned for exploratory and pharmocodynamic analyses. (revised per Amendment 03)

9.7.1.7 Pharmacokinetic, Pharmacodynamic, Pharmacogenomic, and Other Biomarker Analyses

#### 9.7.1.7.1 PHARMACOKINETIC ANALYSES

The Safety Analysis Set will be used for individual lemborexant and its metabolites M4, M9, and M10, as well as zolpidem (where quantified) plasma concentration listings. The PK Analysis Set will be used for summaries of lemborexant and its metabolites M4, M9, and M10, as well as zolpidem (where quantified) plasma concentrations by dose, time and day.

A population PK approach will be used to characterize the PK of lemborexant. For this approach, PK analysis data from this study will be pooled with relevant data from Phase 1 and 2 studies, and other Phase 3 studies if available. To explore sources of variability in lemborexant PK, the effect of covariates (eg, demographics) on the PK of lemborexant will be evaluated. The PK model will be parameterized for clearance (CL) and volumes of distribution. Derived exposure parameters such as AUC,  $C_{max}$ , and any other relevant parameters will be calculated from the model using the individual posterior estimate of CL and dosing history.

#### 9.7.1.7.2 PHARMACODYNAMIC, PHARMACOGENOMIC, AND OTHER BIOMARKER ANALYSES

# Pharmacodynamic Analyses

These analyses are described in the Secondary Efficacy Analyses, and Exploratory and Pharmacodynamic Analyses sections (above).

## Pharmacokinetic/Pharmacodynamic Analyses

The PK/PD relationship between exposure to lemborexant and efficacy variables including but not limited to LPS and WASO, and safety variables including but not limited to morning sleepiness and frequently occurring treatment-emergent adverse events (TEAEs), will be explored graphically. Any emergent PK/PD relationships will be evaluated by population PK/PD modeling. The population PK/PD analysis plan will be described and results will be reported in a separate document.

Eisai 

Population PK and PK/PD analyses will be performed using NONMEM version 7.2 or later.

# Pharmacogenomic Analyses

Not applicable

# Other Biomarker Analyses

Not applicable.

# 9.7.1.8 Safety Analyses

Evaluations of safety will be performed on the relevant Safety Analysis Set.

#### 9.7.1.8.1 EXTENT OF EXPOSURE

The extent of exposure (mean daily dose, cumulative dose, duration of exposure) to study drug will be summarized descriptively for each study drug.

Compliance for each study drug will be calculated on the basis of number of tablets dispensed, lost and returned, separately for each type of tablet. Summaries will provide descriptive summary statistics and number (percentage) of subjects below 80%, between 80% and 120%, and greater than 120%.

#### 9.7.1.8.2 ADVERSE EVENTS

The AE verbatim descriptions (investigator terms from the eCRF) will be classified into standardized medical terminology using the MedDRA. Adverse events will be coded to the MedDRA (Version 17.0 or higher) lower level term closest to the verbatim term. The linked MedDRA PT and primary system organ class (SOC) are also captured in the database.

A TEAE is defined as an AE that emerges during treatment (including the Run-In Period), having been absent at pretreatment (before the PBO Run-In Period) or

- Reemerges during treatment, having been present at pretreatment (before the Run-In Period) but stopped before treatment, or
- Worsens in severity during treatment relative to the pretreatment state, when the AE is continuous.

Only those AEs that are treatment-emergent will be included in summary tables. All AEs, treatment-emergent or otherwise, will be presented in subject data listings. AEs will be classified as TEAEs up to 14 days after the last study treatment.

Adverse events will be summarized by descriptive statistics, using the Safety Analysis Set. The TEAEs will be summarized by treatment group at the start of the TEAE. The incidence of TEAEs will be reported as the number (percentage) of subjects with TEAEs by SOC and PT. A subject will be counted only once within an SOC and PT, even if the subject

Eisai 

experienced more than 1 TEAE within a specific SOC and PT. The number (percentage) of subjects with TEAEs during the Run-In Period will be summarized separately. The number (percentage) of subjects with TEAEs during the Treatment Period will be summarized separately. The number (percentage) of subjects with TEAEs will also be summarized by maximum severity (mild, moderate, or severe).

The number (percentage) of subjects with TEAEs will also be summarized by relationship to study drug (Yes [related] and No [not related]). Treatment-related TEAEs include those events considered by the investigator to be related to study treatment.

The number (percentage) of subjects with treatment-emergent SAEs will be summarized by MedDRA SOC and PT for each treatment group. A subject data listing of all SAEs will be provided.

The number (percentage) of subjects with TEAEs leading to discontinuation from study drug will be summarized by MedDRA SOC and PT for each treatment group. A subject data listing of all AEs leading to discontinuation from study drug will be provided.

The number (percentage) of subjects with TEAEs of cataplexy or other events that are characterized according to the customized MedDRA query PT as potential cataplexy-related events, as well as somnolence and related events, and drug abuse liability will be summarized separately. (revised per Amendment 01)

#### 9.7.1.8.3 CLINICAL LABORATORY VALUES

Clinical laboratory values will be evaluated for each laboratory parameter by subject. Abnormal laboratory values will be identified as those outside (above or below) the normal range. Reference (normal) ranges for laboratory parameters will be included in the clinical study report for this study. Descriptive summary statistics (eg, mean, SD, median, minimum, maximum for continuous variables, and number and percentage for categorical variables) for the laboratory parameters and changes from baseline will be evaluated by treatment group and visit.

Laboratory test results will be assigned a low-normal-high (LNH) classification according to whether the value was below (L), within (N), or above (H) the laboratory parameter's reference range. Within-treatment comparisons will be based on 3 by 3 tables (shift tables) that, for a particular laboratory test, compare the Study Baseline LNH classification to the LNH classification at end of study/early termination, by treatment group.

Clinical laboratory results post-baseline will be evaluated for markedly abnormal values. A laboratory test will be considered markedly abnormal if the result worsens to meet Eisai grading criteria for laboratory values limit of Grade 2 or higher. If the Grade 2 limit is missing, the Grade 1 limit will be considered. Appendix 1 presents the Eisai grading criteria for laboratory values that were used to identify subjects with markedly abnormal laboratory values. For the incidence of markedly abnormal laboratory values, each subject may be counted once in the laboratory parameter value high and in the laboratory parameter low categories as applicable.

Eisai 

## 9.7.1.8.4 VITAL SIGNS, HEIGHT, AND WEIGHT

Descriptive statistics for vital signs parameters (ie, diastolic and systolic BP, pulse, respiration rate, temperature) and weight, and changes from Study Baseline will be presented by visit and treatment group. Height will be measured once at Visit 1.

Vital sign values will be listed. Clinically notable vital sign values will be identified on the listings as those above (H) or below (L) a clinically notable range (Table 5). Categorical analyses of subjects (number and percent) who fall outside the below clinically notable vital sign ranges will also be presented for change from Study Baseline, by treatment group and by time point.

| Table 5 | Vital Sign ( | Criteria |
|---------|--------------|----------|
|---------|--------------|----------|

| Variable | Criterion value <sup>a</sup> | Change relative to baseline <sup>a</sup> | Clinically notable range |
|---|---|---|---|
| Heart rate | >120 bpm | Increase of 15 bpm | Н |
| Heart rate | <50 bpm | Decrease of ≥15 bpm | L |
| Systolic BP | >180 mmHg | Increase of ≥20 mmHg | Н |
| | <90 mmHg | Decrease of ≥20 mmHg | L |
| Diastolic BP | >105 mmHg | Increase of ≥15 mmHg | Н |
| Diastolic BP | <50 mmHg | Decrease of ≥15 mmHg | L |

BP = blood pressure, H = high, L = low.

#### 9.7.1.8.5 ELECTROCARDIOGRAMS

Descriptive statistics for ECG parameters and changes from Study Baseline will be presented by treatment group. Shift tables will present changes from Study Baseline in ECG interpretation (categorized as normal or abnormal) by time point. (revised per Amendment 02)

For each subject, the maximum observed corrected QT interval calculated using Fridericia's formula (QTcF), the corrected QT interval calculated using Bazett's formula (QTcB), and the maximum prolongation from baseline in QTcF will be compiled. Categorical analyses of subjects (number and percent) with maximum observed QTcF values >450 msec, >480 msec, and >500 msec and maximum prolongations (from Study Baseline) in QTcF >30 msec and >60 msec will be presented by treatment group and by time point. Categorical analyses of subjects (number and percent) with maximum observed PR values > 220 msec, and QRS values > 120 msec will be presented by treatment group and by time point.

a. Clinically notable means that a value must meet the criterion value and must attain the specified magnitude of change relative to baseline.

#### 9.7.1.8.6 OTHER SAFETY ANALYSES

To evaluate morning residual sleepiness during study treatment and following completion of treatment, the change from baseline of the mean of morning residual sleepiness item on the Sleep Diary for the first 7 mornings of the Treatment Period, the last 7 mornings of the Treatment Period, as well as the means of each of the 2 weeks after treatment discontinuation will be analyzed using MMRM assuming MAR. (revised per Amendment 03)

The results of eC-SSRS assessments will be listed for each subject. The incidence of suicidal ideation or suicidal behavior will be summarized by treatment group using descriptive statistics as appropriate.

Withdrawal symptoms will be assessed using the T-BWSQ. The mean score will be summarized by treatment group, and number (percentage) of subjects with a score  $\geq 3$  will be summarized.

Urine drug test results will also be listed.

# 9.7.1.9 Other Analyses

Secondary and exploratory endpoints may be additionally presented graphically or analyzed by modeling methods if warranted.

Although zolpidem is included in the study as an active comparator, comparison of ZOL to PBO, and comparison between LEM5 and LEM10 may be made to facilitate evaluation of study results.

## 9.7.2 Determination of Sample Size

The sample size was estimated for the each comparison of LEM10 vs. PBO, and LEM5 vs PBO with respect to the mean change from baseline of LPS at Month 1, on the basis of a 2-sided t-test at the  $0.05 \, \alpha$ -level for each treatment comparison. (revised per Amendment 03)

On the basis of the dose finding study E2006-G000-201 (Study 201), across various lemborexant doses (1 to 25 mg) at Days 14 and 15, the standard deviation (SD) of change from baseline for log-transformed LPS is assumed to be 0.9. The LS mean treatment difference at Days 14/15 from Study 201 for log-transformed LPS of LEM10 and LEM5 compared with PBO was 0.75 and -1.15, respectively. Therefore, a sample size of 250 subjects for LEM5, 250 subjects for LEM10, and 200 subjects for PBO has at least 95% power for each treatment comparison, LEM10 with PBO, and LEM5 with PBO, based on 2-sided, 2-sample t-test at 5% significance level. (revised per Amendment 03)

Power is also estimated for the key secondary objectives, the comparison of LEM10 and LEM5 to PBO on change from baseline of SE and WASO, and LEM10 and LEM5 to ZOL on WASO2H. A sample size of 250 subjects each for LEM5, LEM10, and ZOL, and 200 subjects for PBO has at least a 95% power for detecting a statistically significant difference between LEM and PBO for change from baseline in SE, at least 80% power for detecting a

Eisai 

statistically significant difference between LEM10 and ZOL/PBO for change from baseline in WASO/WASO2H based on 2-sided 2-sample t-test at 5% significance level. (revised per Amendments 03 and 04).

Table 6: Power and Sample Size Calculation for Change from Baseline of LPS, SE, WASO2H, and WASO

| Endpoint (Test) | <b>Estimated Treatment Difference</b> | Estimated SD | Power |
|---|---|---|---|
| Log(LPS) (LEM5 vs PBO) | -0.75 | 0.9 | >95% |
| Log(LPS) (LEM10 vs PBO) | -1.15 | 0.9 | >95% |
| SE (LEM5 vs PBO) | 5% | 14% | >95% |
| SE (LEM10 vs PBO) | 7% | 14% | >95% |
| WASO (LEM5 vs PBO) | -10 min | 55 min | 48% |
| WASO (LEM10 vs PBO) | -15 min | 55 min | 81% |
| WASO2H (LEM5 vs ZOL) | -8 min | 38 min | 65% |
| WASO2H (LEM10 vs ZOL) | -11 min | 38 min | 89% |

NOTE: Estimated treatment difference and SD are based on Study 201.

# 9.7.3 Interim Analysis

An interim analysis is planned to be conducted after approximately 50% of subjects (approximately n=475 subjects) have been randomized and either completed Day 31 assessments or discontinued from the study. This interim analysis will be conducted for administrative reasons as detailed in the separate Interim Analysis charter. When the specified number of subjects has completed the Day 31 assessments, an independent statistician external to the Sponsor will be provided with the relevant PSG dataset and will be unblinded to the primary endpoint, ie, change from baseline in WASO2H for the mean of Days 29 and 30. A conditional power will be calculated to predict the probability that the trial will achieve a significant treatment effect for WASO2H in the LEM10 versus ZOL arms at the end of the study, given what is observed at the time of interim analysis. The interim analysis will be limited to the comparison of LEM10 versus ZOL on the change from baseline in WASO2H for the mean of Days 29 and 30. No other endpoints, dose groups, or timepoints will be analyzed at the interim analysis. The study will not be terminated for either futility or efficacy. Therefore no impact to the type I error rate is expected.

The method of calculating the conditional power will be detailed in the Interim Analysis charter, along with operational procedures, unblinding procedures, procedures for communicating the results of the conditional power calculation and recipients of this information. To preclude potential influence on the conduct of the remainder of the study, disclosure of the conditional power will be limited to a prespecified set of executive-level individuals at the sponsor and sponsor's co-development partner. No individuals involved with the conduct of the study will have access to the interim data or the results of the interim

Eisai 

analysis (i.e., the conditional power of LEM10 versus ZOL on the change from baseline in WASO2H for the mean of Days 29 and 30).

Enrollment of subjects will not be stopped during the interval during which the interim analysis is conducted. The interim analysis may be waived or otherwise not conducted, for reasons including but not limited to a higher than anticipated enrollment rate which would make the interim analysis unnecessary as the majority of subjects would have been enrolled by the time the interim analysis is concluded.

# 9.7.4 Procedure for Revising the Statistical Analysis Plan

If the SAP needs to be revised after the study starts, the sponsor will determine how the revision impacts the study and how the revision should be implemented. The details of the revision will be documented and described in the clinical study report.

## 10 REFERENCE LIST

Abetz L, Arbuckle R, Allen RP, Garcia-Borreguero D, Hening W, Walters AS, et al. The reliability, validity and responsiveness of the International Restless Legs Syndrome Study Group rating scale and subscales in a clinical-trial setting. Sleep Med. 2006;7:340–9.

Allain H, Bentué-Ferrer D, Tarral A, Gandon JM. Effects on postural oscillation and memory functions of a single dose of zolpidem 5 mg, zopiclone 3.75 mg and lormetazepam 1 mg in elderly healthy subjects. A randomized, cross-over, double- blind study versus placebo. Eur J Clin Pharmacol. 2003;59(3):179-88.

Bastien CH, Vallières A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001;2(4):297-307.

Beck AT, Ward CH, Mendelson M, Mock J, Erbaugh J. An inventory for measuring depression. Arch. Gen. Psychiatry. 1961;4(6):561–71.

Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: Psychometric properties J Consult Clinical Psychol. 1988;56: 893–7.

Boyle J, Wolford D, Gargano C, McCrea J, Cummings C, Cerchio K, et al. Next-day residual effects of gaboxadol and flurazepam administered at bedtime: a randomized double-blind study in healthy elderly subjects. Hum Psychophamacol Clin Exp. 2009;24:61-71.

Brooks R. EuroQol: the current state of play. Health Policy 1996;37(1):53-72.

Chung F, Yegneswaran B, Liao P, Chung SA, Vairavanathan S, Islam S, et al. STOP Questionnaire A Tool to Screen Patients for Obstructive Sleep Apnea. Anesthesiology 2008;108:812–21.

Fulda S, Hornyak M, Müller K, Cerny L, Beitinger PA, Wetter TC. Development and validation of the Munich Parasomnia Screening (MUPS). A questionnaire for parasomnias and nocturnal behaviors. Somnologie 2008;12:56–65.

Johns MW. Reliability and factor analysis of the Epworth Sleepiness Scale. Sleep 1992;15(4):376-81.

Jongen S, Vuurman E, Ramaekers J, Vermeeren A. Alcohol calibration of tests measuring skills related to car driving. Psychopharmacology (Berl). 2014;231(12):2435 47.

Mets MA, Volkerts ER, Olivier B, Verster JC. Effect of hypnotic drugs on body balance and standing steadiness. Sleep Med Rev. 2010;14(4):259-67.

Posner K, Brown G.K, Stanley B, Brent DA, Yershova KV, Oquendo MA, et al. The Columbia-Suicide Severity Rating Scale: Initial Validity and Internal Consistency Findings From Three Multisite Studies With Adolescents and Adults. Am J Psychiatry. 2011;168:1266-77
Roth T, Soubrane C, Titeux L, et al. Efficacy and safety of zolpidem-MR: A double-blind, placebo-controlled study in adults with primary insomnia. Sleep Med. 2006;7:397–406.

Schwartz JE, Jandorf L, Krupp LB. The measurement of fatigue: a new instrument. J Psychosom Res. 1993 37(7):753-62.

Stranks EK, Crowe SF. The acute cognitive effects of zopiclone, zolpidem, zaleplon, and eszopiclone: a systematic review and meta analysis. J Clin Exp Neuropsych. 2014;36(7):691-700.

The EuroQol Group (1990). EuroQol-a new facility for the measurement of health-related quality of life. Health Policy. 1990;16(3):199-208.

Tyrer P, Murphy S, Riley P. The benzodiazepine withdrawal symptom questionnaire. J Affect Disord. 1990;19(1):53-61.

Walsh JK, Soubrane C, Roth T. Efficacy and safety of zolpidem extended release in elderly primary insomnia patients. Am J Geriatr Psychiatry. 2008 Jan;16(1):44-57.

Wesnes KA, Garatt C, Wickens M, Gudgoen A, Oliver S. Effects of sibutramine alone and with alcohol on cognitive function in healthy volunteers. Br J Clin Pharmacol. 2000;49:110-7.

eC-SSRS Reference: http://www.cssrs.columbia.edu/ecssrs.html

# 11 PROCEDURES AND INSTRUCTIONS (ADMINISTRATIVE PROCEDURES)

## 11.1 Changes to the Protocol

Any change to the protocol requires a written protocol amendment or administrative change that must be approved by the sponsor before implementation. Amendments specifically affecting the safety of subjects, the scope of the investigation, or the scientific quality of the study require submission to health or regulatory authorities as well as additional approval by the applicable IRBs/IECs. These requirements should in no way prevent any immediate action from being taken by the investigator, or by the sponsor, in the interest of preserving the safety of all subjects included in the study. If the investigator determines that an immediate change to or deviation from the protocol is necessary for safety reasons to eliminate an immediate hazard to the subjects, the sponsor's Medical Monitor and the IRB/IEC for the site must be notified immediately. The sponsor must notify the health or regulatory authority as required per local regulations.

Protocol amendments that affect only administrative aspects of the study may not require submission to health or regulatory authority or the IRB/IEC, but the health or regulatory authority and IRB/IEC (or if regionally required, the head of the medical institution) should be kept informed of such changes as required by local regulations. In these cases, the sponsor may be required to send a letter to the IRB/IEC and the Competent Authorities (or, if regionally required, the head of the medical institution) detailing such changes.

#### 11.2 Adherence to the Protocol

The investigator will conduct the study in strict accordance with the protocol (refer to ICH E6, Section 4.5).

## 11.3 Monitoring Procedures

The sponsor's/CRO's CRA will maintain contact with the investigator and designated staff by telephone, letter, or email between study visits, Monitoring visits to each site and remote monitoring will be conducted between onsite monitoring visits by the assigned CRA as described in the monitoring plan. The investigator (or if regionally required, the head of the medical institution) will allow the CRA to inspect the clinical, laboratory, and pharmacy facilities to assure compliance with GCP and local regulatory requirements. The eCRFs and subject's corresponding original medical records (source documents) are to be fully available for review by the sponsor's representatives at regular intervals. These reviews verify adherence to study protocol and data accuracy in accordance with local regulations. All records at the site are subject to inspection by the local auditing agency and to IRB/IEC review.

In accordance with ICH E6, Section 1.52, source documents include, but are not limited to, the following:

Eisai 

- Clinic, office, or hospital charts
- Copies or transcribed health care provider notes that have been certified for accuracy after production
- Recorded data from automated instruments such as IxRS, x-rays, and other imaging reports (eg., ECGs, rhythm strips, EEGs, polysomnographs) regardless of how these images are stored, including microfiche and photographic negatives (revised per Amendment 01)
- Quality of life or medical history questionnaires completed by subjects (revised per Amendment 01)
- Records of telephone contacts
- Diaries or evaluation checklists
- Drug distribution and accountability logs maintained in pharmacies or by research personnel
- Laboratory results and other laboratory test outputs (eg, urine dipsticks) (revised per Amendment 01)
- Correspondence regarding a study subject's treatment between physicians or memoranda sent to the IRBs/IECs
- eCRF components (eg, questionnaires) that are completed directly by subjects and serve as their own source

#### 11.4 Recording of Data

An eCRF is required and must be completed for each subject by qualified and authorized personnel. All data on the eCRF must reflect the corresponding source document, except when a section of the eCRF itself is used as the source document. Any correction to entries made on the eCRF must be documented in a valid audit trail where the correction is dated, the individual making the correct is identified, the reason for the change is stated, and the original data are not obscured. Only data required by the protocol for the purposes of the study should be collected.

The investigator must sign each eCRF. The investigator will report the eCRFs to the sponsor and retain a copy of the eCRFs.

#### 11.5 Identification of Source Data

All data to be recorded on the eCRF must reflect the corresponding source documents.

#### 11.6 Retention of Records

The circumstances of completion or termination of the study notwithstanding, the investigator (or if regionally required, the head of the medical institution or the designated representative) is responsible for retaining all study documents, including but not limited to the protocol, copies of eCRFs, the Investigator's Brochure, and regulatory agency registration documents (eg, Form FDA 1572 ICFs, and IRB/IEC correspondence). In addition, the

Eisai 

sponsor will send a list of treatment codes by study subject to the investigator after the clinical database for this study has been locked. The site should plan to retain study documents, as directed by the sponsor, for at least 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or at least 3 years have elapsed since the formal discontinuation of clinical development of the investigational product.

It is requested that at the completion of the required retention period, or should the investigator retire or relocate, the investigator contact the sponsor, allowing the sponsor the option of permanently retaining the study records.

## 11.7 Auditing Procedures and Inspection

In addition to routine monitoring procedures, the sponsor's Clinical Quality Assurance department conducts audits of clinical research activities in accordance with the sponsor's SOPs to evaluate compliance with the principles of ICH GCP and all applicable local regulations. If a government regulatory authority requests an inspection during the study or after its completion, the investigator must inform the sponsor immediately.

## 11.8 Handling of Study Drug

All study drug will be supplied to the PI (or a designated pharmacist) by the sponsor. Drug supplies must be kept in an appropriate secure area (eg, locked cabinet) and stored according to the conditions specified on the drug labels. The investigator (or a designated pharmacist) must maintain an accurate record of the shipment and dispensing of the study drug in a drug accountability ledger, a copy of which must be given to the sponsor at the end of the study. An accurate record of the date and amount of study drug dispensed to each subject must be available for inspection at any time. The CRA will visit the site and review these documents along with all other study conduct documents at appropriate intervals once study drug has been received by the site.

All drug supplies are to be used only for this study and not for any other purpose. The investigator (or site personnel) must not destroy any drug labels or any partly used or unused drug supply before approval to do so by the sponsor. At the conclusion of the study and as appropriate during the study, the investigator (or a designated pharmacist) will return all used and unused drug containers, drug labels, and a copy of the completed drug disposition form to the sponsor's CRA or, when approval is given by the sponsor, will destroy supplies and containers at the site.

#### 11.9 Publication of Results

All manuscripts, abstracts, or other modes of presentation arising from the results of the study must be reviewed and approved in writing by the sponsor in advance of submission pursuant to the terms and conditions set forth in the executed Clinical Trial Agreement between the sponsor/CRO and the institution/investigator. The review is aimed at protecting

Eisai 

the sponsor's proprietary information existing either at the date of the commencement of the study or generated during the study.

The detailed obligations regarding the publication of any data, material results, or other information generated or created in relation to the study shall be set out in the agreement between each investigator and the sponsor or CRO, as appropriate.

#### 11.10 Disclosure and Confidentiality

The contents of this protocol and any amendments and results obtained during the study should be kept confidential by the investigator, the investigator's staff, and the IRB/IEC and will not be disclosed in whole or in part to others, or used for any purpose other than reviewing or performing the study, without the written consent of the sponsor. No data collected as part of this study will be used in any written work, including publications, without the written consent of the sponsor. These obligations of confidentiality and non-use shall in no way diminish such obligations as set forth in either the Confidentiality Agreement Agreement the sponsor/CRO Clinical Trial executed between and institution/investigator.

All persons assisting in the performance of this study must be bound by the obligations of confidentiality and non-use set forth in either the Confidentiality Agreement or Clinical Trial Agreement executed between the institution/investigator and the sponsor/CRO.

# 11.11 Discontinuation of Study

The sponsor reserves the right to discontinue the study for medical reasons or any other reason at any time. If a study is prematurely terminated or suspended, the sponsor will promptly inform the investigators/institutions and regulatory authorities of the termination or suspension and the reason(s) for the termination or suspension. The IRB/IEC will also be informed promptly and provided the reason(s) for the termination or suspension by the sponsor or by the investigator/institution, as specified by the applicable regulatory requirement(s).

The investigator reserves the right to discontinue the study should his/her judgment so dictate. If the investigator terminates or suspends a study without prior agreement of the sponsor, the investigator should inform the institution where applicable, and the investigator/institution should promptly inform the sponsor and the IRB/IEC and provide the sponsor and the IRB/IEC with a detailed written explanation of the termination or suspension. Study records must be retained as noted above.

# 11.12 Subject Insurance and Indemnity

The sponsor will provide insurance for any subjects participating in the study in accordance with all applicable laws and regulations.

Eisai  FINAL: (v7.0), 05 Feb 2018

# 12 APPENDICES

Eisai 

# **Appendix 1 Sponsor's Grading for Laboratory Values**

# **Sponsor's Grading for Laboratory Values**

| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| BLOOD/BONE MARROW | | | | |
| Hemoglobin | <lln -="" 10.0="" dl<br="" g=""><lln -="" 100="" g="" l<br=""><lln -="" 6.2="" l<="" mmol="" td=""><td>&lt;10.0 – 8.0 g/dL<br/>&lt;100 – 80 g/L<br/>&lt;6.2 – 4.9 mmol/L</td><td>&lt;8.0 g/dL<br/>&lt;80 g/L<br/>&lt;4.9 mmol/L;<br/>transfusion indicated</td><td>life-threatening<br/>consequences; urgent<br/>intervention<br/>indicated</td></lln></lln></lln> | <10.0 – 8.0 g/dL<br><100 – 80 g/L<br><6.2 – 4.9 mmol/L | <8.0 g/dL<br><80 g/L<br><4.9 mmol/L;<br>transfusion indicated | life-threatening<br>consequences; urgent<br>intervention<br>indicated |
| Leukocytes (total WBC) | <lln -="" 3.0×10<sup="">9/L<br/><lln -="" 3000="" mm<sup="">3</lln></lln> | <3.0 - 2.0×10 <sup>9</sup> /L<br><3000 - 2000/mm <sup>3</sup> | <2.0 - 1.0×10 <sup>9</sup> /L<br><2000 - 1000/mm <sup>3</sup> | <1.0×10 <sup>9</sup> /L<br><1000/mm <sup>3</sup> |
| Lymphocytes | <lln -="" 800="" mm<sup="">3<br/><lln -="" 0.8×10<sup="">9/L</lln></lln> | <800 - 500/mm <sup>3</sup><br><0.8 - 0.5×10 <sup>9</sup> /L | <500 - 200/mm <sup>3</sup><br><0.5 - 0.2×10 <sup>9</sup> /L | <200/mm <sup>3</sup><br><0.2×10 <sup>9</sup> /L |
| Neutrophils | <lln -="" 1.5×10<sup="">9/L<br/><lln -="" 1500="" mm<sup="">3</lln></lln> | <1.5 - 1.0×10 <sup>9</sup> /L<br><1500 - 1000/mm <sup>3</sup> | <1.0 - 0.5×10 <sup>9</sup> /L<br><1000 - 500/mm <sup>3</sup> | <0.5×10 <sup>9</sup> /L<br><500/mm <sup>3</sup> |
| Platelets | <lln -="" 75.0×10<sup="">9/L<br/><lln -="" 75,000="" mm<sup="">3</lln></lln> | <75.0 - 50.0×10 <sup>9</sup> /L<br><75,000 - 50,000/mm <sup>3</sup> | <50.0 - 25.0×10 <sup>9</sup> /L<br><50,000 - 25,000/mm <sup>3</sup> | <25.0×10 <sup>9</sup> /L<br><25,000/mm <sup>3</sup> |
| METABOLIC/LABORATORY | | | | |
| Albumin, serum- low (hypoalbuminemia) | <lln -="" 3="" dl<br="" g=""><lln -="" 30="" g="" l<="" td=""><td>&lt;3 - 2 g/dL<br/>&lt;30 - 20 g/L</td><td>&lt;2 g/dL<br/>&lt;20 g/L</td><td>life-threatening<br/>consequences; urgent<br/>intervention<br/>indicated</td></lln></lln> | <3 - 2 g/dL<br><30 - 20 g/L | <2 g/dL<br><20 g/L | life-threatening<br>consequences; urgent<br>intervention<br>indicated |
| Alkaline phosphatase | >ULN - 3.0×ULN | >3.0 – 5.0×ULN | >5.0 – 20.0×ULN | >20.0×ULN |
| ALT | >ULN - 3.0×ULN | >3.0 – 5.0×ULN | >5.0 – 20.0×ULN | >20.0×ULN |
| AST | >ULN - 3.0×ULN | >3.0 – 5.0×ULN | >5.0 – 20.0×ULN | >20.0×ULN |
| Bilirubin (hyperbilirubinemia) | >ULN – 1.5×ULN | >1.5 – 3.0×ULN | >3.0 – 10.0×ULN | >10.0×ULN |
| Calcium, serum-low (hypocalcemia) | <lln -="" 8.0="" dl<br="" mg=""><lln -="" 2.0="" l<="" mmol="" td=""><td>&lt;8.0 – 7.0 mg/dL<br/>&lt;2.0 – 1.75 mmol/L</td><td>&lt;7.0 – 6.0 mg/dL<br/>&lt;1.75 – 1.5 mmol/L</td><td>&lt;6.0 mg/dL<br/>&lt;1.5 mmol/L</td></lln></lln> | <8.0 – 7.0 mg/dL<br><2.0 – 1.75 mmol/L | <7.0 – 6.0 mg/dL<br><1.75 – 1.5 mmol/L | <6.0 mg/dL<br><1.5 mmol/L |
| Calcium, serum-high (hypercalcemia) | >ULN - 11.5 mg/dL<br>>ULN - 2.9 mmol/L | >11.5 – 12.5 mg/dL<br>>2.9 – 3.1 mmol/L | >12.5 - 13.5 mg/dL<br>>3.1 - 3.4 mmol/L | >13.5 mg/dL<br>>3.4 mmol/L |
| Cholesterol, serum-high (hypercholesterolemia) | >ULN - 300 mg/dL<br>>ULN - 7.75 mmol/L | >300 – 400 mg/dL<br>>7.75 – 10.34 mmol/L | >400 – 500 mg/dL<br>>10.34 – 12.92 mmol/L | >500 mg/dL<br>>12.92 mmol/L |
| Creatinine | >ULN – 1.5×ULN | >1.5 – 3.0×ULN | >3.0 - 6.0×ULN | >6.0×ULN |
| GGT (γ-glutamyl transpeptidase) | >ULN – 3.0×ULN | >3.0 – 5.0×ULN | >5.0 – 20.0×ULN | >20.0×ULN |
| Glucose, serum-high (hyperglycemia) | Fasting glucose value:<br>>ULN – 160 mg/dL<br>>ULN – 8.9 mmol/L | Fasting glucose value:<br>>160 – 250 mg/dL<br>>8.9 – 13.9 mmol/L | >250 – 500 mg/dL;<br>>13.9 – 27.8 mmol/L;<br>hospitalization indicated | >500 mg/dL;<br>>27.8 mmol/L;<br>life-threatening<br>consequences |
| Glucose, serum-low (hypoglycemia) | <lln 55="" dl<br="" mg="" –=""><lln 3.0="" l<="" mmol="" td="" –=""><td>&lt;55 – 40 mg/dL<br/>&lt;3.0 – 2.2 mmol/L</td><td>&lt;40 – 30 mg/dL<br/>&lt;2.2 – 1.7 mmol/L</td><td>&lt;30 mg/dL<br/>&lt;1.7 mmol/L<br/>life-threatening<br/>consequences;<br/>seizures</td></lln></lln> | <55 – 40 mg/dL<br><3.0 – 2.2 mmol/L | <40 – 30 mg/dL<br><2.2 – 1.7 mmol/L | <30 mg/dL<br><1.7 mmol/L<br>life-threatening<br>consequences;<br>seizures |

Eisai 

# **Sponsor's Grading for Laboratory Values**

| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Phosphate, serum-low<br>(hypophosphatemia) | <lln 2.5="" dl<br="" mg="" –=""><lln 0.8="" l<="" mmol="" td="" –=""><td>&lt;2.5 – 2.0 mg/dL<br/>&lt;0.8 – 0.6 mmol/L</td><td>&lt;2.0 – 1.0 mg/dL<br/>&lt;0.6 – 0.3 mmol/L</td><td>&lt;1.0 mg/dL<br/>&lt;0.3 mmol/L<br/>life-threatening<br/>consequences</td></lln></lln> | <2.5 – 2.0 mg/dL<br><0.8 – 0.6 mmol/L | <2.0 – 1.0 mg/dL<br><0.6 – 0.3 mmol/L | <1.0 mg/dL<br><0.3 mmol/L<br>life-threatening<br>consequences |
| Potassium, serum-high (hyperkalemia) | >ULN - 5.5 mmol/L | >5.5 – 6.0 mmol/L | >6.0 – 7.0 mmol/L<br>hospitalization indicated | >7.0 mmol/L<br>life-threatening<br>consequences |
| Potassium, serum-low (hypokalemia) | <lln 3.0="" l<="" mmol="" td="" –=""><td><lln 3.0="" l;<br="" mmol="" –="">symptomatic;<br/>intervention indicated</lln></td><td>&lt;3.0 – 2.5 mmol/L<br/>hospitalization indicated</td><td>&lt;2.5 mmol/L<br/>life-threatening<br/>consequences</td></lln> | <lln 3.0="" l;<br="" mmol="" –="">symptomatic;<br/>intervention indicated</lln> | <3.0 – 2.5 mmol/L<br>hospitalization indicated | <2.5 mmol/L<br>life-threatening<br>consequences |
| Sodium, serum-high (hypernatremia) | >ULN – 150 mmol/L | >150 – 155 mmol/L | >155 – 160 mmol/L<br>hospitalization indicated | >160 mmol/L<br>life-threatening<br>consequences |
| Sodium, serum-low (hyponatremia) | <lln 130="" l<="" mmol="" td="" –=""><td>N/A</td><td>&lt;130 – 120 mmol/L</td><td>&lt;120 mmol/L<br/>life-threatening<br/>consequences</td></lln> | N/A | <130 – 120 mmol/L | <120 mmol/L<br>life-threatening<br>consequences |
| Triglyceride, serum-high (hypertriglyceridemia) | 150 – 300 mg/dL<br>1.71 – 3.42 mmol/L | >300 – 500 mg/dL<br>>3.42 – 5.7 mmol/L | >500 – 1000 mg/dL<br>>5.7 – 11.4 mmol/L | >1000 mg/dL<br>>11.4 mmol/L<br>life-threatening<br>consequences |
| Uric acid, serum-high (hyperuricemia) | >ULN – 10 mg/dL<br>≤0.59 mmol/L without<br>physiologic<br>consequences | N/A | >ULN – 10 mg/dL<br>≤0.59 mmol/L with<br>physiologic<br>consequences | >10 mg/dL<br>>0.59 mmol/L<br>life-threatening<br>consequences |

ALT = alanine aminotransferase (serum glutamic pyruvic transaminase), AST = aspartate aminotransferase (serum glutamic oxaloacetic transaminase), GGT =  $\gamma$ -glutamyl transpeptidase, N/A = not applicable, LLN = lower limit of normal, ULN = upper limit of normal, WBC = white blood cell.

Based on Common Terminology Criteria for Adverse events (CTCAE) Version 4.0. Published: May 28, 2009 (v4.03: June 14, 2010).

# **Appendix 2 Inclusion/Exclusion Criteria Schedule**

Inclusion/exclusion criteria (Section 9.3.1 and Section 9.3.2) will be obtained at study visits as shown below.

#### Schedule of Inclusion/Exclusion Criteria Assessments (revised per Amendment 02)

| | V1 | V2 | V3 | V4 | V5 |
|---|---|---|---|---|---|
| Visit Name | Screening | Screening 2 | During Run-In<br>Period | During Run-<br>In Period | Baseline Period<br>(just prior to<br>Randomization) |
| Inclusion<br>Criterion<br>Number | 11, 12, 13, 14, 15,<br>16, 114, 115 | 17, 18, 19 | I6, I10, I11,<br>I12, I13 | I13 | N/A |
| Exclusion<br>Criterion<br>Number | E1, E2, E3, E5,<br>E6, E7, E8, E9,<br>E10, E11, E12,<br>E13, E14, E15,<br>E16, E17, E18,<br>E19, E20, E21,<br>E23, E24, E25,<br>E26, E27, E28 | E4, E21 ,E22,<br>E24, E25 | E24, E25 | E25 | E24, E25 |

N/A = not applicable, V = visit.

# **Appendix 3 List of Prohibited Concomitant Medications**

If a medication is not presented in the list below, but does fit into a class of medications noted in the list, the Medical Monitor must be consulted to determine whether it is permitted.

| Category | Medication |
|---|---|
| Anticholinergics (centrally-acting) | - |
| Anticonvulsants with known sedating effects | <ul> <li>Barbiturates</li> <li>Benzodiazepines</li> <li>GABA analogues</li> </ul> |
| Antihistamines (centrally-acting H1, including over-the- | <ul> <li>Hydantoins</li> <li>Phenyltriazines</li> <li>Diphenhydramine HCl</li> </ul> |
| counter) | <ul> <li>Carbinoxamine</li> <li>Doxylamine</li> <li>Dimenhyrinate</li> <li>Triprolidine</li> <li>Bromopheniramine</li> <li>Chlorphenamine</li> </ul> |
| | <ul><li>Hydroxazine<br/>(revised per Amendment 02)</li></ul> |
| Antihistamines with known sedating effects | <ul> <li>Non-sedating, eg, Claritin™ is not<br/>prohibited</li> </ul> |
| Anxiolytics with known sedating effects | <ul><li>Lorazepam</li><li>Alprazolam</li><li>Buspirone</li></ul> |
| Strong CYP3A inhibitors | <ul> <li>Amiodarone</li> <li>Bocepravir</li> <li>Clarithomycin</li> <li>Cobicistat</li> </ul> |
| | <ul> <li>Conivaptan</li> <li>Diltiazem</li> <li>Danoprevir</li> <li>Eltegravir</li> </ul> |
| | <ul> <li>Fluvoxamine</li> <li>Grapefruit juice</li> <li>Idelalisib</li> <li>Indinavir</li> </ul> |
| | <ul> <li>Itraconazole</li> <li>Ketoconazole</li> <li>Lopinavir</li> <li>Mibefradil</li> </ul> |
| | <ul><li>Nefazodone</li><li>Nelfinavir</li><li>Posaconazole</li></ul> |
| | <ul> <li>Ritonavir</li> <li>Saquinavir</li> <li>Telapravir</li> <li>Telethromycin</li> </ul> |
| | <ul> <li>Telethromycin</li> <li>Tipranavi</li> <li>Troleandomycin</li> <li>Voriconazole <ul> <li>(revised per Amendment 02)</li> </ul> </li> </ul> |

Eisai 

| Moderate CYP3A inhibitors O Amprenavir O Aprepitant O Atazanavir O Casopitant O Cimetidine O Ciprofloxacin O Clotrimazole O Crizotinib O Cyclosporin O Darunavir O Dronadarone O Erythromycin O Faldaprevir O Fluconazole |
|---|
| <ul> <li>Aprepitant</li> <li>Atazanavir</li> <li>Casopitant</li> <li>Cimetidine</li> <li>Ciprofloxacin</li> <li>Clotrimazole</li> <li>Crizotinib</li> <li>Cyclosporin</li> <li>Darunavir</li> <li>Dronadarone</li> <li>Erythromycin</li> <li>Faldaprevir</li> <li>Fluconazole</li> </ul> |
| <ul> <li>Atazanavir</li> <li>Casopitant</li> <li>Cimetidine</li> <li>Ciprofloxacin</li> <li>Clotrimazole</li> <li>Crizotinib</li> <li>Cyclosporin</li> <li>Darunavir</li> <li>Dronadarone</li> <li>Erythromycin</li> <li>Faldaprevir</li> <li>Fluconazole</li> </ul> |
| <ul> <li>Casopitant</li> <li>Cimetidine</li> <li>Ciprofloxacin</li> <li>Clotrimazole</li> <li>Crizotinib</li> <li>Cyclosporin</li> <li>Darunavir</li> <li>Dronadarone</li> <li>Erythromycin</li> <li>Faldaprevir</li> <li>Fluconazole</li> </ul> |
| <ul> <li>Cimetidine</li> <li>Ciprofloxacin</li> <li>Clotrimazole</li> <li>Crizotinib</li> <li>Cyclosporin</li> <li>Darunavir</li> <li>Dronadarone</li> <li>Erythromycin</li> <li>Faldaprevir</li> <li>Fluconazole</li> </ul> |
| <ul> <li>Ciprofloxacin</li> <li>Clotrimazole</li> <li>Crizotinib</li> <li>Cyclosporin</li> <li>Darunavir</li> <li>Dronadarone</li> <li>Erythromycin</li> <li>Faldaprevir</li> <li>Fluconazole</li> </ul> |
| <ul> <li>Clotrimazole</li> <li>Crizotinib</li> <li>Cyclosporin</li> <li>Darunavir</li> <li>Dronadarone</li> <li>Erythromycin</li> <li>Faldaprevir</li> <li>Fluconazole</li> </ul> |
| <ul> <li>Crizotinib</li> <li>Cyclosporin</li> <li>Darunavir</li> <li>Dronadarone</li> <li>Erythromycin</li> <li>Faldaprevir</li> <li>Fluconazole</li> </ul> |
| <ul> <li>Cyclosporin</li> <li>Darunavir</li> <li>Dronadarone</li> <li>Erythromycin</li> <li>Faldaprevir</li> <li>Fluconazole</li> </ul> |
| <ul> <li>Darunavir</li> <li>Dronadarone</li> <li>Erythromycin</li> <li>Faldaprevir</li> <li>Fluconazole</li> </ul> |
| <ul> <li>Dronadarone</li> <li>Erythromycin</li> <li>Faldaprevir</li> <li>Fluconazole</li> </ul> |
| <ul> <li>Erythromycin</li> <li>Faldaprevir</li> <li>Fluconazole</li> </ul> |
| <ul><li>Faldaprevir</li><li>Fluconazole</li></ul> |
| o Fluconazole |
| l Pi · |
| o Fluvoxamine |
| o Imatinib |
| o Netupitant |
| o Tofisopam |
| o Verapamil |
| (revised per Amendment 02) |
| CYP3A inducers o Avasimibe |
| o Bosentan |
| o Carbamazepine |
| o Efavirenz |
| o Enzaluteamide |
| o Etravirine |
| o Lersivirine |
| o Modafinil |
| o Mitotane |
| o Nafeillin |
| o Phenobarbital |
| o Phenytoin |
| o Rifabutin |
| o Rifampin |
| o St. John's Wort |
| o Troglitazone |
| o Talviraline |
| <ul> <li>Thiroiridazine</li> </ul> |
| (revised per Amendment 02) |
| Aypnotics O Melatonin |
| o Prescribed or OTC |
| Herbal preparations with sedating effects - |
| MAOIs - |
| Opioid Analgesics - |
| Muscle relaxants (centrally-acting) with known sedating O GABA analogues |
| effects o Hydantoins |
| o Phenyltriazines |
| Stimulants • Amphetamines |
| o Modafinil |
| o Armodafinil |
| <ul> <li>Methylfenidate</li> </ul> |

Eisai 

| Category | Medication |
|----------|----------------------------------------------------|
| Other | <ul> <li>Warfarin, heparin, ticlopidine</li> </ul> |
| | <ul> <li>Non-stimulant diet pills</li> </ul> |
| | <ul> <li>Systemic isoretinoin</li> </ul> |
| | <ul> <li>Systemic glucocorticoids</li> </ul> |
| | o Tryptophan |
| | (revised per Amendment 01) |

#### PROTOCOL SIGNATURE PAGE

**Study Protocol Number:** E2006-G000-304

**Study Protocol Title:** A Multicenter, Randomized, Double-Blind, Placebo-Controlled,

Active Comparator, Parallel-Group Study of the Efficacy and Safety of Lemborexant in Subjects 55 Years and Older with Insomnia

Disorder

**Investigational Product** 

Name:

E2006/lemborexant

**IND Number:** 111,871

**EudraCT Number:** 2015-004347-39



#### **INVESTIGATOR SIGNATURE PAGE**

**Study Protocol Number:** E2006-G000-304

**Study Protocol Title:** A Multicenter, Randomized, Double-Blind, Placebo-Controlled,

Active Comparator, Parallel-Group Study of the Efficacy and Safety of Lemborexant in Subjects 55 Years and Older with Insomnia

Disorder

**Investigational Product** 

Name:

E2006/lemborexant

**IND Number:** 111,871

**EudraCT Number:** 2015-004347-39

I have read this protocol and agree to conduct this study in accordance with all stipulations of the protocol and in accordance with International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) and all applicable local Good Clinical Practice (GCP) guidelines, including the Declaration of Helsinki.

| Medical Institution | | |
|---------------------|-----------|------|
| Investigator | Signature | Date |